# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for

DMID Protocol: 14-0031 Study Title:

A Phase 1 Double-Blinded, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety and Immunogenicity of Double Mutant Heat-Labile Toxin LTR192G/L211A (dmLT) from Enterotoxigenic *Escherichia coli* (ETEC) by Oral, Sublingual, or Intradermal Vaccination in Adults Residing in an Endemic Area

NCT03548064

Version 1.0

**DATE: 16 AUG-2021** 

THIS COMMUNICATION IS PRIVILEGED AND CONFIDENTIAL

# **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 14-0031 |
|---|---|
| <b>Development Phase:</b> | Phase 1 |
| Products: | Attenuated, Recombinant Double Mutant Heat-Labile Toxin (dmLT) from Enterotoxigenic <i>Escherichia coli</i> (ETEC), LT(R192G/L211A) |
| Form/Route: | Oral, Sublingual, and Intradermal |
| Indication Studied: | Escherichia coli (E. coli) |
| Sponsor: | Division of Microbiology and Infectious Diseases National Institute of Allergy and Infectious Diseases National Institutes of Health |
| Clinical Trial Initiation Date: | 11 January 2018 |
| Clinical Trial Completion Date: | |
| Date of the Analysis Plan: | August 16 <sup>th,</sup> 2021 |
| Version Number: | Version 1.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# TABLE OF CONTENTS

| STUDY | TITLE | П |
|---|---|---|
| TABLE | OF CONTENTS | III |
| LIST OF | F ABBREVIATIONS | VI |
| 1. | PREFACE | 1 |
| 2. | INTRODUCTION | 2 |
| 2.1. | Purpose of the Analyses. | 3 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 4 |
| 3.1. | Study Objectives | 4 |
| 3.2. | Endpoints | 4 |
| 3.2.1. | Primary Outcome Measures | 4 |
| 3.2.2. | 3.2.2 Secondary Outcome Measures | 4 |
| 3.2.3. | Exploratory Outcome Measures | 5 |
| 3.3. | Study Definitions and Derived Variables | 5 |
| 4. | INVESTIGATIONAL PLAN | 8 |
| 4.1. | Overall Study Design and Plan | 8 |
| 4.2. | Discussion of Study Design, Including the Choice of Control Groups | 8 |
| 4.3. | Selection of Study Population | 8 |
| 4.4. | Treatments | 10 |
| 4.4.1. | Treatments Administered. | 10 |
| 4.4.2. | Identity of Investigational Product(s) | 10 |
| 4.4.3. | Method of Assigning Subjects to Treatment Groups (Randomization) | 11 |
| 4.4.4. | Selection of Doses in the Study | 11 |
| 4.4.5. | Selection and Timing of Dose for Each Subject | 11 |
| 4.4.6. | Blinding | 11 |
| 4.4.7. | Prior and Concomitant Therapy | 12 |
| 4.4.8. | Treatment Compliance | 12 |
| 4.5. | Immunogenicity and Safety Variables | 12 |
| 4.5.1. | Safety Variables | 12 |
| 4.5.2. | Immunogenicity Variables | 13 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 14 |

# **Table of Contents** (continued)

| 6. | GENERAL STATISTICAL CONSIDERATIONS | 15 |
|---|---|---|
| 6.1. | General Principles | 15 |
| 6.2. | Timing of Analyses be stratified by route of administration with a column | |
| | for each | |
| 6.3. | Analysis Populations | |
| 6.3.1. | Safety Population | 15 |
| 6.3.2. | Modified-Intention-To-Treat (mITT) Immunogenicity Population | 15 |
| 6.3.3. | Per Protocol (PP) Immunogenicity Population | 15 |
| 6.4. | Covariates and Subgroups | 16 |
| 6.5. | Missing Data | 16 |
| 6.6. | Interim Analyses and Data Monitoring | 16 |
| 6.6.1. | Safety Review | 16 |
| 6.6.2. | Immunogenicity Review | 16 |
| 6.6.3. | Halting Rules | 17 |
| 6.7. | Multicenter Studies | 17 |
| 6.8. | Multiple Comparisons/Multiplicity | 18 |
| 7. | STUDY SUBJECTS | 19 |
| 7.1. | Disposition of Subjects | 19 |
| 7.2. | Protocol Deviations | 19 |
| 8. | IMMUNOGENICITY EVALUATION | 20 |
| 8.1. | Primary Immunogenicity Analysis | 20 |
| 8.2. | Secondary Immunogenicity Analyses | 20 |
| 8.3. | Exploratory Immunogenicity Analyses | 21 |
| 9. | SAFETY EVALUATION | 24 |
| 9.1. | Demographic and Other Baseline Characteristics | 24 |
| 9.1.1. | Prior and Concurrent Medical Conditions | 24 |
| 9.1.2. | Prior and Concomitant Medications | 24 |
| 9.2. | Measurements of Treatment Compliance | 24 |
| 9.3. | Adverse Events | 24 |
| 9.3.1. | Solicited Events and Symptoms | 24 |
| 9.3.2. | Unsolicited Adverse Events | 25 |

# **Table of Contents** (continued)

| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 25 |
|---|---|---|
| 9.5. | Pregnancies | 26 |
| 9.6. | Clinical Laboratory Evaluations | 26 |
| 9.7. | Vital Signs and Physical Evaluations | 26 |
| 9.8. | Concomitant Medications | 27 |
| 9.9. | Other Safety Measures | 27 |
| 10. | PHARMACOKINETICS | 28 |
| 11. | IMMUNOGENICITY | 29 |
| 12. | OTHER ANALYSES | 30 |
| 13. | REPORTING CONVENTIONS | 31 |
| 14. | TECHNICAL DETAILS | 32 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 33 |
| 16. | REFERENCES | 34 |
| 17. | LISTING OF TABLES, FIGURES, AND LISTINGS | 35 |
| APPENI | DICES | 36 |
| APPENI | DIX 1. TABLE MOCK-UPS | 37 |
| APPENI | DIX 2. FIGURE MOCK-UPS | 247 |
| APPENI | DIX 3. LISTINGS MOCK-UPS | 303 |

# LIST OF ABBREVIATIONS

| AE | Adverse Event/Adverse Experience |
|---------|--------------------------------------------------------------------|
| ALS | Antibodies in Lymphocyte Supernatant |
| ALT | Alanine Aminotransferase, formerly called SGPT |
| ANC | Absolute Neutrophil Count |
| ASC | Antibody Secreting Cells |
| CI | Confidence Interval |
| CRF | Case Report Form |
| CVD | Center for Vaccine Development-Global Health |
| CyTOF | Cytometry by Time-of-Flight, or Mass Cytometry |
| DHHS | Department of Health and Human Services |
| DMID | Division of Microbiology and Infectious Diseases, NIAID, NIH, DHHS |
| dmLT | Double-Mutant Heat-Labile Toxin |
| DSMB | Data and Safety Monitoring Board |
| eCRF | Electronic Case Report Form |
| ELISA | Enzyme-Linked Immunosorbent Assay |
| ELISpot | Enzyme-Linked ImmunoSpot Assay |
| ETEC | Enterotoxigenic Escherichia coli |
| FDA | Food and Drug Administration, DHHS |
| HBsAg | Hepatitis B Virus Surface Antigen |
| HCV | Hepatitis C Virus |
| icddr,b | International Centre for Diarrhoeal Disease Research, Bangladesh |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| ID | Intradermal |
| Ig | Immunoglobulin |
| ISM | Independent Safety Monitor |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MM | Medical Monitor |
| NIAID | National Institute of Allergy and Infectious Diseases, NIH, DHHS |
| NIH | National Institutes of Health |
| PATH | Program for Appropriate Technology in Health, now simply "PATH" |
| PBMC | Peripheral Blood Mononuclear Cells |
| • | • |

# **List of Abbreviations** (continued)

| PI | Principal Investigator |
|------|--------------------------------------------------|
| SAE | Serious Adverse Event/Serious Adverse Experience |
| SDCC | Statistical and Data Coordinating Center |
| SL | Sublingual |
| WBC | White Blood Cell |
| WHO | World Health Organization |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Phase 1 Double-Blinded, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety and Immunogenicity of Double Mutant Heat-Labile Toxin LTR192G/L211A (dmLT) from Enterotoxigenic Escherichia coli (ETEC) by Oral, Sublingual, or Intradermal Vaccination in Adults Residing in an Endemic Area" (DMID Protocol 14-0031) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for immunogenicity and safety outcomes, and (4) a list of proposed tables and figures. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

ETEC remains a major cause of childhood diarrhea in low-middle income (i.e., developing) countries and is endemic to areas with poor infrastructure for sanitation and without access to clean water. The use of dmLT is proposed as an oral, sublingual (SL), or intradermal (ID) traveler's diarrhea vaccine for persons from industrialized (i.e., developed) countries that visit high-risk developing (non-industrialized) countries. It is envisioned that dmLT may also be used as a component of candidate ETEC vaccines under development for use in infants and young children living in ETEC endemic areas. The National Institute of Allergy and Infectious Disease (NIAID) sponsored a Phase 1 dose-escalation study of healthy adult participants who received a single oral dose of dmLT (DMID Protocol 09-0066). No participants experienced diarrhea in any dosage group and the vaccine was well tolerated. Although the immune responses were limited in those receiving 5 µg or 25 µg of dmLT, the immune response was greater in those receiving 50 µg or 100 µg of dmLT, with a possible plateauing of immune responses at 50 µg.[1] A Phase 1 study of an inactivated oral multivalent ETEC vaccine (ETVAX, expressing CFA/I, CS3, CS5, CS6, and LTB) with dmLT as an adjuvant was conducted in 129 healthy Swedish adults. The vaccine with dmLT was safe and well tolerated; dmLT appeared to further enhance mucosal immune responses to CF antigens which were present in low amounts in the vaccine.[2] A Phase 1/2 study (VAC 014/OEV-122) of oral administration of an inactivated ETEC vaccine (ETVAX) with and without dmLT and a Phase 2 study (NCT02531802) of the oral ETEC vaccine (ETVAX) administered with dmLT among healthy adults in Bangladesh are ongoing at the International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b). A Phase 1/2b study of a live, attenuated oral ETEC vaccine (ACE527) adjuvanted with dmLT was conducted in the United States (VAC 006). The trial results have not yet been published, but the data have been presented at scientific conferences. Immunization with ACE527 administered with dmLT was safe and immunogenic and protecting against diarrhea upon challenge.[3] NIAID sponsored a Phase 1 dose-escalation study in healthy adult participants who received three sequential SL or Oral doses of dmLT (DMID Protocol 12-0023). Delivery of dmLT to Cohorts 1-4 were completed and no safety concerns were identified with up to the 3 doses of 50 µg dmLT delivered orally. The study is completed; there have been no noted safety concerns. There are no other human trials, to our knowledge, that have been completed using SL route of administration of dmLT as a vaccine or adjuvant. NIAID is currently sponsoring a Phase 1 dose-escalation trial with dmLT administered in three sequential doses via the ID route (DMID Protocol 13-0013), the first in human trial with dmLT administered via the ID route. The trial has progressed through doses up to 2.0 µg without safety concerns. The aforementioned DMID-sponsored studies on dmLT have been or are being conducted in the United States (an industrialized country) and there are unanswered questions regarding the immune responses through different routes of administration in a non-industrialized country. This study was designed to assess the safety and immune responses of a range of doses of dmLT when administered by the oral, SL, or ID route, in participants residing in an endemic country for ETEC disease. Compared to oral immunization, SL or ID immunization may increase dose-sparing, which would help reduce the cost of the final vaccine product, and potentially eliminate the need for buffering to neutralize gastric acid, therefore providing greater protein antigen stability. Both the SL and ID routes may also help bypass gut enteropathy, a major barrier to oral vaccination. The proposed indication for dmLT is to protect against ETEC diarrhea associated with infection by strains expressing the E. coli heat-labile enterotoxin alone or in combination with the heat-stable toxin as a component of an oral, sublingual, or intradermal diarrhea vaccine for those residing in high risk endemic regions as well as international travelers to these high-risk regions.

# 2.1. Purpose of the Analyses

These analyses assess the safety, reactogenicity, and immunogenicity of a range of doses of dmLT administered via the oral, sublingual, or intradermal route and will be included in the clinical study report.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

#### **Primary**

• To assess the reactogenicity, safety and tolerability of dmLT when administered in three sequential doses, over a range of dosages by oral, sublingual, or intradermal routes

#### **Secondary**

- To assess the long-term safety, from first vaccination through 6 months following the last dose of vaccine
- To evaluate the serum anti-dmLT Immunoglobulin IgG and IgA response
- To evaluate the IgG and IgA anti-dmLT Antibody Secreting Cell (ASC) response
- To evaluate the IgG and IgA anti-dmLT Antibodies in Lymphocyte Supernatant (ALS) response
- To evaluate the total fecal IgA and fecal anti-dmLT IgA response
- To evaluate the total salivary IgA and the saliva-derived anti-dmLT IgA response

#### **Exploratory**

- To measure the mucosal homing of IgA anti-dmLT ASC
- To measure the serum toxin neutralizing antibody response
- To measure the dmLT-specific IgG and IgA memory B cell response
- To determine the dmLT-specific effector and memory T cell responses

# 3.2. Endpoints

#### 3.2.1. Primary Outcome Measures

The **Primary Safety Endpoints** to be used to evaluate reactogenicity, safety and tolerability are as follows:

- The occurrence of solicited local site and systemic reactogenicity events from vaccination through 7 days after each dose of vaccine is administered
- The occurrence of study withdrawals throughout the study
- The occurrence of discontinuation of study vaccination during the study
- The occurrence of unsolicited vaccine-related adverse events (AE), including laboratory AE, from first vaccination through 28 days after the last dose of vaccine is administered

#### 3.2.2 Secondary Outcome Measures

The **Secondary Safety Endpoints** to be used to evaluate the safety of this study are:

• The occurrence of vaccine-related serious adverse events (SAE) from the first vaccination through 6 months after the last dose of vaccine was administered

•

The **Secondary Immunogenicity Endpoints** to be used to evaluate the immune response to vaccination consist of the following:

- At any time after vaccination, the proportion of participants with a ≥4-fold rise in dmLT-specific serum IgG and IgA titers over baseline measured by Enzyme-Linked Immunosorbent Assay (ELISA)
- At any time after vaccination the proportion of participants with ≥8 dmLT-specific IgA or IgG ASC / 10<sup>6</sup> peripheral blood mononuclear cells (PBMC) as measured by Enzyme-Linked ImmunoSpot Assay (ELISpot)
- At any time after vaccination, the proportion of participants with ≥2-fold rise in ALS anti-dmLT-specific IgG and IgA titers over baseline measured by ELISA
- At any time after vaccination, the proportion of participants with a ≥4-fold rise over baseline in dmLT-specific fecal IgA titers measured by ELISA
- At any time after vaccination, the proportion of participants with a ≥4-fold rise over baseline in dmLT-specific salivary IgA titers measured by ELISA

## 3.2.3. Exploratory Outcome Measures

The **Exploratory Endpoints** to be used to evaluate the immune response to vaccination consist of the following:

- Geometric mean titers of dmLT-specific IgG and IgA in ALS measured by ELISA
- Geometric mean titers of dmLT-specific serum IgG and IgA measured by ELISA
- Mean and median number of dmLT-specific IgG and IgA ASC measured by EliSpot
- Geometric mean titers of dmLT-specific fecal IgA measured by ELISA
- Geometric mean titers of dmLT-specific salivary IgA measured by ELISA
- The proportion of participants with dmLT-specific memory B cell response as measured by ELISpot
- At any time after vaccination, the proportion of participants with anti-dmLT IgG and IgA ASC in circulation expressing gut homing receptors (integrin  $\alpha 4\beta 7$  in the absence or presence of CD62L) measured by EliSpot assay
- At any time after vaccination, proportion of participants with ≥4-fold rise over baseline in toxin neutralization titers measured by Y-1 cell assay
- At any time after vaccination, the proportion of participants with dmLT-specific effector and memory T cell responses as measured by Cytometry by Time-of-Flight, or Mass Cytometry (CyTOF).

# 3.3. Study Definitions and Derived Variables

The baseline value will be defined as the last value obtained prior to the first vaccination/dose of study product. If a participant has repeated laboratory values on the same day, the value from the last evaluation will be used for analysis. Post-baseline, in the case of multiple observations (for example, from supplemental visits), the assessment value that is closest to the scheduled visit window will be used in the analyses. All the recorded data will be listed. If observations have the same distance to the scheduled assessment, the latest one will be used.

An adverse event (AE) is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product. Any medical condition that is present at the time that the participant is screened will be considered as baseline and not reported as an AE. However, if the severity of any pre-existing medical condition increases, it will be reported as an AE.

AEs are graded for severity and assessed for relationship to study product as defined below.

The severity of Laboratory, Vital Sign, and Solicited AEs are to be graded according to the standard criteria shown in Table 7, Table 8, and Table 9. For all other AEs severity is defined as follows:

- Mild (Grade 1): Events require minimal or no treatment and do not interfere with the participant's daily activities.
- Moderate (Grade 2): Events result in a low level of inconvenience or concern with therapeutic measures. Moderate events may cause some interference with functioning and daily activities.
- Severe (Grade 3): Events interrupt the participant's usual daily activities and may require systemic drug therapy or other treatment. Severe events are usually incapacitating.

For all AEs relationship to study product is defined as follow:

- Related There is a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event.
- Not Related There is not a reasonable possibility that the administration of the study product caused the event.

A SAE will be defined as an adverse event or suspected adverse reaction that, in the view of either the site principal investigator or sponsor, results in any of the following outcomes:

- Death,
- A life-threatening adverse event, defined as an adverse event the occurrence of which, in the view of either the site principal investigator or sponsor, places the participant at immediate risk of death. It does not include an adverse event that, had it occurred in a more severe form, might have caused death.
- Inpatient hospitalization (defined by local practice as the study participant being present in the hospital greater than 24 hours) or prolongation of existing hospitalization,
- A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
- A congenital anomaly/birth defect.
- Important medical events that may not result in death, be life-threatening, or require hospitalizations may be considered serious when, based upon appropriate medical judgment they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

Serum dmLT-specific Ig response is defined as a ≥4-fold rise in dmLT-specific serum

Ig titers over baseline.

ASC dmLT-specific Ig response is defined as ≥8 dmLT-specific Ig ASC /10<sup>6</sup> PBMC.

Serum dmLT-specific toxin neutralization response is defined as a ≥4-fold rise over baseline in toxin neutralization titers.

ALS response is defined as a  $\geq$ 2-fold rise in ALS anti-dmLT-specific Ig titers over baseline.

Salivary response is defined as a  $\geq$ 4-fold rise over baseline in dmLT-specific salivary IgA titers.

Fecal response is defined as a  $\geq$ 4-fold rise over baseline in dmLT-specific fecal IgA titers.

ASC Homing response is defined as the presence of dmLT-specific circulating ASC expressing gut homing receptors (integrin  $\alpha 4\beta 7$  in the absence or presence of CD62L).

B memory response is defined as a  $\geq$ 0.05% increase from baseline in the percentage of antigen-specific Ig /total Ig B memory cells.

T cell response is defined as an increase of >0.05% from baseline cell percentage.

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

This is a phase 1, single center, randomized, double-blinded, placebo controlled, dose escalation clinical trial in which 135 healthy males and non-pregnant females ages 18-45 who met all eligibility criteria were to receive 3 doses of either dmLT vaccine or placebo, randomized in a 4:1 ratio. Cohort A and Cohort B participants received study product via oral administration. Cohort C and Cohort D participants received study product via sublingual administration. Cohort E participants received two of three planned doses of study product via intradermal administration prior to the study being terminated due to the COVID-19 pandemic. No participants were enrolled in planned Cohorts F, G, H, or I. Participants were screened by history, physical exam, and clinical laboratory tests, including a urine or serum pregnancy test for women of childbearing potential. A schematic of the planned study design is presented in Table 1.

# 4.2. Discussion of Study Design, Including the Choice of Control Groups

This study was designed to assess the safety and immune responses of a range of doses of dmLT when administered by the oral, SL, or ID route; in participants residing in an endemic country for ETEC disease. Cohorts A and B received 3 vaccinations via the oral route at escalating doses. Cohorts C and D received 3 vaccinations via the sublingual route at escalating doses. Cohorts E received 2 vaccinations via the intradermal route. Three placebo recipients per cohort were included in the study in order to blind the participants and observer and not as a comparison group.

# 4.3. Selection of Study Population

The study population for DMID protocol 14-0031 is males and non-pregnant females, 18 to 45 years old, inclusive, who are in good health and meet all eligibility criteria. Potential participants were screened from the general population at the International Centre for Diarrheal Disease Research, Mirpur, Bangladesh.

#### **Subject Inclusion Criteria**

Study participants were eligible for this study if they fulfilled the inclusion criteria below:

- 1. Male or female age 18-45 years old, inclusive.
- 2. Provides written informed consent before initiation of any study procedures.
- 3. Healthy as judged by the site investigators and determined by medical history, medication history, and physical examination.
- 4. Capable of understanding, consenting, and complying with all the study visits and procedures.
- 5. Body Mass Index of no less than 18.5
- 6. Agrees not to participate in another clinical trial during the study period.
- 7. Agrees to complete all study visits and procedures.
- 8. Agrees not to donate blood to a blood bank for 12 months after receiving the last vaccine.

#### **Subject Exclusion Criteria**

Participants were ineligible for any of the following conditions or reasons:

- 1. Women who are pregnant or lactating or have a positive urine pregnancy test at screening or on the day of vaccinations.
  - \*Note: all women presenting for screening will have urine pregnancy testing. "Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control from screening and through 28 days post last dose of vaccine. Abstinence is also acceptable."
- 2. Presence or history of a chronic medical condition\* that would, in the opinion of the investigator, render vaccination unsafe or interfere with the evaluation of the vaccine.
  - \* Note: this may include, but is not limited to: significant renal disease, unstable or progressive neurological disorders, diabetes, heart disease, asthma, lung disease, liver disease, organ transplant recipients and cancer.
- 3. Presence of a significant dermatologic condition\*, or tattoo(s), scarring or significant skin damage at the vaccination site that would impede evaluation of local reactogenicity.
  - \* Note: this may include severe eczema, psoriasis or history of keloid formation. Participants with history of squamous cell or basal cell skin cancer that has been surgically excised and considered cured may be enrolled in the study if the skin cancer site is healed and is not at proposed vaccine administration site.
- 4. Any developmental abnormality of the palate.
- 5. Participants diagnosed with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation.
- 6. Use of long-term (≥2 weeks) oral steroids, intranasal or topical prednisone (or equivalent), parenteral steroids, or high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months.
- 7. Has major psychiatric illness\* during last 12 months that in the investigator's opinion would preclude participation.
  - \* Note: Participants taking antipsychotic or antimanic drugs should not be enrolled. These include: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, lamotrigine, gabapentin, topiramate, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate, or lithium citrate. Participants taking a single antidepressant drug and are stable without decompensating symptoms in the preceding 3 months can be enrolled in the study.
- 8. Use of prescription or over-the-counter (OTC) anti-inflammatory medications\* 48 hours prior to receiving the investigational product.
  - \* Note: This includes naproxen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs.
- 9. Gastrointestinal symptoms\* in the past 24 hours or abdominal pain lasting for more than 2 weeks in the past 6 months.
  - \*Note: this may include, but is not limited to: abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting.
- 10. Moderate or severe diarrheal illness\* during the 6 weeks prior to enrollment.
  - \*Note: Moderate or severe diarrheal illness is defined by the passage of  $\geq$  4 unformed or loose stools (mix of liquid and solid components) in a 24-hour period

- 11. History of chronic gastrointestinal illness\*.
  - \*Note: this includes severe dyspepsia or gastroesophageal reflux disease, constipation, irritable bowel syndrome (IBS), hemorrhoids, diverticular disease, colitis, colon polyps, colon cancer, and inflammatory bowel disease. Mild or moderate heartburn or epigastric pain occurring no more than three times per week is permitted.
- 12. Regular use (weekly or more often) of laxatives, anti-diarrheal, anti-constipation, or antacid therapy.
- 13. History of major gastrointestinal surgery, excluding uncomplicated appendectomy or cholecystectomy.
- 14. History of systemic antimicrobial treatment (i.e., topical treatments are not an exclusion) during the week prior to any administration of dmLT.
- 15. Acute febrile illness (body temperature ≥38°C) during the week prior to enrollment.
- 16. Abnormal screening laboratories\*.
  - \*Note: screening labs include white blood cell count (WBC), absolute neutrophil count (ANC), hemoglobin (Hg), platelet count, serum creatinine, serum albumin, alanine aminotransferase (ALT, also known as SGPT), and serologic testing for Hepatitis B virus surface antigen (HBsAg) and Hepatitis C virus (HCV) antibody.
- 17. Isolation of specific bacteria\* from screening stool cultures.

  \*Note: bacteria include ETEC, Vibrio cholerae, and Shigella spp. Salmonella and Campylobacter will not be evaluated as part this criterion.
- 18. Received an inactivated licensed vaccine within 2 weeks of enrollment or live licensed vaccine within 4 weeks of enrollment.
- 19. Received a cholera (licensed or experimental) vaccine, *E. coli* vaccine, or *Shigella* vaccine in the last 3 years.
- 20. History of receiving immune globulin or other blood product within the 3 months before enrollment in this study.
- 21. Currently enrolled in another study, involving an experimental agent. Participants involved in observational studies or surveys remain eligible.
- 22. Any condition that would, in the opinion of the Site Investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.
- 23. Known allergies to study compound or components of the study vaccine.
- 24. Donating blood in the 8 weeks prior to study entry.

#### 4.4. Treatments

#### 4.4.1. Treatments Administered

Participants were to be administered three doses of dmLT vaccine or placebo. Cohort E participants were administered two of three planned doses.

#### 4.4.2. Identity of Investigational Product(s)

LT(R192G/L211A), or dmLT, is a derivative of wild-type ETEC heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at

amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules. The protein has been designated LT(R192G/L211A) and has been extensively evaluated in pre-clinical animal studies for its ability to induce anti-dmLT antibody responses, as well as its capacity to adjuvant the immune responses for co-administered antigens.

The dmLT vaccine was provided by PATH Vaccine Solutions. All Cohorts received lot number 001-08-16 manufactured at IDT Biologika Dessau. Placebo (0.9% Sodium Chloride Injection, United States Pharmacopeia) and sodium bicarbonate (NaHCO3) buffer (used in delivery of the orally administered dmLT) were provided by Fisher BioServices.

## 4.4.3. Method of Assigning Subjects to Treatment Groups (Randomization)

The randomization code was prepared by the Statistical and Data Coordinating Center (SDCC), Emmes. Enrollment/randomization were performed through the enrollment module in the electronic data capture system, maintained by the SDCC.

For each cohort, eligible participants were randomized and assigned in a 4:1 ratio to dmLT (n = 12) or placebo (n = 3) groups. The randomization was based on a variable blocked scheme to provide an approximately balanced allocation to the treatment groups during the study.

#### 4.4.4. Selection of Doses in the Study

Oral dmLT administered alone in a dose of up to  $100~\mu g$  and together with an inactivated ETEC vaccine and live attenuated ETEC vaccine in a dose of up to  $25~\mu g$  have been found to be safe in Phase 1 studies. In DMID Protocol 09-0066 a single oral dose of dmLT in escalating doses of  $5~\mu g$ ,  $25~\mu g$ ,  $50~\mu g$ , and  $100~\mu g$  was found to be well tolerated and immunogenic, with immune responses plateauing at the  $50~\mu g$  dose. [1] In DMID Protocol 12-0023 three sublingual doses of dmLT in escalating doses of  $1~\mu g$ ,  $5~\mu g$ ,  $25~\mu g$ , and  $50~\mu g$  were found to be well tolerated with  $25~\mu g$  eliciting the most consistent immogenic response. [4] In DMID Protocol 13-0013 (CSR pending) three intradermal doses of dmLT in escalating doses of  $0.1~\mu g$ ,  $0.3~\mu g$ ,  $1.0~\mu g$ , and  $2.0~\mu g$  dmLT were administered with no safety signals observed.

#### 4.4.5. Selection and Timing of Dose for Each Subject

Cohort A and B participants received 3 doses administered orally in clinic on Day 1, Day 15, and Day 29. Cohort C and Cohort D received 3 doses administered sublingually in clinic on Day 1, Day 15, and Day 29. Cohort E participants received 2 doses administered intradermally in clinic on Day 1, Day 22.

## 4.4.6. Blinding

This is a double-blind study. While participants and study personnel were not blinded to cohort and route of administration, they were blinded to group assignment (i.e., placebo vs. vaccine) within a cohort. Study product was administered by an unblinded study product administrator, a study personnel licensed, registered, or certified to administer vaccines, who was not involved in study-related assessments and had no participant contact for data collection following study injection. Participants, investigators, and study personnel who performed any study-related assessments following study product administration, and laboratory personnel who performed immunologic assessments were blinded to the administration of vaccine or placebo, within each cohort. The randomization scheme was generated by the SDCC and provided only to the assigned unblinded study personnel (e.g., pharmacist who prepared study products and unblinded study product administrators). According to DMID policy, the study medical monitor (MM) responds to requests for

emergency unblinding, and instructs the SDCC to release treatment codes only if necessary to ensure that the participant receives appropriate clinical care. No emergency or other unplanned unblinding events occurred during the conduct of this study.

### 4.4.7. Prior and Concomitant Therapy

Participants were permitted to take birth control pills and vitamins throughout the course of the study; herbal supplements were not permitted. In addition, participants were instructed that prescription or OTC anti-inflammatory medications were not permitted in the 48 hours prior to receiving the investigational product. This included medications that contain naproxen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs. All concomitant medications (e.g., vitamins, antacids, analgesics, prescription medications) taken 28 days prior to vaccination were recorded in the concomitant medication data collection form. Any medications taken during the 7 days following a dose of vaccine were to be recorded on the participant's memory aid and/or reported to a research team member upon follow up clinic visit. All analgesics and prescription medications from 8 to 28 days post-vaccination were recorded in the concomitant medication data collection form.

If the investigator learned that a participant had taken a prohibited medication (see Section 4.3 inclusion/exclusion criteria) during the time immediately around the dosing of the investigational product, the investigator was to contact the DMID Clinical Project Manager and MO for instructions regarding the participant's continuation in the study.

## 4.4.8. Treatment Compliance

All participants received each dose of study product administered in the clinic. Participants were directly observed at the time of dosing by a member of the clinical research team who was licensed to administer vaccines.

# 4.5. Immunogenicity and Safety Variables

See Table 2 and Table 3 for a schedule of study procedures.

#### 4.5.1. Safety Variables

Safety, reactogenicity, and tolerability will be assessed by:

- 1. Frequency and Severity of Solicited Adverse Events reactogenicity events occurring from vaccination through 7 days after each dose of vaccine is administered:
  - a) Local solicited events include: irritation of the oral cavity or tongue, diarrhea, nausea, vomiting, and abdominal discomfort for Oral Cohorts; irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort for Sublingual Cohorts; and injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass for Intradermal Cohorts.
  - b) Systemic solicited events include: fever, feverishness, fatigue, malaise, myalgia, or headache for Oral and Sublingual Cohorts; and fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort for Intradermal Cohorts.
- 2. Frequency of participant withdrawals from first vaccination through the end of follow-up (Day 209 for Oral and Sublingual Cohorts, Day 223 for Intradermal Cohorts)
- 3. Frequency of discontinuation of study vaccination during the study

- 4. Frequency and severity of unsolicited vaccine-related non-serious adverse events (AE), including laboratory AE, from first vaccination through 28 days after the last dose of vaccine is administered (Day 57 for Oral and Sublingual Cohorts, Day 71 for Intradermal Cohorts)
- 5. Frequency of vaccine-related SAEs from the first vaccination through the end of follow-up (Day 209 for Oral and Sublingual Cohorts, Day 223 for Intradermal Cohorts)

#### 4.5.2. Immunogenicity Variables

Secondary and exploratory immunogenicity variables will be measured by the following assays:

- dmLT-specific serum IgG and IgA results as measured using ELISA will be reported by icddr,b lab for samples collected Days 1, 8, 15, 22, 29, 36, 57, and 114 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, 71, and 128 for Intradermal Cohorts.
- IgG and IgA anti-dmLT Antibody Secreting Cell (ASC) results as measured using ELISpot will be reported by icddr,b lab for samples collected Days 1, 8, 15, 22, 29, and 36 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, and 50 for Intradermal Cohorts.
- IgG and IgA anti-dmLT Antibodies in Lymphocyte Supernatant (ALS) results as measured using ELISA will be reported by icddr,b lab for samples collected Days 1, 8, 15, 22, 29, and 36 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, and 50 for Intradermal Cohorts.
- Total fecal IgA and fecal anti-dmLT IgA results as measured using ELISA will be reported by icddr,b lab for samples collected Days 1, 8, 15, 22, 29, 36, and 57 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, and 71 for Intradermal Cohorts.
- Total salivary IgA and the saliva-derived anti-dmLT IgA results as measured using ELISA will be reported by icddr,b lab for samples collected Days 1, 8, 15, 22, 29, 36, and 57 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, and 71 for Intradermal Cohorts.
- Mucosal homing of and IgG and IgA anti-dmLT ASC results as measured using ELISpot will be reported by icddr,b lab for samples collected Days 8, 22, and 36 for Oral and Sublingual Cohorts and at Days 8, 29, and 50 for Intradermal Cohorts.
- Serum toxin neutralizing antibody results as measured using Y-1 cell assay will be reported by the Center for Vaccine Development-Global Health (CVD) lab at the University of Maryland, Baltimore for samples collected Days 1, 8, 15, 22, 29, 36, 57, and 114 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, 71, and 128 for Intradermal Cohorts.
- dmLT-specific IgG and IgA memory B cell results as measured using ELISpot will be reported by icddr,b lab for samples collected Days 1, 22, 36, 57, 114, and 209 for Oral and Sublingual Cohorts and at Days 1, 29, 50, 71, 128, and 223 for Intradermal Cohorts.
- dmLT-specific effector and memory T cell results as measured using CyTOF will be reported by the Cellular Immunology Group of the CVD for samples collected at screening and on Days 22, 36, 57, 114, and 209 for Oral and Sublingual Cohorts and at screening and on Days 29, 50, 71, 128, and 223 for Intradermal Cohorts.

#### 5. SAMPLE SIZE CONSIDERATIONS

The sample size for each cohort was chosen based on the number of participants deemed appropriate for a Phase 1 study in which the vaccine has had limited experience by the different routes of administration in humans. Sample size was limited to at least 11 evaluable participants and up to 15 participants for each cohort (each of the nine planned cohorts A through I).

The DMID Data and Safety Monitoring Board (DSMB) was scheduled to review cumulative data after Cohorts A through F had completed safety data through 7 days post-third dose of vaccine. At which time each cohort had been expected to have at least 10 evaluable vaccinees (10 per cohort). Among the 10 vaccinees per dose, the absence of a dose-limiting AE provides for an upper 95% exact (Clopper-Pearson) confidence bound of 30.8%. The absence of a dose-limiting AE among 20 vaccinees per route (e.g., combining safety data from Cohort A and B) provides for an upper 95% confidence bound of 16.8%. If at the time of data review, there had been no dose-limiting AEs among 60 vaccinees (e.g., combining safety data from Cohorts A through F), this would have provided an upper 95% confidence bound of 6.0% (Table 4). There were no dose-limiting AEs among the 40 vaccinees (Cohort A through D) who received all three planned doses which provides an upper 95% confidence bound of 8.8%.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard deviation, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by site, treatment and participant, and when appropriate by visit number within participant. Summary tables will be structured with a column (or row) for each treatment in the order from left to right (or top to bottom): Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, All Oral Cohorts: Placebo, Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, All Sublingual Cohorts: Placebo, Cohort E: Intradermal 0.3 µg dmLT, Cohort E: Intradermal Placebo. Where necessary, summary tables will be stratified with oral and sublingual cohort columns presented in one table and intradermal cohort columns presented in the table immediately following. Tables will be annotated with the total population size relevant to that table/treatment, including any missing observations.

## 6.2. Timing of Analyses be stratified by route of administration with a column for each

The final analysis will be performed after database lock. No interim analysis was planned or performed.

# 6.3. Analysis Populations

Summaries and analysis of safety data will be presented for the Safety Population. Summaries and analysis of immunogenicity data will be presented for the mITT and Per Protocol Immunogenicity Population. A tabular listing of all participants, visits, and observations excluded from the analysis populations will be provided in the CSR (Listing 4).

#### **6.3.1.** Safety Population

The Safety Analysis population will include all eligible participants who received at least one dose of study product.

#### 6.3.2. Modified-Intention-To-Treat (mITT) Immunogenicity Population

The modified-intention-to-treat (mITT) immunogenicity population includes all eligible participants who received at least one dose of study product and contributed both pre- and at least one post-vaccination samples for immunogenicity testing for which valid results were reported.

## 6.3.3. Per Protocol (PP) Immunogenicity Population

The per protocol (PP) immunogenicity population includes all participants in the mITT subset with the following exclusions:

- Data from all available visits for participants found to be ineligible at baseline
- Data from all visits subsequent to major protocol deviations, such as:
  - Second or third vaccination not received
  - Second or third vaccination received out of window
  - o Receipt of non-study vaccines during the timeframe prohibited by the protocol
- Data from any visit that occurs substantially out of window

# 6.4. Covariates and Subgroups

The protocol did not define any formal subgroup analyses, and the study is not adequately powered to perform subgroup analyses.

## 6.5. Missing Data

All attempts were made to collect all data per protocol. No imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier. If data points are identified as outliers, sensitivity analyses will be performed to examine the impact of including or excluding the outliers. Any substantive differences in these analyses will be reported.

# 6.6. Interim Analyses and Data Monitoring

#### 6.6.1. Safety Review

There was no formal statistical interim analysis based on the safety data. Prior to dose escalation, safety data through 7 days post vaccination of the third dose was reviewed by the principal investigator (PI), MM, and DMID Independent Safety Monitor (ISM). A local DSMB reviewed safety data and provided a recommendation with enrollment and vaccination of the next successive dosage and route of administration cohort. The DMID DSMB was notified when the decision was made to progress to the next cohort. A meeting of the DMID DSMB was planned between Cohort F and Cohort G, but not held because the study was terminated after Cohort E.

#### 6.6.2. Immunogenicity Review

The immunology data was not a required element of the data for the DMID DSMB or local DSMB to review. There was no formal statistical interim analysis based on the immunology data planned or performed.

## 6.6.3. Dose Escalation Halting Criteria

Prior to dose escalation to the next cohort within a route of administration group (see Table 1), safety data through 7 days post vaccination of the third dose was reviewed. Specifically, the SDCC provided the cumulative safety data and notified the PI, MM, and DMID (ISM), that the following criteria had not been met based on a review of the safety data collected in the seven days after the third vaccination of the last participant in the current cohort. Only one cohort was enrolled at a time, and enrollment proceed from Cohort A to B; Cohort C to D, and Cohort E if the halting criteria described below are NOT met.

In addition, there would have been no progression to the next cohort within a route of administration group if the following dose escalation halting criteria had been met:

• The site PI, protocol PI, MM, DMID ISM or local DSMB identify a safety concern that would prompt a review by the DMID DSMB.

If the above dose escalation halting criteria were NOT met, the dose escalation proceed to the next successive route of administration cohort.

If any of the above dose escalation halting criteria had been met, then escalation to the next successive route of administration cohort would not have proceeded and the data would have been reviewed by the DMID DSMB.

## 6.6.3. Halting Rules

Further dosing of any participant only for the route (oral, SL, ID) would have been halted if any of the following criteria were met. The study would have been halted, and all further vaccine administration halted for DSMB review/recommendation if any of the following criteria had been met for each route of administration:

- Any participant experiences vaccine-related SAE (e.g., excluding trauma or accident) from the time of the first study vaccination through the participant's last study visit.
- Any participant experiences an injection site necrosis within 7 days of vaccination.
- Any participant experiences an anaphylactic reaction related to vaccine occurring within 24 hours after vaccination.
- Any participant experiences urticaria, laryngospasm, bronchospasm, or anaphylaxis determined to be related to vaccine and within 7 days of vaccination.
- Any participant experiences facial nerve neuropathy, within 28 days of vaccination, confirmed by an investigator and determined to be related to vaccine.
- Any participant experiences a death for any reason excluding trauma or accident.

In addition, the study would have been halted if two or more participants in the same cohort or three participants across all cohorts within a route of administration (who received at least one dose of study product) experienced:

- The same severe (Grade 3) study vaccine-related local solicited event,
- The same severe (Grade 3) study vaccine-related systemic solicited event,
- The same severe (Grade 3) study vaccine-related clinical laboratory test,
- The same severe (Grade 3) study vaccine-related vital sign, or
- Any other severe (Grade 3) AE of the same system organ class

Exceptions to this would have been:

• If there are obvious and acceptable physiological explanation for a Grade 3 abnormality (example, grade 3 hematuria in menstruating females)

If a halting rule had been met, further dosing of the respective route would have ceased, but follow-up visits would have continued. An *ad hoc* DMID DSMB meeting and local DSMB meeting would have been convened to discuss the halting event. If, following review by both the DMID DSMB and local DSMB, it had been deemed acceptable to restart the study, the study would have resumed, upon DMID's approval and authorization.

#### 6.7. Multicenter Studies

Not applicable. This study took place at a single site.

# 6.8. Multiple Comparisons/Multiplicity

This study was not designed to test any specific null hypothesis, and as such no adjustments for multiple testing are planned.

#### 7. STUDY SUBJECTS

# 7.1. Disposition of Subjects

Table 16 will present a summary of the reasons that participants were screened but not enrolled.

The composition of analysis populations, including reasons for participant exclusion, by treatment arm, is presented in Table 12 and Table 13.

The disposition of participants in the study will be tabulated by treatment group (Table 10 and Table 11). The table shows the total number of participants screened, enrolled, receiving at least 1 dose, receiving at least 2 doses, receiving all 3 doses, discontinued dosing or terminated from study follow-up and the number completing the study.

A flowchart showing the disposition of study participants, adapted from the Consort Statement [5] will be included (Figure 1, Figure 2, and Figure 3). This figure will present the number of participants screened, enrolled, lost to follow-up, and analyzed, by treatment arm.

A listing of participants who discontinued dosing or terminated from study follow-up and the reason will be included in Listing 1.

#### 7.2. Protocol Deviations

A summary of participant-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and treatment group for all participants (Table 5 and Table 6). Deviations that are considered major deviations that will be reviewed for possible participant exclusion from the per protocol population include: second or third vaccination not received or received out of window and receipt of non-study vaccines during the timeframe prohibited by the protocol. All participant-specific protocol deviations and non-participant specific protocol deviations will be included in as data listings (Listing 2 and Listing 3, respectively).

#### 8. IMMUNOGENICITY EVALUATION

Immune responses will be summarized at each time point within each route by treatment, pooling participants who received placebo. The number and percentage of participants with responses, as defined for each outcome measure in Section 3.3, will be presented.

All immunogenicity variables will be listed by treatment group, participant, and visit (Listing 7, Listing 8, Listing 9, Listing 10, Listing 11, Listing 12, Listing 13, Listing 14, and Listing 15). N, Geometric or Arithmetic Mean, Standard Deviation, Minimum and Maximum will summarize continuous immunogenicity variables, whereas number and percent will summarize categorical immunogenicity variables. Measurements that are titers or concentrations will be summarized by geometric means and 95% confidence intervals (CI). This study was not designed to test a specific null hypothesis, rather the study is designed to assess the safety and immune responses of a range of doses of dmLT when administered by the oral, SL, or ID route in participants residing in an endemic country for ETEC disease.

Immunogenicity data summaries and analysis will be presented for the mITT and PP populations.

# 8.1. Primary Immunogenicity Analysis

Not applicable.

# 8.2. Secondary Immunogenicity Analyses

Serum dmLT-specific IgA by ELISA

The number and percentage of participants showing ≥4-fold rise from the baseline in serum dmLT-specific IgA concentration determined by ELISA will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 15, 22, 29, 36, 57, 114, and any time post first dose for Oral and Sublingual Cohorts and at Days 8, 22, 29, 43, 50, 71, 128, and any time post first dose for Intradermal Cohorts (Table 43 and Table 44). Box and whisker plots of fold-rise over time will be presented (Figure 58, Figure 59, Figure 60, Figure 61, Figure 62, and Figure 63).

Serum dmLT-specific IgG by ELISA

The number and percentage of participants showing ≥4-fold rise from the baseline in serum dmLT-specific IgG concentration determined by ELISA will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 15, 22, 29, 36, 57, 114, and any time post first dose for Oral and Sublingual Cohorts and at Days 8, 22, 29, 43, 50, 71, 128, and any time post first dose for Intradermal Cohorts (Table 45 and Table 46). Box and whisker plots of fold-rise over time will be presented (Figure 64 Figure 65 Figure 66 Figure 67 Figure 68, and Figure 69).

dmLT-specific IgA ASC by ELISpot

The number and percentage of participants showing with  $\geq 8$  dmLT-specific IgA ASC /  $10^6$  PBMC as measured by ELISpot will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 1, 8, 15, 22, 29, 36, and any time for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, and any time for Intradermal Cohorts (Table 49 and Table 50).

dmLT-specific IgG ASC by ELISpot

The number and percentage of participants showing with ≥8 dmLT-specific IgG ASC / 10<sup>6</sup> PBMC as measured by ELISpot will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at

Days 1, 8, 15, 22, 29, 36, and any time for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, and any time for Intradermal Cohorts (Table 51 and Table 52).

ALS anti-dmLT-specific IgA by ELISA

The number and percentage of participants showing ≥2-fold rise from the baseline in ALS anti-dmLT-specific IgA titers determined by ELISA will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 15, 22, 29, 36, and any time post first dose for Oral and Sublingual Cohorts and at Days 8, 22, 29, 43, 50, and any time post first dose for Intradermal Cohorts (Table 53 and Table 54). Box and whisker plots of fold-rise over time will be presented (Figure 76, Figure 77, Figure 78, Figure 79, Figure 80, and Figure 81).

ALS anti-dmLT-specific IgG by ELISA

The number and percentage of participants showing ≥2-fold rise from the baseline in ALS anti-dmLT-specific IgG titers determined by ELISA will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 15, 22, 29, 36, and any time post first dose for Oral and Sublingual Cohorts and at Days 8, 22, 29, 43, 50, and any time post first dose for Intradermal Cohorts (Table 55 and Table 56). Box and whisker plots of fold-rise over time will be presented (Figure 82, Figure 83, Figure 84, Figure 85, Figure 86, and Figure 87).

Fecal dmLT-specific IgA by ELISA

The number and percentage of participants showing ≥4-fold rise from the baseline in dmLT-specific fecal IgA titers determined by ELISA will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 15, 22, 29, 36, 57, and any time post first dose for Oral and Sublingual Cohorts and at Days 8, 22, 29, 43, 50, 71, and any time post first dose for Intradermal Cohorts (Table 61, Table 62, Table 63, and Table 64). Box and whisker plots of fold-rise over time will be presented (beginning at Figure 88 and concluding with Figure 99).

Salivary dmLT-specific IgA by ELISA

The number and percentage of participants showing ≥4-fold rise from the baseline in dmLT-specific salivary IgA titers determined by ELISA will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 15, 22, 29, 36, 57, and any time post first dose for Oral and Sublingual Cohorts and at Days 8, 22, 29, 43, 50, 71, and any time post first dose for Intradermal Cohorts (Table 65, Table 66, Table 67, and Table 68). Box and whisker plots of fold-rise over time will be presented (beginning at Figure 100 and concluding with Figure 111).

# 8.3. Exploratory Immunogenicity Analyses

ALS anti-dmLT-specific IgA by ELISA

Geometric mean titers and corresponding 95% confidence intervals of dmLT-specific IgA in ALS measured by ELISA will be presented by treatment arm at Days 1, 8, 15, 22, 29, and 36 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, and 50 for Intradermal Cohorts (Table 31 and Table 32) will be presented. Box and whisker plots of log-titers over time will be presented (Figure 22, Figure 23, Figure 24, Figure 25, Figure 26, and Figure 27).

ALS anti-dmLT-specific IgG by ELISA

Geometric mean titers and corresponding 95% confidence intervals of dmLT-specific IgG in ALS measured by ELISA will be presented by treatment arm at Days 1, 8, 15, 22, 29, and 36 for Oral and Sublingual Cohorts

and at Days 1, 8, 22, 29, 43, and 50 for Intradermal Cohorts (Table 33 and Table 34) will be presented. Box and whisker plots of log-titers over time will be presented (Figure 28, Figure 29, Figure 30, Figure 31, Figure 32, and Figure 33).

## Serum dmLT-specific IgA by ELISA

Geometric mean titers and corresponding 95% confidence intervals of serum dmLT-specific IgA determined by ELISA will be presented by treatment arm at Days 1, 8, 15, 22, 29, 36, 57, and 114 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, 71, and 128 for Intradermal Cohorts (Table 21 and Table 22). Box and whisker plots of log-titers over time will be presented (Figure 4, Figure 5, Figure 6, Figure 7, Figure 8, and Figure 9).

#### Serum dmLT-specific IgG by ELISA

Geometric mean titers and corresponding 95% confidence intervals of serum dmLT-specific IgG determined by ELISA will be presented by treatment arm at Days 1, 8, 15, 22, 29, 36, 57, and 114 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, 71, and 128 for Intradermal Cohorts (Table 23 and Table 24). Box and whisker plots of log-titers over time will be presented (Figure 10, Figure 11, Figure 12, Figure 13, Figure 14, and Figure 15).

#### dmLT-specific IgA ASC by ELISpot

Mean and median number of dmLT-specific IgA ASC as measured by ELISpot will be presented by treatment arm at Days 1, 8, 15, 22, 29, and 36 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, and 50 for Intradermal Cohorts (Table 27 and Table 28).

## dmLT-specific IgG ASC by ELISpot

Mean and median number of dmLT-specific IgG ASC as measured by ELISpot will be presented by treatment arm at Days 1, 8, 15, 22, 29, and 36 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, and 50 for Intradermal Cohorts (Table 29 and Table 30).

#### Fecal dmLT-specific IgA by ELISA

Geometric mean titers and corresponding 95% confidence intervals of dmLT-specific fecal IgA determined by ELISA will be presented by treatment arm at Days 1, 8, 15, 22, 29, 36, and 57 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, and 71 for Intradermal Cohorts (Table 35, Table 36, Table 37, and Table 38). Box and whisker plots of log-titers over time will be presented (beginning at Figure 34 and concluding with Figure 45).

#### Salivary dmLT-specific IgA by ELISA

Geometric mean titers and corresponding 95% confidence intervals of dmLT-specific salivary IgA determined by ELISA will be presented by treatment arm at Days 1, 8, 15, 22, 29, 36, and 57 for Oral and Sublingual Cohorts and at Days 1, 8, 22, 29, 43, 50, and 71 for Intradermal Cohorts (Table 39, Table 40, Table 41, and Table 42). Box and whisker plots of log-titers over time will be presented (beginning at Figure 46 and concluding with Figure 57).

#### Memory B Cell dmLT-specific IgA by ELISpot

The number and percentage of participants with memory B cell dmLT-specific/total IgA response as measured by ELISpot will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 1, 22, 36, 57, 114, 209, and any time for Oral and Sublingual Cohorts and at Days 1, 29, 50, 71, 128, 223, and any time for Intradermal Cohorts (Table 69 and Table 70).

## Memory B Cell dmLT-specific IgG by ELISpot

The number and percentage of participants with memory B cell dmLT-specific/total IgG response as measured by ELISpot will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 1, 22, 36, 57, 114, 209, and any time for Oral and Sublingual Cohorts and at Days 1, 29, 50, 71, 128, 223, and any time for Intradermal Cohorts (Table 71 and Table 72).

## ASC Homing Markers IgA by EliSpot

The number and percentage of participants with anti-dmLT IgA ASC in circulation expressing gut homing receptors (integrin  $\alpha4\beta7$  in the absence or presence of CD62L) measured by EliSpot assay will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 22, 36, and any time for Oral and Sublingual Cohorts and at Days 8, 29, 50, and any time for Intradermal Cohorts (Table 57 and Table 58).

# ASC Homing Markers IgG by EliSpot

The number and percentage of participants with anti-dmLT IgG ASC in circulation expressing gut homing receptors (integrin  $\alpha4\beta7$  in the absence or presence of CD62L) measured by EliSpot assay will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 22, 36, and any time for Oral and Sublingual Cohorts and at Days 8, 29, 50, and any time for Intradermal Cohorts (Table 59 and Table 60).

## Toxin Neutralization by Y-1 cell assay

The number and percentage of participants with ≥4-fold rise over baseline in toxin neutralization titers measured by Y-1 cell assay will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 8, 15, 22, 29, 36, 57, 114, and any time post first dose for Oral and Sublingual Cohorts and at Days 8, 22, 29, 43, 50, 71, 128, and any time post first dose for Intradermal Cohorts (Table 47 and Table 48). GMTs and corresponding 95% confidence intervals will be reported (Table 25 and Table 26). Box and whisker plots of log-titers over time (Figure 16, Figure 17, Figure 18, Figure 19, Figure 20, and Figure 21) and fold-rise over time (Figure 70, Figure 71, Figure 72, Figure 73, Figure 74, and Figure 75) will be presented.

## dmLT-specific effector and memory T cell responses by CyTOF

The number and percentage of participants with dmLT-specific effector and memory T cell responses as measured by CyTOF will be presented with exact (Clopper-Pearson) two-sided 95% CI by treatment arm at Days 22, 36, 57, 114, 209, and any time post first dose for Oral and Sublingual Cohorts and at Days 29, 50, 71, 128, 223, and any time post first dose for Intradermal Cohorts (Table 73 and Table 74). Box and whisker plots of % ratio to baseline over time (beginning at Figure 112 and concluding with Figure 237) will be presented.

#### Comparison of Immunogenicity Responses

Spearman rank correlations with 95% CI for peak immunogenicity responses will be presented by Cohort (beginning at Table 75 and concluding with Table 90).

#### 9. SAFETY EVALUATION

Safety listings will be sorted by treatment group, participant, and timepoint. N, Mean, Standard Deviation, Minimum and Maximum will summarize continuous safety variables, whereas number and percent will summarize categorical safety variables. Safety data will be summarized for the Safety Analysis Population.

# 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, and race will be presented by treatment group and overall (Table 17, Table 18, Table 19, and Table 20). Ethnicity is categorized as Bengali or Other. In accordance with NIH reporting policy, participants may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the case report form (CRF) as "No" to each racial option.

Individual participant listings will be presented for all demographics (Listing 5); pre-existing medical conditions (Listing 6); vital signs and oral temperature (Listing 25); and concomitant medications (Listing 27).

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be Medical Dictionary for Regulatory Activities (MedDRA®) coded using MedDRA dictionary version 22.0 or higher. Participants' pre-existing medical conditions will be presented as individua participant listings (Listing 6).

#### 9.1.2. Prior and Concomitant Medications

Individual participant listings will be presented for all concomitant medications that were started prior to dosing and continuing at the time of dosing (Listing 27).

# 9.2. Measurements of Treatment Compliance

The number of doses of study product administered to participants will be presented by treatment group as part of the participant disposition table (Table 10 and Table 11).

Table 14 and Table 15 present the number of participants who received first dose, by treatment arm.

#### 9.3. Adverse Events

When calculating the incidence of adverse events (i.e., on a per participant basis), each participant will only be counted once and any repetitions of adverse events within a participant will be ignored; the denominator will be the total population size. All adverse events reported will be included in the summaries and analyses.

An overall summary of adverse events by treatment group is presented in Table 91 and Table 92. Unsolicited adverse events occurring in more than 5% of participants in any treatment group are presented in Table 93 and Table 94.

## 9.3.1. Solicited Events and Symptoms

Solicited adverse events were collected pre-vaccination, 90 minutes post-vaccination following oral dosing or 30 minutes post-vaccination following SL and ID dosing, and then daily for 7 days after each vaccination and graded on a scale of 0 (none), 1 (mild), 2 (moderate) and 3 (severe). Grading scales for solicited adverse events are presented in Table 7. Systemic events for the oral and sublingual routes include: fever, feverishness, fatigue, malaise, myalgia, or headache. Systemic events for the intradermal route include: fever,

feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local events for the oral route include: irritation of the oral cavity or tongue, diarrhea, nausea, vomiting, and abdominal discomfort. Local events for the sublingual route include: irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort. Local events for the intradermal route include: injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.

The proportion of participants reporting at least one solicited adverse event will be summarized for each solicited adverse event, any systemic symptom, any local symptom, and any symptoms. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (beginning at Table 97 and concluding with Table 104).

For each systemic and local event, any systemic event, any local event, and any solicited event, the maximum severity over 7 days after each vaccination will be summarized for the Safety population. The number and percentage of participants reporting each event will be summarized by the maximum severity and treatment group, separately for each vaccination and over all vaccinations. For each event the denominator is the number of participants with non-missing data for the specific event (beginning at Table 105 and concluding with Table 112).

The number of participants reporting a solicited adverse event will be summarized for each day post vaccination for each vaccination and for all vaccinations combined both in a summary table (beginning at Table 113 and concluding with Table 134) and graphically in a bar chart (beginning at Figure 238 and concluding with Figure 253). A comparison of the event rate for each treatment group between vaccination 1 and vaccination 2, vaccination 2 and vaccination 3, and vaccination 1 and vaccination 3 will be presented (Table 135, Table 136, and Table 137).

Solicited adverse events by participant will be presented in Listing 16, Listing 17, Listing 18, Listing 19, Listing 20, and Listing 21.

#### 9.3.2. Unsolicited Adverse Events

The proportion of participants reporting at least one unsolicited adverse event will be summarized by MedDRA system organ class and preferred term and treatment group for each vaccination and over all vaccinations. Denominators for percentages are the number of participants who received the vaccination being summarized.

Unsolicited adverse events by participant will be presented in Listing 22.

The following summaries for unsolicited adverse events will be presented by MedDRA system organ class, preferred term, vaccination and treatment group:

• Participant listing of non-serious adverse events of moderate or greater severity (Table 139);

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Participant ID, Adverse Event Description, Last Dose Received/Days Post Dose, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

• Deaths and Serious Adverse Events (Table 138);

# 9.5. Pregnancies

For any participants in the Safety population who became pregnant during the study, every attempt was made to follow the participants to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. Listings of pregnancies and outcomes will be presented (Listing 28, Listing 29, Listing 30, Listing 31, and Listing 32).

## 9.6. Clinical Laboratory Evaluations

The baseline value will be defined as the last value obtained prior to the first vaccination/dose of study product. If a participant has repeated laboratory values on the same day, the value from the last evaluation will be used for analysis. Post-baseline, in the case of multiple observations (for example, from supplemental visits), the assessment value that is closest to the scheduled visit window will be used in the analyses. All the recorded data will be listed. If observations have the same distance to the scheduled assessment, the latest one will be used.

Chemistry parameters evaluated were creatinine, ALT, Albumin, and Total Bilirubin. Hematology parameters evaluated were WBC, ANC, hemoglobin, and platelets.

All clinical laboratory parameters were evaluated at baseline (screening visit) and Day 57 for Oral and Sublingual Cohorts and at baseline (screening visit) and Day 71 for Intradermal Cohorts. ALT creatinine, and total bilirubin were also evaluated at Day 36 for Oral and Sublingual Cohorts and at Day 50 for Intradermal Cohorts. The distribution of laboratory results by severity, time point, and treatment group will be presented in Table 142, Table 143, Table 144, Table 145, and Table 146 for chemistry and in Table 151, Table 152, Table 153, Table 154, and Table 155 for hematology. Descriptive statistics including mean, standard deviation, median, minimum and maximum values and changes from baseline by time point, for each laboratory parameter, will be summarized in Table 147, Table 148, Table 149, and Table 150 for chemistry and in Table 156, Table 157, Table 158, and Table 159 for hematology. Changes in laboratory values will be presented beginning at Figure 254 and concluding with Figure 276.

Grading scales for safety laboratory parameters are presented in Table 8.

Listing 23 and Listing 24 will provide a complete listing of individual clinical laboratory results with applicable reference ranges. Table 140 and Table 141 will provide a listing of only abnormal individual clinical laboratory results.

# 9.7. Vital Signs and Physical Evaluations

The baseline value will be defined as the last value obtained prior to the first vaccination/dose of study product. If a participant has repeated vital sign measurements on the same day, the value from the last evaluation will be used for analysis. Post-baseline, in the case of multiple observations (for example, from supplemental visits), the assessment value that is closest to the scheduled visit window will be used in the analyses. All the recorded data will be listed. If observations have the same distance to the scheduled assessment, the latest one will be used.

Vital sign measurements include systolic blood pressure, diastolic blood pressure, pulse, and oral temperature. Grading scales for vital signs are presented in Table 9. Vital signs were assessed at Day 1, Day 8, Day 15, Day 22, Day 29, Day 36, Day 57, Day 114 and Day 209 for Oral and Sublingual Cohorts and at Day 1, Day 8, Day 22, and Day 29 for Intradermal Cohorts. Vital signs will be tabulated by severity, visit, and treatment group (Table 160, Table 161, Table 162, Table 163, and Table 164; Listing 25).

Physical Examinations were performed at screening to assess general wellness. The following body systems were assessed: head, eyes, ears, nose, and throat; lymph nodes; skin; pulmonary; cardiovascular; abdominal; neurological; and musculoskeletal systems. At subsequent visits including enrollment a targeted physical examination was conducted if indicated based on review of medical history. Findings will be presented in Listing 26.

#### 9.8. Concomitant Medications

Concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study was recorded on the CRFs. A by-participant listing of concomitant medication use will be presented (Listing 27).

# 9.9. Other Safety Measures

Not applicable.

# 10. PHARMACOKINETICS

Not applicable.

# 11. IMMUNOGENICITY

See Section 8.
# 12. OTHER ANALYSES

Not applicable.

### 13. REPORTING CONVENTIONS

The mean, standard deviation, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%.

# 14. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

### **Changes to Study Conduct**

- At the request of the local (icddr,b) DSMB, collection of serum bilirubin at screening and Visit 6 and collection of ALT and creatinine at Visit 6 were added to the safety labs. These results were not obtained for Cohorts A through C which were enrolled prior to the request.
- Due to a country-wide lockdown instituted in Bangladesh to combat the COVID-19 pandemic all Cohort E participants did not receive a third dose of study product. Cohort D participant Visits 8 and 9 and Cohort E participant Visits 6 through 9 were not conducted and no further cohorts were enrolled due to the pandemic.

#### 16. REFERENCES

- 1. El-Kamary SS, Cohen MB, Bourgeois AL, et al. Safety and immunogenicity of a single oral dose of recombinant double mutant heat-labile toxin derived from enterotoxigenic Escherichia coli. Clin Vaccine Immunol 2013;20:1764-70.
- 2. Lundgren A, Bourgeois L, Carlin N, et al. Safety and immunogenicity of an improved oral inactivated multivalent enterotoxigenic Escherichia coli (ETEC) vaccine administered alone and together with dmLT adjuvant in a double-blind, randomized, placebo-controlled Phase I study. Vaccine 2014;32:7077-84.
- 3. Harro C, Sack DA, Chakraborty S, et al. Evaluation of a Lyophilized Formulation of Enterotoxigenic Escherichia coli (ETEC) ACE527 Vaccine Administered Alone or With a Double-Mutant E. coli Heat-Labile Toxin (dmLT) in Healthy Adult Subjects (NCT01739231). In: The Seventh International Conference on: Vaccines for Enteric Diseases. Bangkok, Thailand; 2013.
- 4. Bernstein, D., M. Pasetti, R. Brady, et al. A Phase 1 dose escalating study of double mutant heat-labile toxin LTR192G/L211A (dmLT) from Enterotoxigenic *Escherichia coli* (ETEC) by sublingual or oral immunization. Vaccine. <a href="https://doi.org/10.1016/j.vaccine.2018.12.011">https://doi.org/10.1016/j.vaccine.2018.12.011</a>
- 5. Drummond R. CONSORT Revised: Improving the Reporting of Randomized Clinical Trials. JAMA. 2001; 285(15):2006-2007.

# 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

# **APPENDICES**

# APPENDIX 1. TABLE MOCK-UPS

# LIST OF TABLES

| Table 1: | Study Design | 46 |
|---|---|---|
| Table 2: | Schedule of Study Procedures – Oral & Sublingual Cohorts | 47 |
| Table 3: | Schedule of Study Procedures – Intradermal Cohort | 49 |
| Table 4: | Sample Size/Probability Estimates | 51 |
| Table 5: | Distribution of Protocol Deviations by Category, Type, and Treatment<br>Group – Oral & Sublingual Cohorts | 52 |
| Table 6: | Distribution of Protocol Deviations by Category, Type, and Treatment<br>Group – Intradermal & Pooled Cohorts | 54 |
| Table 7: | Solicited Adverse Event Grading Scale | 55 |
| Table 8: | Laboratory Adverse Event Grading Scale | 56 |
| Table 9: | Vital Sign Adverse Event Grading Scale | 57 |
| Table 10: | Subject Disposition by Treatment Group - Oral & Sublingual Cohorts | 58 |
| Table 11: | Subject Disposition by Treatment Group - Intradermal & Pooled Cohorts | 58 |
| Table 12: | Analysis Populations by Treatment Group – Oral & Sublingual Cohorts | 59 |
| Table 13: | Analysis Populations by Treatment Group – Intradermal & Pooled Cohorts | 59 |
| Table 14: | Dates of First Treatment by Treatment Group - Oral & Sublingual Cohorts | 60 |
| Table 15: | Dates of First Treatment by Treatment Group – Intradermal & Pooled Cohorts | 60 |
| Table 16: | Ineligibility Summary of Screen Failures | 61 |
| Table 17: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - Oral & Sublingual Cohorts | 62 |
| Table 18: | Summary of Categorical Demographic and Baseline Characteristics by Treatment Group – Intradermal & Pooled Cohorts | 62 |
| Table 19: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group – Oral & Sublingual Cohorts | 63 |
| Table 20: | Summary of Continuous Demographic and Baseline Characteristics by Treatment Group – Intradermal & Pooled Cohorts | 63 |
| Table 21: | Serum IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population | 64 |
| Table 22: | Serum IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 65 |
| Table 23: | Serum IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population | 66 |

| Table 24: | Serum IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 67 |
|---|---|---|
| Table 25: | Serum LT Toxin Neutralization GMT Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, mITT Population | 68 |
| Table 26: | Serum LT Toxin Neutralization GMT Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, Per Protocol Population | 69 |
| Table 27: | ASC IgA Results by Time Point and Treatment Group, mITT Population | 70 |
| Table 28: | ASC IgA Results by Time Point and Treatment Group, Per Protocol Population | 71 |
| Table 29: | ASC IgG Results by Time Point and Treatment Group, mITT Population | 72 |
| Table 30: | ASC IgG Results by Time Point and Treatment Group, Per Protocol Population | 73 |
| Table 31: | ALS IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population | 74 |
| Table 32: | ALS IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 75 |
| Table 33: | ALS IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population | 76 |
| Table 34: | ALS IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 77 |
| Table 35: | Fecal dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population | 78 |
| Table 36: | Fecal dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 79 |
| Table 37: | Fecal dmLT-specific/Total IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population | 80 |
| Table 38: | Fecal dmLT-specific/Total IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 81 |
| Table 39: | Salivary dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population | 82 |
| Table 40: | Salivary dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 83 |
| Table 41: | Salivary dmLT-specific/Total IgA GMT Results with 95% Confidence<br>Intervals by Time Point and Treatment Group, mITT Population | 84 |
| Table 42: | Salivary dmLT-specific/Total IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population | 85 |
| Table 43: | Serum IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population | 86 |

| Table 44: | Serum IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 88 |
|---|---|---|
| Table 45: | Serum IgG GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population | 89 |
| Table 46: | Serum IgG GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 91 |
| Table 47: | Serum LT Toxin Neutralization GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population | 92 |
| Table 48: | Serum LT Toxin Neutralization GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 94 |
| Table 49: | ASC IgA Response Results by Time Point and Treatment Group, mITT Population | 95 |
| Table 50: | ASC IgA Response Results by Time Point and Treatment Group, Oral & Sublingual Cohorts, Per Protocol Population | 96 |
| Table 51: | ASC IgG Response Results by Time Point and Treatment Group, mITT Population | 97 |
| Table 52: | ASC IgG Response Results by Time Point and Treatment Group, Per Protocol Population | 98 |
| Table 53: | ALS IgA GMFR and 2-Fold Rise Results by Time Point and Treatment Group, mITT Population | 99 |
| Table 54: | ALS IgA GMFR and 2-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 100 |
| Table 55: | ALS IgG GMFR and 2-Fold Rise Results by Time Point and Treatment Group, mITT Population | 101 |
| Table 56: | ALS IgG GMFR and 2-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 102 |
| Table 57: | ASC Homing Markers IgA by Time Point and Treatment Group, mITT Population | |
| Table 58: | ASC Homing Markers IgA by Time Point and Treatment Group, Per Protocol Population | |
| Table 59: | ASC Homing Markers IgG by Time Point and Treatment Group, mITT Population | |
| Table 60: | ASC Homing Markers IgG by Time Point and Treatment Group, Per Protocol Population | |
| Table 61: | Fecal dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population | |
| Table 62: | Fecal dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | |

| Table 63: | Fecal dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population | 109 |
|---|---|---|
| Table 64: | Fecal dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 110 |
| Table 65: | Salivary dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population | 111 |
| Table 66: | Salivary dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 112 |
| Table 67: | Salivary dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population | 113 |
| Table 68: | Salivary dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population | 114 |
| Table 69: | Anti-dmLT IgA Memory B Cell Response – mITT Population | 115 |
| Table 70: | Anti-dmLT IgA Memory B Cell Response – Per Protocol Population | 117 |
| Table 71: | Anti-dmLT IgG Memory B Cell Response – mITT Population | 118 |
| Table 72: | Anti-dmLT IgG Memory B Cell Response – Per Protocol Population | 120 |
| Table 73: | T Cell Memory Responses by CyTOF – mITT Population | 121 |
| Table 74: | T Cell Memory Responses by CyTOF – Per Protocol Population | 180 |
| Table 75: | Correlation of Serum IgA GMFR vs Fecal dmLT-specific IgA GMFR by Time Point and Treatment Group, Immunogenicity Population | 181 |
| Table 76: | Correlation of Serum IgA GMFR vs Fecal dmLT-specific IgA GMFR by Time Point and Treatment Group, Per Protocol Population | 181 |
| Table 77: | Correlation of Serum IgA GMFR vs Fecal dmLT-specific/Total IgA GMFR by Time Point and Treatment Group, Immunogenicity Population | 181 |
| Table 78: | Correlation of Serum IgA GMFR vs Fecal dmLT-specific/Total IgA GMFR by Time Point and Treatment Group, Per Protocol Population | 181 |
| Table 79: | Correlation of Serum IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population | 182 |
| Table 80: | Correlation of Serum IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population | 182 |
| Table 81: | Correlation of Serum IgG GMFR vs ALS IgG Titers GMFR by Time Point and Treatment Group, Immunogenicity Population | 183 |
| Table 82: | Correlation of Serum IgG GMFR vs ALS IgG Titers GMFR by Time Point and Treatment Group, Per Protocol Population | 183 |
| Table 83: | Correlation of Fecal dmLT-specific IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population | 184 |
| Table 84: | Correlation of Fecal dmLT-specific IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population | 184 |

| Table 85: | Correlation of Fecal dmLT-specific/Total IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population | 185 |
|---|---|---|
| Table 86: | Correlation of Fecal dmLT-specific/Total IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population | 185 |
| Table 87: | Correlation of ASC IgA Count vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population | 186 |
| Table 88: | Correlation of ASC IgA Count vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population | 186 |
| Table 89: | Correlation of ASC IgG Count vs ALS IgG Titers GMFR by Time Point and Treatment Group, Immunogenicity Population | 187 |
| Table 90: | Correlation of ASC IgG Count vs ALS IgG Titers GMFR by Time Point and Treatment Group, Per Protocol Population | 187 |
| Table 91: | Overall Summary of Adverse Events - Oral & Sublingual Cohorts | 188 |
| Table 92: | Overall Summary of Adverse Events - Intradermal & Pooled Cohorts | 189 |
| Table 93: | Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Oral & Sublingual Cohorts | 190 |
| Table 94: | Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Intradermal & Pooled Cohorts | 190 |
| Table 95: | Serious Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Oral & Sublingual Cohorts | 190 |
| Table 96: | Serious Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Intradermal & Pooled Cohorts | 190 |
| Table 97: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort A: Oral 5 µg dmLT | 191 |
| Table 98: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort B: Oral 25 µg dmLT | 191 |
| Table 99: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – All Oral Cohorts: Placebo | 191 |
| Table 100: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort C: Sublingual 5 µg dmLT | 192 |
| Table 101: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort D: Sublingual 25 µg dmLT | 192 |

| Table 102: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – All Sublingual Cohorts: Placebo | 192 |
|---|---|---|
| Table 103: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort E: Intradermal 0.3 µg dmLT | 192 |
| Table 104: | Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort E: Intradermal Placebo | 192 |
| Table 105: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort A: Oral 5 µg dmLT | 193 |
| Table 106: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort B: Oral 25 µg dmLT | 195 |
| Table 107: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – All Oral Cohorts: Placebo | 195 |
| Table 108: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort C: Sublingual 5 µg dmLT | 195 |
| Table 109: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort D: Sublingual 25 µg dmLT | 195 |
| Table 110: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – All Sublingual Cohorts: Placebo | 196 |
| Table 111: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort E: Intradermal 0.3 µg dmLT | 196 |
| Table 112: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort E: Intradermal Placebo | 196 |
| Table 113: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort A: Oral 5 µg dmLT, Dose 1 | 197 |
| Table 114: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort A: Oral 5 µg dmLT, Dose 2 | 200 |
| Table 115: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort A: Oral 5 µg dmLT, Dose 3 | 200 |
| Table 116: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort B: Oral 25 µg dmLT, Dose 1 | 200 |
| Table 117: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort B: Oral 25 µg dmLT, Dose 2 | 200 |

| Table 118: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort B: Oral 25 µg dmLT, Dose 3 | 200 |
|---|---|---|
| Table 119: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Oral Cohorts: Placebo, Dose 1 | 200 |
| Table 120: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Oral Cohorts: Placebo, Dose 2 | 200 |
| Table 121: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Oral Cohorts: Placebo, Dose 3 | 200 |
| Table 122: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort C: Sublingual 5 µg dmLT, Dose 1 | 200 |
| Table 123: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort C: Sublingual 5 µg dmLT, Dose 2 | 201 |
| Table 124: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort C: Sublingual 5 µg dmLT, Dose 3 | 201 |
| Table 125: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort D: Sublingual 25 µg dmLT, Dose 1 | 201 |
| Table 126: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort D: Sublingual 25 µg dmLT, Dose 2 | 201 |
| Table 127: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort D: Sublingual 25 µg dmLT, Dose 3 | 201 |
| Table 128: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Sublingual Cohorts: Placebo Dose 1 | 201 |
| Table 129: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Sublingual Cohorts: Placebo, Dose 2 | 201 |
| Table 130: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Sublingual Cohorts: Placebo, Dose 3 | |

| Table 131: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal 0.3 µg dmLT, Dose 1 | 202 |
|---|---|---|
| Table 132: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal 0.3 µg dmLT, Dose 2 | 202 |
| Table 133: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal Placebo, Dose 1 | 202 |
| Table 134: | Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal Placebo, Dose 2 | 202 |
| Table 135: | Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 2 by Treatment Group | 203 |
| Table 136: | Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 3 by Treatment Group | 205 |
| Table 137: | Number and Percentage of Subjects Experiencing Solicited Events for Dose 2 Compared with Dose 3 by Treatment Group | 205 |
| Table 138: | Listing of Serious Adverse Events | 206 |
| | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | |
| Table 140: | Listing of Abnormal Laboratory Results - Chemistry | 209 |
| | Listing of Abnormal Laboratory Results - Hematology | |
| Table 142: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter | 211 |
| Table 143: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Creatinine | 212 |
| Table 144: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Alanine Aminotransferase | 213 |
| Table 145: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Albumin | 214 |
| Table 146: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Total Bilirubin | 215 |
| Table 147: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Creatinine (µmol/L) | 216 |
| Table 148: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Alanine Aminotransferase (U/L) | 217 |
| Table 149: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Albumin (g/dL) | |

| Table 150: | $Laboratory\ Summary\ Statistics\ by\ Parameter,\ Time\ Point,\ and\ Treatment$ $Group-Total\ Bilirubin\ (\mu mol/L)\$ | 219 |
|---|---|---|
| Table 151: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter | 220 |
| Table 152: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cell Count | 221 |
| Table 153: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Absolute Neutrophil Count | 222 |
| Table 154: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Hemoglobin | 223 |
| Table 155: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelets | 224 |
| Table 156: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – White Blood Cell Count (10 <sup>9</sup> /L) | 225 |
| Table 157: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Absolute Neutrophil Count (10 <sup>9</sup> /L) | 226 |
| Table 158: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Hemoglobin (mg/dL) | 227 |
| Table 159: | Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Platelets (10 <sup>9</sup> /L) | 228 |
| Table 160: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Any Assessment | 229 |
| Table 161: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Temperature | 232 |
| Table 162: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Pulse | 235 |
| Table 163: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Systolic Blood Pressure | 239 |
| Table 164: | Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Diastolic Blood Pressure | 243 |

#### **Overall Study Design and Plan Description** 9.1

Table 1: **Study Design** 

| Cohort | Group | Route | dmLT dose<br>(μg) | Target No.<br>Participant<br>Enrollment | Minimum No.<br>Participants<br>Evaluable* | Vaccination Days |
|---|---|---|---|---|---|---|
| A | A1<br>A2 | Oral | 5<br>placebo | 12<br>3 | 10<br>1 | 1, 15, 29 |
| ISM, MM, and the protoc | col PI will rev | | data collected thro | | ination of third dose | of last participant for |
| В | B1<br>B2 | Oral | 25<br>placebo | 12<br>3 | 10<br>1 | 1, 15, 29 |
| С | C1<br>C2 | Sublingual | 5<br>placebo | 12<br>3 | 10<br>1 | 1, 15, 29 |
| ISM, MM, and the pr | rotocol PI wi | ll review Cohort C sat | fety data collected<br>lation to proceed t | | on of third dose of la | st participant for |
| D | D1<br>D2 | Sublingual | 25<br>placebo | 12<br>3 | 10<br>1 | 1, 15, 29 |
| Eª | E1<br>E2 | Intradermal | 0.3<br>placebo | 12<br>3 | 10<br>1 | 1, 22, 43 |
| ISM, MM, and the protoc | col PI will re | | data collected thro<br>dation to proceed t | | ination of third dose | of last participant for |
| F <sup>b</sup> | F1<br>F2 | Intradermal | 1.0<br>placebo | 12<br>3 | 10<br>1 | 1, 22, 43 |
| Scheduled DMID DSMB | meeting will | | ulative safety data<br>d proceed to Coho | | the third dose of vac | cine and determine if |
| $G_p$ | G1<br>G2 | Oral | 50<br>placebo | 12<br>3 | 10<br>1 | 1, 15, 29 |
| $H_p$ | H1<br>H2 | Sublingual | 50<br>placebo | 12<br>3 | 10<br>1 | 1, 15, 29 |
| $I_p$ | I1<br>I2 | Intradermal | 2.0<br>placebo | 12<br>3 | 10<br>1 | 1, 22, 43 |
| Scheduled DMID DSMB | meeting will | be held to review the | aggregate safety o | data through 28 days | after the third dose o | f vaccine for all nine |

A Final DMID DSMB meeting will be held to review the safety data following the completion of the study

cohorts (A-I)b

a Halted prior to Dose 3 because of COVID-19 Pandemic b Not done due to COVID-19 Pandemic

# 9.5.1 Immunogenicity and Safety Measurements Assessed and Flow Chart

 Table 2:
 Schedule of Study Procedures – Oral & Sublingual Cohorts

| | | | | Oral and | d Subling | ual coho | rts | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit (V) | screen | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | |
| Study Day | -7 to -4 | 1 | 8 | 15 | 22 | 29 | 36 | 57 | 114 | 209 | Unscheduled visit, upo | Early Tamain ation 10 |
| Window | | | ±1d | ±2d | ±1d | ±2d | ±1d | ±3d | ±1w | ±2w | investigator judgement | Early Termination <sup>10</sup> |
| Study Week | | 0 | 1 | 2 | 3 | 4 | 5 | 8 | 16 | 30 | | |
| Informed Consent | X | | | | | | | | | | | |
| Confirm Ongoing Consent | | X | X | X | X | X | X | X | X | X | | |
| Eligibility Review | X | X | X | X | X | X | X | X | X | | | |
| Collection of demographics | X | | | | | | | | | | | |
| Medical History | X | X | X | X | X | X | X | X | X | X | X | [X] |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | [X] |
| Physical Exam | X | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | | X | [X] |
| Vitals Signs | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | X | [X] |
| Urine pregnancy test <sup>4,9</sup> | X | X | | X | | X | | | | | | |
| VACCINATION | | #1 | | #2 | | #3 | | | | | | |
| Pre-vaccination & Post-vaccination assessment | | X <sup>5</sup> | | X <sup>5</sup> | | X <sup>5</sup> | | | | | | |
| Memory Aid and thermometer (d)distribute, (c) collect Memory Aid | | d | С | d | С | D | с | | | | | [c] <sup>7</sup> |
| Confirm date & time of next Visit | | X | X | X | X | X | X | X | X | | | |
| Adverse Event (AE)/Serious AE review | | X | $X^6$ | X | $X^6$ | X | $X^6$ | $X^6$ | X <sup>1</sup> | $X^1$ | X <sup>8</sup> | X |
| Screening stool | X | | | | | | | | | | | |
| Saliva/Oral Fluid for Ab | | X | X | X | X | X | X | X | | | Also may occur: | |
| Stool for ELISA Ab | | X | X | X | X | X | X | X | | | Stool culture when | |
| Stool for future use (Microbiome studies) | X | X | X | X | X | X | X | X | | | indicated; Exam and Photo of | |
| Clinical labs/chemistry | 2 mL | | | | | | 2 mL | 2 mL | | | local reactogenicity | |
| Blood-Serum for ELISA Ab & Neut. | | 3 mL | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | 3 mL | 2 mL | | when indicated | |

| Oral and Sublingual cohorts | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Blood-PBMC for ASC | | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | | | | | |
| Blood-PBMC for ASC w/ homing | | | 2 mL | | 2 mL | | 2 mL | | | | I | |
| Blood-PBMC for ALS | | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | | | | I | |
| Blood-PBMC for Memory B assays | | 8mL | | | 5 mL | | 5 mL | 5 mL | 5 mL | 5 mL | I | Ī |
| Blood-PBMC for effector T cell assays | 13 mL | | | | 8mL | | 7 mL | 7 mL | 8 mL | 10 mL | I | Ī |
| Store plasma from PBMC | | X | X | | X | | X | X | X | X | I | |
| Total Blood Volume up to ~140 mL/participant | 15 mL | 15 mL | 8 mL | 6 mL | 21 mL | 6 mL | 22 mL | 17 mL | 15 mL | 15 mL | | Ī |

<sup>[]</sup> Make every effort to collect at Early Termination visit. If not collected, this will not result in a protocol deviation.

<sup>&</sup>lt;sup>1</sup>review for Serious Adverse Events only

<sup>&</sup>lt;sup>2</sup>Targeted physical examination, if indicated based on review of medical history

<sup>&</sup>lt;sup>3</sup>Vital signs: collect oral temperature, pulse, and blood pressure

<sup>&</sup>lt;sup>4</sup>Urine pregnancy test required for all women

<sup>&</sup>lt;sup>5</sup>Exam at end of 30 min observation period post-vaccination for SL and ID, at end of a 90 min observation period for Oral

<sup>&</sup>lt;sup>6</sup>Review to include assessments of: 1) injection site necrosis within 7 days of vaccination, 2) urticaria, laryngospasm, bronchospasm, or anaphylaxis determined to be related to vaccine and within 7 days of vaccination, 3) facial nerve neuropathy, confirmed by an investigator and determined to be related to vaccine.

<sup>&</sup>lt;sup>7</sup>Assess reactogenicity and review memory aid if early termination occurs within 7 days of any vaccination

<sup>&</sup>lt;sup>8</sup> AE assessment to include (as applicable): 1) Assess reactogenicity (if within 7 days of last vaccination), unsolicited non-serious AE information (if within 28 days of last vaccination), or any SAE information (anytime within study) 2) Upon judgement of the clinical investigator, clinical laboratory assessments may be performed to evaluate an AE and medications (e.g. analgesics) may be recommended to treat an AE.

<sup>&</sup>lt;sup>9</sup>Visits 1-7: Provide instructions to women participants to avoid pregnancy through the 28 days from receipt of the last dose of vaccine.

<sup>&</sup>lt;sup>10</sup>Early Termination Visit is to include: assess reactogenicity and review memory aid if early termination occurs within 7 days of any vaccination; assess for SAE during all early termination visits; obtain serum samples for laboratory safety assays if visit occurs <28 days after third vaccination.

 Table 3:
 Schedule of Study Procedures – Intradermal Cohort

| Intradermal Cohort Study Visit (V) screen 1 2 3 4 5 6 7 8 9 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit (V) | screen | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | | |
| Study Day | -7 to -4 | 1 | 8 | 22 | 29 | 43 | 50 | 71 | 128 | 223 | Unscheduled visit, upon | |
| Window | | | ±1d | ±2d | ±1d | ±2d | ±1d | ±3d | ±1w | ±2w | investigator judgement | Early Termination <sup>11</sup> |
| Study Week | | 0 | 1 | 3 | 4 | 6 | 7 | 10 | 18 | 32 | | |
| Informed Consent | X | | | | | | | | | | | |
| Confirm Ongoing Consent | | X | X | X | X | X | X | X | X | X | | |
| Eligibility Review | X | X | X | X | X | X | X | X | X | | | |
| Collection of demographics | X | | | | | | | | | | | |
| Medical History | X | X | X | X | X | X | X | X | X | X | X | [X] |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | [X] |
| Physical Exam | X | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ | | X | [X] |
| Vitals Signs | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | $X^3$ | X | [X] |
| Urine pregnancy test <sup>4,10</sup> | X | X | | X | | X | | | | | | |
| VACCINATION | | #1 | | #2 | | #3 | | | | | | |
| Pre-vaccination & Post-vaccination assessment | | X <sup>6</sup> | | $X^6$ | | X <sup>6</sup> | | | | | | |
| Memory Aid and thermometer (d)distribute, (c) collect Memory Aid | | d | с | d | с | d | с | | | | | [c] <sup>8</sup> |
| Confirm date & time of next Visit | | X | X | X | X | X | X | X | X | | | |
| Adverse Event (AE) / Serious AE review | | X | X <sup>5,7</sup> | X | X <sup>5,7</sup> | X | X <sup>5,7</sup> | X <sup>7</sup> | X <sup>1</sup> | $X^1$ | X <sup>5,9</sup> | X |
| Screening stool | X | | | | | | | | | | | |
| Saliva/Oral Fluid for Ab | | X | X | X | X | X | X | X | | | Also may occur: | |
| Stool for ELISA Ab | | X | X | X | X | X | X | X | | | Stool culture when | |
| Stool for future use (Microbiome studies) | X | X | X | X | X | X | X | X | | | indicated;<br>Exam and Photo of | |
| Clinical labs/chemistry | 2 mL | | | | | | 2 mL | 2 mL | | | local reactogenicity | |
| Blood-Serum for ELISA Ab & Neut. | | 3 mL | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | 3 mL | 2 mL | | when indicated | |

| | Intradermal Cohort | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Blood-PBMC for ASC | | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | | | |
| Blood-PBMC for ASC w/ homing | | | 2 mL | | 2 mL | | 2 mL | | | |
| Blood-PBMC for ALS | | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | 2 mL | | | |
| Blood-PBMC for Memory B assays | | 8mL | | | 5 mL | | 5 mL | 5 mL | 5 mL | 5 mL |
| Blood-PBMC for effector T cell assays | 13 mL | | | | 8 mL | | 7 mL | 7 mL | 8 mL | 10 mL |
| Store plasma from PBMC | | X | X | | X | | X | X | X | X |
| Total Blood Volume up to ~140 mL/participant | 15 mL | 15 mL | 8 mL | 6 mL | 21 mL | 6 mL | 22 mL | 17 mL | 15 mL | 15 mL |

Make every effort to collect at Early Termination visit. If not collected, this will not result in a protocol deviation.

<sup>&</sup>lt;sup>1</sup>review for Serious Adverse Events only

<sup>&</sup>lt;sup>2</sup>Targeted physical examination, if indicated based on review of medical history

<sup>&</sup>lt;sup>3</sup>Vital signs: collect oral temperature, pulse, and blood pressure

<sup>&</sup>lt;sup>4</sup>Urine pregnancy test required for all women

<sup>&</sup>lt;sup>5</sup>For grade 3 local site reactions, a photo should be taken on a daily basis until the injection site reaction is deemed stable or returns back to a grade 2 or lower severity, if the event occurs within 7 days of an intradermal dose administration

<sup>&</sup>lt;sup>6</sup>Exam at end of 30 min observation period post-vaccination

<sup>&</sup>lt;sup>7</sup>Review to include assessments of: 1) injection site necrosis within 7 days of vaccination, 2) urticaria, laryngospasm, bronchospasm, or anaphylaxis determined to be related to vaccine and within 7 days of vaccination, 3) facial nerve neuropathy, confirmed by an investigator and determined to be related to vaccine.

<sup>&</sup>lt;sup>8</sup> Assess reactogenicity and review memory aid if early termination occurs within 7 days of any vaccination

<sup>&</sup>lt;sup>9</sup>AE assessment to include (as applicable): 1) Assess reactogenicity (if within 7 days of last vaccination), unsolicited non-serious AE information (if within 28 days of last vaccination), or any SAE information (anytime within study) 2) Upon judgement of the clinical investigator, clinical laboratory assessments may be performed to evaluate an AE and medications (e.g. analgesics) may be recommended to treat an AE.

<sup>&</sup>lt;sup>10</sup>Visits 1-7: Provide instructions to women participants to avoid pregnancy through the 28 days from receipt of the last dose of vaccine.

<sup>&</sup>lt;sup>11</sup>Early Termination Visit is to include: assess reactogenicity and review memory aid if early termination occurs within 7 days of any vaccination; assess for SAE during all early termination visits; obtain serum samples for laboratory safety assays if visit occurs <28 days after third vaccination.

# 9.7.1 Sample Size

Table 4: Sample Size/Probability Estimates

| | Evaluable Vaccinees (N) | Upper 95% Confidence Bound in the Absence of Observed Dose-Limiting AE |
|---|---|---|
| Per Cohort | 10 | 30.8% |
| Per Route <sup>a</sup> | 20 | 16.8% |
| Cohorts A-D <sup>b</sup> | 40 | 8.8% |
| Cohorts A-F <sup>c</sup> | 60 | 6.0% |

<sup>&</sup>lt;sup>a</sup>Oral, sublingual or intradermal <sup>b</sup>Received all three doses

<sup>&</sup>lt;sup>c</sup>Planned prior to safety data review

### 10.2 Protocol Deviations

Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group – Oral & Sublingual Cohorts

| | | | ort A:<br>.g dmLT<br>=X) | Oral<br>dm | ort B:<br>25 μg<br>LT<br>=X) | Coh<br>Plac | Oral<br>orts:<br>cebo<br>=X) | Sub | ll Route<br>jects<br>=X) | Subling<br>dm | ort C:<br>ual 5 µg<br>iLT<br>=X) | Sublingt<br>dm | ort D:<br>nal 25 μg<br>LT<br>=X) | Coh<br>Plac | olingual<br>orts:<br>cebo<br>=X) | Route S | olingual<br>Subjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. |
| Eligibility/<br>enrollment | Any type | | | | | | | | | | | | | | | | |
| | Did not meet inclusion criterion | х | X | X | X | X | X | X | X | X | X | X | X | X | X | х | Х |
| | Met exclusion criterion | | | | | | | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | | | |
| Treatment administration schedule | Any type | | | | | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | | | | | |
| | Missed treatment administration | | | | | | | | | | | | | | | | |
| | Delayed treatment administration | | | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | | | |

Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group (continued)

| | | Coho<br>Oral 5 µ<br>(N= | g dmLT | Oral<br>dm | ort B:<br>25 μg<br>LT<br>=X) | Coh<br>Plac | Oral<br>orts:<br>cebo<br>=X) | Sub | ll Route<br>jects<br>=X) | | | dm | ort D:<br>nal 25 μg<br>LLT<br>=X) | Coh<br>Plac | olingual<br>orts:<br>cebo<br>=X) | Route S | blingual<br>Subjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. |
| Protocol<br>procedure/<br>assessment | Any type | | | | | | | | | | | | | | | | |
| | Incorrect version of ICF signed | | | | | | | | | | | | | | | | |
| | Blood not collected | | | | | | | | | | | | | | | | |
| | Urine not collected | | | | | | | | | | | | | | | | |
| | Stool not collected | | | | | | | | | | | | | | | | |
| | Other specimen not collected | | | | | | | | | | | | | | | | |
| | Too few aliquots obtained | | | | | | | | | | | | | | | | |
| | Specimen result not obtained | | | | | | | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | | | | | |
| | Study product temperature excursion | | | | | | | | | | | | | | | | |
| | Specimen temperature excursion | | | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | | | |
| Treatment administration | Any type | | | | | | | | | | | | | | | | |
| | Required procedure done incorrectly | | | | | | | | | | | | | | | | |

Table 5: Distribution of Protocol Deviations by Category, Type, and Treatment Group (continued)

| | | Oral 5 µ | ort A:<br>ug dmLT<br>=X) | Oral<br>dm | ort B:<br>25 μg<br>LT<br>=X) | Coh<br>Plac | Oral<br>orts:<br>cebo<br>=X) | Sub | l Route<br>jects<br>=X) | Coho<br>Subling<br>dm<br>(N= | ual 5 µg | Sublings<br>dm | ort D:<br>ual 25 µg<br>LT<br>=X) | Coh<br>Plac | olingual<br>orts:<br>cebo<br>=X) | Route S | olingual<br>Subjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. | No. of<br>Subj. | No. of<br>Dev. |
| | Study product temperature excursion | | | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | | | |
| Blinding policy/<br>procedure | Any type | | | | | | | | | | | | | | | | |
| | Treatment unblinded | | | | | | | | | | | | | | | | |
| | Other | | | | | | | | | | | | | | | | |

Note: N= Number of subjects in the Safety Population

Tables with similar format:

### Table 6: Distribution of Protocol Deviations by Category, Type, and Treatment Group – Intradermal & Pooled Cohorts

# 12.2.2 Displays of Adverse Events

**Table 7:** Solicited Adverse Event Grading Scale

| Solicited Adverse Event | Normal | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|---|
| Fever (Oral °C) | 35-37.9 | 38.0 to 38.4 | 38.5 to 38.9 | ≥39.0 |
| Feverishness (Chills/Shivering/Sweating) | none | Mild, but no interference with function | Some interference with daily activity | Significant interference, prevents daily activity |
| Fatigue<br>(Tiredness) | Normal activity reduced slightly | Normal activity decreased 25-50% | Unable to perform daily activity | Urgent care visit or hospitalization |
| Malaise<br>(General Unwell Feeling) | No interference with daily activity | Some interference with daily activity | Significant interference with daily activity | Urgent care visit or hospitalization |
| Myalgia<br>(Body/Muscle Aches) | Mild, but no interference with function | Moderate, interferes with function, but not with daily activity | Severe, interferes with daily activity | Severe and disabling,<br>unable to perform daily<br>activity |
| Headache | Mild and brief or easily tolerated | Moderate with limited effect to daily activity | Severe and prevents daily activity | Urgent care visit or hospitalization |
| Diarrhea | Normal or 1-2<br>loose stool per 24<br>hr | 3 loose stools per 24 hr | 4-7 loose stools per 24 hr | 8 or more loose/watery<br>stools per 24 hr or<br>requires outpatient IV<br>hydration, ED visit or<br>hospitalization for<br>diarrhea |
| Nausea | none | Mild, but no interference with activity or intake | Moderate, interferes with activity or intake | Severe, unable to perform activity or no intake |
| Vomiting | none | 1-2 episodes<br>per 24 hr. | 3-4 episodes<br>per 24 hr. | ≥5 episodes<br>per 24 hr. |
| Abdominal Discomfort | No interference with daily activity | Some interference with daily activity | Significant interference with daily activity | Urgent care visit or hospitalization |
| Irritation of Oral Cavity<br>(Mouth Pain/Sores) | none | Mild or transient, no limitation of oral intake | Moderate, slight interference with oral intake | Severe, unable to tolerate oral intake |
| Facial Nerve Disturbance | none | Mild or transient, no limitation | Moderate disturbance but no overt facial nerve palsy | Severe, obvious facial nerve palsy |
| Injection Site Pain | none | Aware of pain but no interference with activity | Slight interference with activity, may require analgesic | Pain that prevents daily activity |
| Injection Site Redness | none | Less than 5x5 cm | Greater than 5x5 cm but less than 9x9 cm | Greater than 9x9 cm |
| Injection Site Swelling | none | Less than 5x5 cm | Greater than 5x5 cm but less than 9x9 cm | Greater than 9x9 cm or ulceration or necrosis |
| Injection Site Bruising (Ecchymosis) | none | Less than 5x5 cm | Greater than 5x5 cm but less than 9x9 cm | Greater than 9x9 cm |
| Injection Site Itching | none | Aware of sensation but no interference with activity | Slight interference with activity, may require medication | Itching that prevents daily activity |
| Injection Site Induration (limited to the dermal layer) | none | Less than 5x5 cm | Greater than 5x5 cm but less than 9x9 cm | Greater than 9x9 cm |
| Injection Site<br>Hypo/Hyperpigmentation | none | Less than 1x1 cm | Greater than 1x1 cm but less than 5x5 cm | Greater than 5x5 cm |
| Injection Site Vesicles | none | | >5 vesicles and localized to injection site | Any number of vesicles which are generalized in distribution |
| Injection Site Hardened Mass (deeper than dermal layer) | none | Less than 1x1 cm | Greater than 1x1 cm but less than 5x5 cm | Greater than 5x5 cm |

# 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

**Table 8:** Laboratory Adverse Event Grading Scale

| Solicited Lab AEs | Grade 1 – Mild | Grade 2 – Moderate | Grade 3 - Severe |
|---|---|---|---|
| WBC, Decreased (cells x10 <sup>9</sup> /Liter) | 2.0 – 3.9 | 1.5 – 1.9 | ≤1.4 |
| WBC, Increased (cells x10 <sup>9</sup> /Liter) | 11.1 – 15.0 | 15.1 – 20.0 | ≥20.1 |
| ANC, Decreased (cells x10 <sup>9</sup> /Liter) | 1.0 – 1.9 | 0.75 – 0.99 | ≤0.74 |
| Hemoglobin, female (mg/dL) | 9.0- 9.4 | 8.0 - 8.9 | 6.5 – 7.9 |
| Hemoglobin, male (mg/dL) | 10.0 - 10.9 | 9.0 – 9.9 | 7.0 – 8.9 |
| Platelets<br>(cells x 10 <sup>9</sup> /Liter) | 100 – 149 | 50 – 99 | ≤49 |
| Creatinine (μmol/Liter) | 1.1 – 1.3 x ULN* | >1.3 – 1.8 x ULN* | >1.8 – 3.4 x ULN* |
| ALT (SGPT)<br>(U/L) | 1.25 – 2.5 x ULN* | >2.5 – 5.0 x ULN* | >5.0 – 10.0 x ULN* |
| Albumin<br>(g/dL) | 2.8 - 3.1 | 2.5 - 2.7 | < 2.5 |

<sup>\*</sup>ULN = upper limit of normal, from the laboratory reference range

**Table 9: Vital Sign Adverse Event Grading Scale** 

| Vital Sign | Normal | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) |
|---|---|---|---|---|
| Temperature, °C | 35-37.9 | 38.0 to 38.4 | 38.5 to 38.9 | ≥39.0 |
| Tachycardia, bpm* | ≤100 | 101 to 115 | 116 to 130 | >130 |
| Bradycardia, bpm* | ≥50 | 45 to 49 | 40 to 44 | <40 |
| Hypertension, systolic, mmHg | ≤140 | 141 to 150 | 151 to 155 | >155 |
| Hypotension, systolic, mmHg | ≥90 | 85-89 | 80-84 | <80 |
| Hypertension, diastolic, mmHg | ≤90 | 91-95 | 96-100 | >100 |
| Hypotension, diastolic, mmHg | ≥60 | 45-59 | 35-44 | <35 |

<sup>\*</sup>bpm = beats per minute

#### 14.1 Description of Study Subjects

#### 14.1.1 Disposition of Subjects

**Table 10:** Subject Disposition by Treatment Group - Oral & Sublingual Cohorts

| Subject | Oral 5 µ | ort A:<br>ug dmLT<br>=X) | Oral 25 | ort B:<br>ug dmLT<br>=X) | Pla | Cohorts:<br>cebo<br>=X) | Sub | al Route<br>jects<br>=X) | Subling<br>dm | ort C:<br>gual 5 μg<br>aLT<br>=X) | Sublings<br>dm | ort D:<br>ual 25 μg<br>LT<br>=X) | Cohorts | olingual<br>: Placebo<br>=X) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Disposition | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Screened | | | | | | | | | х | | | | | | | |
| Enrolled/Randomized | x | 100 | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 | х | 100 |
| Received Dose 1 <sup>a</sup> | x | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx |
| Received Dose 2 <sup>a</sup> | | | | | | | | | | | | | | | | |
| Received Dose 3 <sup>a</sup> | | | | | | | | | | | | | | | | |
| Completed Final<br>Blood Draw (Study<br>Day 209) | | | | | | | | | | | | | | | | |
| Completed Follow-up (Study Day 209) <sup>a</sup> | | | | | | | | | | | | | | | | |
| Completed Per<br>Protocol <sup>b</sup> | | | | | | | | | | | | | | | | |

Note: N=Number of subjects enrolled

#### Tables with similar format:

#### **Table 11:** Subject Disposition by Treatment Group - Intradermal & Pooled Cohorts

[Implementation note: Study Day for "Completed Final Blood Draw" and "Completed Follow-Up" is Day 223 for Intradermal Cohort. Treatment groups are Cohort E: Intradermal 0.3  $\mu$ g dmLT (N=X), Cohort E: Intradermal Placebo (N=X), and All Intradermal Route Subjects (N=X). All Subjects (N=X) will be added at the end.]

<sup>&</sup>lt;sup>a</sup> Refer to Listing 16.2.1 for reasons subjects discontinued or terminated early.

<sup>&</sup>lt;sup>b</sup> Refer to Listing 16.2.3 for reasons subjects are excluded from the Analysis populations.

**Table 12:** Analysis Populations by Treatment Group – Oral & Sublingual Cohorts

| | Reason Subjects | Oral 5 µ | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | | All Oral<br>Cohorts: Placebo<br>(N=X) | | All Oral Route<br>Subjects<br>(N=X) | | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | | olingual<br>: Placebo<br>=X) | Route S | olingual<br>Subjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Analysis Populations</b> | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| [Population 1, for<br>example: Per Protocol<br>Immunogenicity<br>Analysis Cohort] | Any Reason | xx | XX | XX | XX | xx | xx | XX | xx | xx | xx | xx | xx | xx | XX | xx | xx |
| | [Reason 1, for example:<br>Did not meet eligibility<br>criteria] | | | | | | | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | | | | | | | |
| | [Reason 4] | | | | | | | | | | | | | | | | |
| [Population 2, for<br>example: Safety<br>Analysis Cohort] | Any Reason | | | | | | | | | | | | | | | | |
| | [Reason 1] | | | | | | | | | | | | | | | | |
| | [Reason 2] | | | | | | | | | | | | | | | | |

Note: N=Number of subjects enrolled

Tables with similar format:

## **Table 13:** Analysis Populations by Treatment Group – Intradermal & Pooled Cohorts

Table 14: Dates of First Treatment by Treatment Group - Oral & Sublingual Cohorts

| Dates of Dosing | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 μg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo<br>(N=X) | All Oral Route<br>Subjects<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts: Placebo<br>(N=X) | All Sublingual<br>Route Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
| Total (Entire period of enrollment) | | X | X | X | X | | | |
| DDMMMYYYY-<br>DDMMMYYYY | | | | | | | | |
| [categorize based on length of enrollment period] | X | | | | | | | |

Note: N=Number of subjects enrolled

Tables with similar format:

#### **Table 15:** Dates of First Treatment by Treatment Group – Intradermal & Pooled Cohorts

**Table 16: Ineligibility Summary of Screen Failures** 

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | ₀∕₀ <sup>b</sup> |
|---|---|---|---|
| Inclusion and Exclusion | Number of subjects failing any eligibility criterion | X | 100 |
| Inclusion | Any inclusion criterion | X | XX |
| | [inclusion criterion 1] | X | xx |
| | [inclusion criterion 2] | X | XX |
| | [inclusion criterion 3] | X | xx |
| Exclusion | Any exclusion criterion | X | xx |
| | [exclusion criterion 1] | X | xx |
| | [exclusion criterion 2] | X | xx |
| | [exclusion criterion 3] | X | xx |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per subject.

<sup>b</sup> Denominator for percentages is the total number of screen failures.

### 14.1.2 Demographic Data by Study Group

Table 17: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group - Oral & Sublingual Cohorts

| Variable | Characteristic | Characteristic Cohort A: Oral 5 μg dmLT (N=X) | | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | | All Oral Route<br>Subjects<br>(N=X) | | Cohort C:<br>Sublingual 5<br>µg dmLT<br>(N=X) | | Cohort D:<br>Sublingual 25<br>µg dmLT<br>(N=X) | | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | | All Sublingual<br>Route<br>Subjects<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | X | XX | х | XX | х | xx | х | XX | X | XX | х | XX | х | XX | х | XX |
| | Female | | | | | | | | | | | | | | | | |
| Ethnicity | Bengali | X | XX | х | XX | Х | xx | х | XX | X | XX | х | XX | х | XX | х | XX |
| | Other | | | | | | | | | | | | | | | | |
| Race | American Indian or Alaska Native | X | xx | х | XX | х | XX | X | XX | X | XX | х | XX | х | XX | х | XX |
| | Asian | | | | | | | | | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | | | | | | | | | |
| | Black or African American | | | | | | | | | | | | | | | | |
| | White | | | | | | | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | | | | | | | |
| | Unknown | | | | | | | | | | | | | | | | |

Note: N=Number of subjects enrolled

Tables with similar format:

### Table 18: Summary of Categorical Demographic and Baseline Characteristics by Treatment Group – Intradermal & Pooled Cohorts

Table 19: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group – Oral & Sublingual Cohorts

| Variable | Statistic | Cohort A:<br>Oral 5 μg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo<br>(N=X) | All Oral Route<br>Subjects<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts: Placebo<br>(N=X) | All Sublingual<br>Route Subjects<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Age (units) | Mean | XX | XX | XX | xx | XX | xx | XX | xx |
| | Standard Deviation | XX | XX | XX | xx | XX | XX | XX | xx |
| | Median | X | X | X | X | X | X | X | x |
| | Minimum | х | х | X | X | X | X | X | х |
| | Maximum | х | х | х | х | X | X | х | х |

Note: N=Number of subjects enrolled

Tables with similar format:

# Table 20: Summary of Continuous Demographic and Baseline Characteristics by Treatment Group – Intradermal & Pooled Cohorts

### 14.2 Immunogenicity Data

Table 21: Serum IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1a | N | x | X | х | X | X | X | х | X |
| | GMT | x.x | x.x | x.x | X.X | X.X | X.X | x.x | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3e | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day<br>28g | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day<br>85 <sup>h</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

Note: N=Number of subjects in the mITT Population

#### Tables with similar format:

Serum IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population **Table 22:** 

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>h</sup>Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort
Table 23: Serum IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A: Oral 5<br>µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | N | X | X | Х | X | x | X | x | Х |
| | GMT | x.x | x.x | x.x | X.X | X.X | x.x | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3e | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| Time Point | Statistic | Cohort A: Oral 5 µg dmLT (N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day<br>28g | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day<br>85 <sup>h</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

**Table 24:** Serum IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>h</sup>Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

Table 25: Serum LT Toxin Neutralization GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A: Oral 5 µg dmLT (N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | N | x | X | X | X | X | X | X | X |
| | GMT | x.x | x.x | x.x | X.X | x.x | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3 <sup>e</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A: Oral 5 µg dmLT (N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 28g | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 85h | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

Table 26: Serum LT Toxin Neutralization GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

eDay 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup>Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>h</sup>Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

 Table 27:
 ASC IgA Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 μg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | n | х | х | X | х | x | X | х | X |
| | Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Median | x.x | x.x | X.X | X.X | x.x | x.x | x.x | X.X |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3 <sup>e</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| | | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT | All Oral<br>Cohorts:<br>Placebo | Cohort C:<br>Sublingual 5 μg<br>dmLT | Cohort D:<br>Sublingual 25 μg<br>dmLT | All Sublingual<br>Cohorts:<br>Placebo | Cohort E:<br>Intradermal 0.3<br>µg dmLT | Cohort E:<br>Intradermal<br>Placebo |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | (11 21) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |

Tables with similar format:

ASC IgA Results by Time Point and Treatment Group, Per Protocol Population **Table 28:** 

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort <sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

eDay 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

Table 29: ASC IgG Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 μg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 μg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | n | Х | х | х | х | X | х | X | X |
| | Mean (SD) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) | x.x (x.x) |
| | Median | x.x | x.x | x.x | x.x | x.x | x.x | x.x | X.X |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3 <sup>e</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| | | Cohort A:<br>Oral 5 μg | Cohort B:<br>Oral 25 µg | All Oral<br>Cohorts: | Cohort C:<br>Sublingual 5 µg | Cohort D:<br>Sublingual 25 µg | All Sublingual<br>Cohorts: | Cohort E:<br>Intradermal 0.3 | Cohort E:<br>Intradermal |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | dmLT<br>(N=X) | dmLT<br>(N=X) | Placebo<br>(N=X) | dmLT<br>(N=X) | dmLT<br>(N=X) | Placebo<br>(N=X) | μg dmLT<br>(N=X) | Placebo<br>(N=X) |

# Tables with similar format:

Table 30: ASC IgG Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort <sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

eDay 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

Table 31: ALS IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | N | х | x | x | x | Х | Х | X | х |
| | GMT | x.x | X.X | X.X | x.x | x.x | x.x | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3 <sup>e</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E: Intradermal Placebo (N=X) |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

Tables with similar format:

Table 32: ALS IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

Table 33: ALS IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | N | x | x | х | X | x | x | х | x |
| | GMT | x.x | x.x | x.x | x.x | x.x | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | | | | | | | | |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3 <sup>e</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 μg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

Tables with similar format:

ALS IgG GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population **Table 34:** 

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

eDay 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

Table 35: Fecal dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1a | N | Х | х | х | х | х | X | х | х |
| | GMT | x.x | x.x | x.x | X.X | X.X | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3 <sup>e</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day<br>28g | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

## Tables with similar format:

**Table 36:** Fecal dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol **Population** 

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

Table 37: Fecal dmLT-specific/Total IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | N | X | Х | x | х | X | x | X | х |
| | GMT | x.x | x.x | X.X | X.X | x.x | X.X | x.x | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7d | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3e | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 28g | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

Table 38: Fecal dmLT-specific/Total IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup>Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

Table 39: Salivary dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | N | х | x | X | X | X | X | X | x |
| | GMT | x.x | X.X | x.x | X.X | X.X | X.X | x.x | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3e | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 28g | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

Table 40: Salivary dmLT-specific IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup>Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

Table 41: Salivary dmLT-specific/Total IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 μg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | N | X | X | X | x | х | х | X | X |
| | GMT | x.x | x.x | x.x | X.X | x.x | x.x | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | [Min,Max] | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Post-Dose 1 Day 7 <sup>b</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Pre-Dose 3e | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | [Min,Max] | | | | | | | | |
| Post-Dose 3 Day 28g | N | | | | | | | | |
| | GMT | | | | | | | | |
| | 95% CI | | | | | | | | |
| | [Min,Max] | | | | | | | | |

Table 42: Salivary dmLT-specific/Total IgA GMT Results with 95% Confidence Intervals by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup>Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

Table 43: Serum IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | х | X | X | X | X | X | X | X |
| | GMFR <sup>h</sup> | x.x | x.x | X.X | X.X | X.X | X.X | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 4-Fold Rise <sup>i</sup> | x.x | x.x | x.x | X.X | x.x | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Risei | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>d</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 28 <sup>f</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 85g | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

Table 44: Serum IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort <sup>d</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup> Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

<sup>&</sup>lt;sup>h</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

<sup>&</sup>lt;sup>1</sup>4 -Fold Rise represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to pre-dose 1.

Table 45: Serum IgG GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | Х | X | х | X | X | X | Х | x |
| | GMFR <sup>g</sup> | x.x | X.X | x.x | X.X | X.X | X.X | x.x | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 4-Fold Riseh | x.x | X.X | x.x | X.X | X.X | X.X | x.x | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>d</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 28 <sup>f</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 85g | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 μg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

Table 46: Serum IgG GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort <sup>d</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup> Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

<sup>&</sup>lt;sup>h</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

<sup>&</sup>lt;sup>1</sup>4-Fold Rise represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to pre-dose 1.

Table 47: Serum LT Toxin Neutralization GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | х | X | X | X | X | X | X | X |
| | GMFR <sup>h</sup> | x.x | x.x | x.x | X.X | X.X | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 4-Fold Rise <sup>i</sup> | x.x | x.x | x.x | X.X | X.X | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3d | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 28 <sup>f</sup> | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 85g | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>i</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

Tables with similar format:

Table 48: Serum LT Toxin Neutralization GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup>Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup>Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

<sup>&</sup>lt;sup>h</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

<sup>&</sup>lt;sup>1</sup>4-Fold Rise represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to pre-dose 1.

Table 49: ASC IgA Response Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5<br>µg dmLT<br>(N=X) | Cohort D:<br>Sublingual 25<br>µg dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal<br>0.3 µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | n | Х | X | X | X | х | X | X | X |
| | Proportion with ASC Response <sup>g</sup> | X.XX | X.XX | x.xx | x.xx | x.xx | X.XX | X.XX | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Post-Dose 1 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>e</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| | | Cohort A: | Cohort B: | All Oral | Cohort C: | Cohort D: | All Sublingual | Cohort E: | Cohort E: |
|---|---|---|---|---|---|---|---|---|---|
| | | Oral 5 µg | Oral 25 µg | Cohorts: | Sublingual 5 | Sublingual 25 | Cohorts: | Intradermal | Intradermal |
| | | dmLT | dmLT | Placebo | μg dmLT | μg dmLT | Placebo | 0.3 µg dmLT | Placebo |
| Time Point | Statistic | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |

Tables with similar format:

ASC IgA Response Results by Time Point and Treatment Group, Oral & Sublingual Cohorts, Per Protocol Population **Table 50:** 

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort <sup>d</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

f Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort g Defined as  $\geq$ 8 IgA ASC/10<sup>6</sup> PBMCs

Table 51: ASC IgG Response Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5<br>µg dmLT<br>(N=X) | Cohort D:<br>Sublingual 25<br>µg dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal<br>0.3 µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Pre-Dose 1 <sup>a</sup> | n | X | Х | х | Х | Х | X | X | Х |
| | Proportion with ASC Response <sup>g</sup> | X.XX | x.xx | x.xx | X.XX | x.xx | X.XX | X.XX | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Post-Dose 1 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 2 <sup>c</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2 Day 7 <sup>d</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3e | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3 Day 7 <sup>f</sup> | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time Post Dose | n | | | | | | | | |
| | Proportion with ASC Response <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| | | Cohort A: | Cohort B: | All Oral | Cohort C: | Cohort D: | All Sublingual | Cohort E: | Cohort E: |
|---|---|---|---|---|---|---|---|---|---|
| | | Oral 5 µg | Oral 25 µg | Cohorts: | Sublingual 5 | Sublingual 25 | Cohorts: | Intradermal | Intradermal |
| | | dmLT | dmLT | Placebo | μg dmLT | μg dmLT | Placebo | 0.3 μg dmLT | Placebo |
| Time Point | Statistic | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |

Tables with similar format:

ASC IgG Response Results by Time Point and Treatment Group, Per Protocol Population **Table 52:** 

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 8

<sup>&</sup>lt;sup>c</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort <sup>d</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

e Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort f Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort g Defined as ≥8 IgA ASC/10<sup>6</sup> PBMCs

Table 53: ALS IgA GMFR and 2-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | X | X | X | X | X | X | X | X |
| | GMFR <sup>f</sup> | X.X | X.X | X.X | x.x | X.X | X.X | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 2-Fold Rise <sup>g</sup> | X.X | x.x | x.x | X.X | x.x | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Rise <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2,<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Rise <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>d</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Riseg | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3,<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | | | |
| | 2-Fold Rise <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Riseg | | | | | | | | |
| | 95% CI | | | | | | | | |

Table 54: ALS IgA GMFR and 2-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

g 2-Fold Rise represents the percentage of subjects with at least a 2-Fold Rise in antibody compared to pre-dose 1.

Table 55: ALS IgG GMFR and 2-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1 Day<br>7 <sup>a</sup> | N | x | X | X | X | X | X | X | X |
| | GMFR <sup>f</sup> | x.x | x.x | x.x | x.x | X.X | x.x | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 2-Fold Riseg | x.x | x.x | x.x | x.x | x.x | x.x | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Riseg | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2, Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Riseg | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>d</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Riseg | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3, Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| Time Point | Statistic | Cohort A:<br>Oral 5 μg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 95% CI | | | | | | | | |
| | 2-Fold Riseg | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time Post<br>Dose 1 | N | | | | | | | | |
| | GMFR <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 2-Fold Rise <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

Tables with similar format:

Table 56: ALS IgG GMFR and 2-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

f GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

g 2-Fold Rise represents the percentage of subjects with at least a 2-Fold Rise in antibody compared to pre-dose 1.

Table 57: ASC Homing Markers IgA by Time Point and Treatment Group, mITT Population

| 1 | | 8 | | | 1 / | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 μg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
| dmLT-specij | fic IgA Gut Homing AS | SC (a4/β7+) | | | | | | | |
| Day 8 | n | х | х | Х | х | х | Х | х | X |
| | IgA ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Post-Dose<br>2 Day 7 <sup>a</sup> | n | x | x | x | x | x | х | X | x |
| | IgA ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Post-Dose<br>3 Day 7 <sup>b</sup> | n | x | X | х | х | Х | Х | Х | х |
| | IgA ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX | x.xx | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Any Time | n | х | х | х | x | х | X | х | X |
| | IgA ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Total IgA G | ut Homing ASC (α4/β7 | ·<br>/+) | | | | | | | |
| Day 8 | n | | | | | | | | |
| | IgA ASC Response <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose<br>2 Day 7 <sup>a</sup> | n | | | | | | | | |
| | IgA ASC Response <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose<br>3 Day 7 <sup>b</sup> | n | | | | | | | | |

| IgA ASC Response <sup>f</sup> | | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| 95% CI | | | | | | | | |
| n | | | | | | | | |
| IgA ASC Response <sup>f</sup> | | | | | | | | |
| 95% CI | | | | | | | | |
| ic / Total IgA Gut Hon | ning ASC (\alpha4/\beta7+) | | | | | | | |
| n | | | | | | | | |
| IgA ASC Response <sup>f</sup> | | | | | | | | |
| 95% CI | | | | | | | | |
| | 95% CI n IgA ASC Response <sup>f</sup> 95% CI ic / Total IgA Gut Hon n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> | 95% CI n IgA ASC Response <sup>f</sup> 95% CI ic / Total IgA Gut Homing ASC (a4/\beta 7+) n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> | 95% CI n IgA ASC Response <sup>f</sup> 95% CI ic / Total IgA Gut Homing ASC (α4/β7+) n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n | 95% CI n IgA ASC Response <sup>f</sup> 95% CI ic / Total IgA Gut Homing ASC (α4/β7+) n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n | 95% CI n IgA ASC Response <sup>f</sup> 95% CI ic / Total IgA Gut Homing ASC (α4/β7+) n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n | 95% CI n IgA ASC Response <sup>f</sup> 95% CI ig / Total IgA Gut Homing ASC (α4/β7+) n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n IgA ASC Response <sup>f</sup> 95% CI n | 95% CI n IgA ASC Response <sup>c</sup> 95% CI 95% CI 10 11 12A ASC Response <sup>c</sup> 95% CI 11 12A ASC Response <sup>c</sup> 95% CI 12A ASC Response <sup>c</sup> 95% CI 13A ASC Response <sup>c</sup> 95% CI 14A ASC Response <sup>c</sup> 95% CI 15A ASC Response <sup>c</sup> 95% CI 16A ASC Response <sup>c</sup> | 95% CI n lgA ASC Response <sup>f</sup> 95% CI psylon 1gA ASC Response <sup>f</sup> 95% CI n lgA ASC Response <sup>f</sup> 95% CI n |

Tables with similar format:

**Table 58:** ASC Homing Markers IgA by Time Point and Treatment Group, Per Protocol Population

N=Number of subjects in the mITT Population

<sup>a</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>b</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

Table 59: ASC Homing Markers IgG by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| dmLT-specifi | ic IgG Gut Homing ASC | $C(\alpha 4/\beta 7+)$ | | | | | | | |
| Day 8 | n | х | х | X | X | х | х | х | X |
| | IgG ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Post-Dose 2<br>Day 7 <sup>a</sup> | n | x | x | х | х | х | x | х | X |
| | IgG ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Post-Dose 3<br>Day 7 <sup>b</sup> | n | x | X | х | Х | х | X | X | x |
| | IgG ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Any Time | n | х | х | X | х | х | х | х | X |
| | IgG ASC Response <sup>f</sup> | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | x.xx | X.XX |
| | 95% CI | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| Total IgG Gu | ut Homing ASC (α4/β7+ | ) | | | | | | | |
| Day 8 | n | | | | | | | | |
| | IgG ASC Response <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>a</sup> | n | | | | | | | | |
| | IgG ASC Response <sup>f</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>b</sup> | n | | | | | | | | |

| | IgG ASC Response <sup>f</sup> | | | | | |
|---|---|---|---|---|---|---|
| | 95% CI | | | | | |
| Any Time | n | | | | | |
| | IgG ASC Response <sup>f</sup> | | | | | |
| | 95% CI | | | | | |
| dmLT-specif | ic / Total IgG Gut Homi | ing ASC (α4/β7+) | | | | |
| Day 8 | n | | | | | |
| | IgG ASC Response <sup>f</sup> | | | | | |
| | 95% CI | | | | | |
| Post-Dose 2<br>Day 7 <sup>a</sup> | n | | | | | |
| | IgG ASC Response <sup>f</sup> | | | | | |
| | 95% CI | | | | | |
| Post-Dose 3<br>Day 7 <sup>b</sup> | n | | | | | |
| | IgG ASC Response <sup>f</sup> | | | | | |
| | 95% CI | | | | | |
| Any Time | n | | | | | |
| | IgG ASC Response <sup>f</sup> | | | | | |
| | 95% CI | | | | | |
| NI NI 1 | f subjects in the mITT D | 1 (* | • | • | • | • |

Tables with similar format:

Table 60: ASC Homing Markers IgG by Time Point and Treatment Group, Per Protocol Population

N=Number of subjects in the mITT Population

<sup>a</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>b</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

Table 61: Fecal dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | Х | Х | X | Х | Х | Х | х | X |
| | GMFR <sup>g</sup> | X.X | X.X | x.x | X.X | X.X | X.X | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 4-Fold Riseh | X.X | X.X | X.X | X.X | X.X | X.X | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3d | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 μg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 28 <sup>f</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

Tables with similar format:

Table 62: Fecal dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

h 4-Fold Rise represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to pre-dose 1.

Table 63: Fecal dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 μg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | X | х | X | X | X | X | X | x |
| | GMFR <sup>g</sup> | X.X | X.X | X.X | X.X | X.X | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 4-Fold Riseh | X.X | X.X | X.X | X.X | X.X | X.X | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>d</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 28 <sup>f</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |

## Tables with similar format:

Table 64: Fecal dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

d Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

h 4-Fold Rise represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to pre-dose 1.

Table 65: Salivary dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | X | X | х | X | X | X | х | Х |
| | GMFR <sup>g</sup> | X.X | x.x | x.x | X.X | X.X | x.x | x.x | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 4-Fold Rise <sup>h</sup> | X.X | X.X | x.x | X.X | X.X | X.X | x.x | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>d</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 28 <sup>f</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |

## Tables with similar format:

Table 66: Salivary dmLT-specific IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

h 4-Fold Rise represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to pre-dose 1.

Table 67: Salivary dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, mITT Population

| | | | | Calcad Co. Calcad Do | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
| Post-Dose 1<br>Day 7 <sup>a</sup> | N | X | X | X | X | X | X | X | X |
| | GMFR <sup>g</sup> | X.X | X.X | x.x | X.X | X.X | X.X | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| | 4-Fold Riseh | X.X | X.X | x.x | X.X | X.X | X.X | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Pre-Dose 2 <sup>b</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 2<br>Day 7 <sup>c</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Pre-Dose 3 <sup>d</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 7 <sup>e</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | 4-Fold Rise <sup>h</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| Post-Dose 3<br>Day 28 <sup>f</sup> | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | | | | | | | | |
| Any Time<br>Post Dose 1 | N | | | | | | | | |
| | GMFR <sup>g</sup> | | | | | | | | |
| | 95% CI | | | | | | | | |
| | 4-Fold Riseh | | | | | | | | |
| | 95% CI | the mITT Demulation | | | | | | | |

Tables with similar format:

Table 68: Salivary dmLT-specific/Total IgA GMFR and 4-Fold Rise Results by Time Point and Treatment Group, Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 29 for Oral & Sublingual Cohorts; Day 43 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>g</sup> GMFR represents the geometric mean fold rise in antibody compared to pre-dose 1.

h 4-Fold Rise represents the percentage of subjects with at least a 4-Fold Rise in antibody compared to pre-dose 1.

**Table 69:** Anti-dmLT IgA Memory B Cell Response – mITT Population

| Time Point | Statistic | Cohort A: Oral 5<br>µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| dmLT-specific IgA | (spot-forming cells pe | r 10 <sup>6</sup> PBMC) | | | | | | | |
| Baseline, Pre-<br>Dose 1 <sup>a</sup> | n | х | х | х | х | х | х | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 2 Day<br>7 <sup>b</sup> | n | X | Х | Х | Х | х | х | х | Х |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 3 Day 7c | n | х | х | х | х | х | х | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 3 Day<br>28 <sup>d</sup> | n | х | Х | X | х | х | х | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 3 Day<br>85° | n | х | х | х | х | х | X | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |

| Time Point | Statistic | Cohort A: Oral 5<br>µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day<br>180 <sup>f</sup> | n | х | X | х | X | х | Х | X | х |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| dmLT-specific/tota | l IgA (%) | | | | | | | | |
| Baseline, Pre-<br>Dose 1 <sup>a</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| Post-Dose 2 Day<br>7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day<br>7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day<br>28 <sup>d</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |

| Time Point | Statistic | Cohort A: Oral 5<br>µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day<br>85° | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day<br>180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

Tables with similar format:

**Table 70:** Anti-dmLT IgA Memory B Cell Response – Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup> Day 209 for Oral & Sublingual Cohorts; Day 223 for Intradermal Cohort

g Response represents the percentage of subjects with at least a 0.05% increase in percentage of antigen-specific IgA/total IgA B memory cells from pre-vaccination

 Table 71:
 Anti-dmLT IgG Memory B Cell Response – mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| dmLT-specific IgG (spo | t-forming cells per 10 <sup>6</sup> PB | MC) | | | | | | | |
| Baseline, Pre-Dose 1a | n | х | X | X | x | x | Х | x | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 2 Day 7 <sup>b</sup> | n | х | X | X | X | Х | Х | X | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 3 Day 7 <sup>c</sup> | n | х | X | X | X | х | Х | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 3 Day 28d | n | х | X | X | X | х | Х | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 3 Day 85e | n | х | X | X | X | х | Х | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| Post-Dose 3 Day 180f | n | х | X | X | X | х | Х | х | X |
| | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median [Min, Max] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] | xx [xx,xx] |
| dmLT-specific/total IgG | G (%) | | | | 1 | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg<br>dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg<br>dmLT<br>(N=X) | All Oral<br>Cohorts:<br>Placebo<br>(N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3<br>µg dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7c | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| | | Cohort A:<br>Oral 5 μg | Cohort B:<br>Oral 25 μg | All Oral<br>Cohorts: | Cohort C:<br>Sublingual 5 μg | Cohort D:<br>Sublingual 25 μg | | Cohort E:<br>Intradermal 0.3 | Cohort E:<br>Intradermal |
|---|---|---|---|---|---|---|---|---|---|
| Time Point | Statistia | dmLT | dmLT | Placebo | dmLT | dmLT | Placebo | μg dmLT | Placebo |
| Time Point | Statistic | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) | (N=X) |

## Tables with similar format:

## **Table 72:** Anti-dmLT IgG Memory B Cell Response – Per Protocol Population

<sup>&</sup>lt;sup>a</sup> Day 1

<sup>&</sup>lt;sup>b</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup> Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup> Day 209 for Oral & Sublingual Cohorts; Day 223 for Intradermal Cohort

g Response represents the percentage of subjects with at least a 0.05% increase in percentage of antigen-specific IgG/total IgG B memory cells from pre-vaccination

**Table 73:** T Cell Memory Responses by CyTOF – mITT Population

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Effector function - CD4 | !/IFNg (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | х | x | х | х | X | X | x | Х |
| | Mean (SD) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) |
| | Median<br>[Min, Max] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] |
| Post-Dose 2 Day 7 <sup>b</sup> | n | x | x | х | X | X | X | х | Х |
| | Mean (SD) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) |
| | Median<br>[Min, Max] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] |
| | Response <sup>g</sup> - % (95% CI) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| Post-Dose 3 Day 7 <sup>c</sup> | n | х | x | x | х | x | X | x | Х |
| | Mean (SD) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) |
| | Median<br>[Min, Max] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] |
| | Response <sup>g</sup> - % (95% CI) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| Post-Dose 3 Day 28d | n | X | X | X | X | x | X | X | X |
| | Mean (SD) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) |
| | Median<br>[Min, Max] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] |
| | Response <sup>g</sup> - % (95% CI) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| Post-Dose 3 Day 85e | n | X | X | X | X | X | X | x | X |
| | Mean (SD) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] |
| | Response <sup>g</sup> - % (95% CI) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| Post-Dose 3 Day 180 <sup>f</sup> | n | x | X | x | x | x | X | x | X |
| | Mean (SD) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) | xxx.xx (xxx.xx) |
| | Median<br>[Min, Max] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] | xxx.xx<br>[xxx.xx, xxx.xx] |
| | Response <sup>g</sup> - % (95% CI) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| Any Time Post-Dose 1 | n | x | x | x | x | x | X | х | X |
| | Response <sup>g</sup> - % (95% CI) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) | xx.x (xx.x,xx.x) |
| Effector function - CD4 | /TNFa (%) | | | | | | | | |
| Baseline, Pre-Dose 1 <sup>a</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | /MIP1b (%) | | | | | | | • | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | /CD107a (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | 4/IL-2 (%) | | | | | | | | |
| Baseline, Pre-Dose 1 <sup>a</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7c | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | _ | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | /IL-17A (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | Tem/IFNg (%) | ) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | Tem/TNFa (% | 5) | | • | | | | <u>. </u> | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | , | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Effector function - CD4 | Tem/MIP1b (% | %) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Effector function - CD4 | Tem/CD107a | (%) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | Tem/IL-2 (%) | | | | | | | | |
| Baseline, Pre-Dose 1 <sup>a</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD4 | Tem/IL-17A ( | %) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Effector function - CD8. | /IFNg (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | /TNFa (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | /MIP1b (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | /CD107a (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | /IL-2 (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Effector function - CD8 | /IL-17A (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | Tem/IFNg (%) | ) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | Tem/TNFa (% | <i>(</i> ) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | Tem/MIP1b (9 | %) | | | | | | | |
| Baseline, Pre-Dose 1 <sup>a</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | Tem/CD107a | (%) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85 <sup>e</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median<br>[Min, Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | Tem/IL-2 (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Effector function - CD8 | Tem/IL-17A (S | %) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Homing - CD4/integrin | a4b7 (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Homing - CD4/CCR6 ( | %) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Homing - CD4/CCR4 (% | %) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Homing - CD4/CXCR3 | (%) | | | | | | | <u> </u> | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Homing - CD4 Tem/inte | egrin a4b7 (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Homing - CD8/integrin | a4b7 (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Homing - CD8 Tem/int | egrin a4b7 (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh - CD4/CXCR5 (%) | | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-homing - CXCR5/ | integrin a4b7 ( | %) | | | | | | • | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-homing - CXCR5/ | CCR6 (%) | | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-homing - CXCR5/ | CCR4 (%) | | | | | | | | |
| Baseline, Pre-Dose 1 <sup>a</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-homing - CXCR5/ | CXCR3 (%) | | | | | | | | |
| Baseline, Pre-Dose 1 <sup>a</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-effector function - | CXCR5/IFNg | (%) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-effector function - | CXCR5/TNFa | (%) | | | | | | · | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-effector function - | CXCR5/IL-2 | (%) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-effector function - | CXCR5/IL-21 | (%) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-effector function - | CXCR5/CD15 | 4 (%) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85e | n | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| pTfh-effector function - | CXCR5/ICOS | (%) | | | | | | | |
| Baseline, Pre-Dose 1a | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| Post-Dose 2 Day 7 <sup>b</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 7 <sup>c</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 µg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|---|
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - %<br>(95% CI) | | | | | | | | |
| Post-Dose 3 Day 28d | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 85° | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Post-Dose 3 Day 180 <sup>f</sup> | n | | | | | | | | |
| | Mean (SD) | | | | | | | | |
| | Median [Min,<br>Max] | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |
| Any Time Post-Dose 1 | n | | | | | | | | |
| | Response <sup>g</sup> - % (95% CI) | | | | | | | | |

| Time Point | Statistic | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts:<br>Placebo (N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT (N=X) | All Sublingual<br>Cohorts:<br>Placebo (N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

N=Number of subjects in the mITT Population

**Table 74:** T Cell Memory Responses by CyTOF – Per Protocol Population

<sup>&</sup>lt;sup>a</sup>Screening visit

<sup>&</sup>lt;sup>b</sup>Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort <sup>c</sup>Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup>Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

<sup>&</sup>lt;sup>e</sup>Day 114 for Oral & Sublingual Cohorts; Day 128 for Intradermal Cohort

<sup>&</sup>lt;sup>f</sup>Day 209 for Oral & Sublingual Cohorts; Day 223 for Intradermal Cohort

gResponse represents the percentage of subjects with a post-vaccination increase of >0.05%

Table 75: Correlation of Serum IgA GMFR vs Fecal dmLT-specific IgA GMFR by Time Point and Treatment Group, Immunogenicity Population

| | | Spearman Correlation (95% CI) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 μg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal Placebo<br>(N=X) |
| Max Any Time<br>Post Dose 1 | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) |

- Table 76: Correlation of Serum IgA GMFR vs Fecal dmLT-specific IgA GMFR by Time Point and Treatment Group, Per Protocol Population
- Table 77: Correlation of Serum IgA GMFR vs Fecal dmLT-specific/Total IgA GMFR by Time Point and Treatment Group, Immunogenicity Population
- Table 78: Correlation of Serum IgA GMFR vs Fecal dmLT-specific/Total IgA GMFR by Time Point and Treatment Group, Per Protocol Population

Table 79: Correlation of Serum IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population

| | | | | Spearman Corre | elation (95% CI) | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal Placebo<br>(N=X) |
| Max Any Time<br>Post Dose 1 | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) |

Table 80: Correlation of Serum IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population

Table 81: Correlation of Serum IgG GMFR vs ALS IgG Titers GMFR by Time Point and Treatment Group, Immunogenicity Population

| | | Spearman Correlation (95% CI) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 μg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 μg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal Placebo<br>(N=X) |
| Max Any Time<br>Post Dose 1 | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) |

Table 82: Correlation of Serum IgG GMFR vs ALS IgG Titers GMFR by Time Point and Treatment Group, Per Protocol Population

Table 83: Correlation of Fecal dmLT-specific IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population

| | | | | Spearman Corr | elation (95% CI) | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal<br>Placebo<br>(N=X) |
| Max Any Time<br>Post Dose 1 | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx) -x.xxx | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) |

Table 84: Correlation of Fecal dmLT-specific IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population

Table 85: Correlation of Fecal dmLT-specific/Total IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population

| | | Spearman Correlation (95% CI) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal Placebo<br>(N=X) |
| Max Any Time<br>Post Dose 1 | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) |

Table 86: Correlation of Fecal dmLT-specific/Total IgA GMFR vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population

Table 87: Correlation of ASC IgA Count vs ALS IgA Titers GMFR by Time Point and Treatment Group, Immunogenicity Population

| | | | | Spearman Corre | elation (95% CI) | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 μg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal Placebo<br>(N=X) |
| Max Any Time<br>Post Dose 1 | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) |

Table 88: Correlation of ASC IgA Count vs ALS IgA Titers GMFR by Time Point and Treatment Group, Per Protocol Population

Table 89: Correlation of ASC IgG Count vs ALS IgG Titers GMFR by Time Point and Treatment Group, Immunogenicity Population

| | | | | Spearman Corre | elation (95% CI) | | | |
|---|---|---|---|---|---|---|---|---|
| Time Point | Cohort A:<br>Oral 5 µg dmLT<br>(N=X) | Cohort B:<br>Oral 25 µg dmLT<br>(N=X) | All Oral Cohorts: Placebo (N=X) | Cohort C:<br>Sublingual 5 µg<br>dmLT<br>(N=X) | Cohort D:<br>Sublingual 25 µg<br>dmLT<br>(N=X) | All Sublingual<br>Cohorts:<br>Placebo<br>(N=X) | Cohort E:<br>Intradermal 0.3 μg<br>dmLT<br>(N=X) | Cohort E:<br>Intradermal Placebo<br>(N=X) |
| Max Any Time<br>Post Dose 1 | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) | x.xx<br>(x.xxx-x.xxx) |

Table 90: Correlation of ASC IgG Count vs ALS IgG Titers GMFR by Time Point and Treatment Group, Per Protocol Population

#### 14.3 Safety Data

### 14.3.1 Displays of Adverse Events

**Table 91:** Overall Summary of Adverse Events - Oral & Sublingual Cohorts

| | 5 μg | A: Oral<br>dmLT<br>=X) | Oral<br>dn | ort B:<br>25 µg<br>1LT<br>=X) | Coh<br>Pla | Oral<br>orts:<br>cebo<br>=X) | Sub | nl Route<br>jects<br>=X) | Subling<br>dm | ort C:<br>gual 5 μg<br>nLT<br>=X) | Sublin<br>µg d | ort D:<br>gual 25<br>mLT<br>=X) | Coh<br>Pla | olingual<br>orts:<br>cebo<br>=X) | Route S | olingual<br>Subjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one local solicited adverse event | x | X | x | х | x | x | x | x | х | X | X | х | х | Х | X | x |
| At least one systemic solicited adverse event | х | Х | х | х | х | Х | Х | х | Х | X | X | х | х | Х | х | х |
| At least one unsolicited adverse event | X | X | X | X | X | X | X | X | X | X | Х | X | X | X | X | X |
| At least one related unsolicited<br>adverse event, through 28 days<br>after the last dose | х | X | х | x | х | х | х | х | х | X | X | X | X | X | X | х |
| Mild (Grade 1) | х | x | х | х | х | х | х | х | х | X | X | х | х | X | х | х |
| Moderate (Grade 2) | х | x | х | х | х | х | х | х | х | x | X | х | х | х | х | х |
| Severe (Grade 3) | х | X | х | х | х | х | х | х | х | X | X | х | х | х | х | х |
| Not yet assessed | | | | | | | | | | | | | | | | |
| At least one related unsolicited adverse event, from first vaccination through 6 months after the last dose | X | X | X | X | X | X | X | X | X | x | Х | X | X | X | X | X |
| Mild (Grade 1) | х | X | х | х | х | х | х | х | х | X | X | х | х | х | х | х |
| Moderate (Grade 2) | х | X | X | Х | х | х | х | х | х | X | X | х | х | X | X | х |
| Severe (Grade 3) | х | X | X | X | X | Х | х | X | X | X | X | X | X | X | X | X |
| Not yet assessed | | | | | | | | | | | | | | | | |

| | 5 μg ( | A: Oral<br>dmLT<br>=X) | Oral<br>dm | ort B:<br>25 μg<br>aLT<br>=X) | Coh<br>Pla | Oral<br>orts:<br>cebo<br>=X) | Sub | ll Route<br>jects<br>=X) | Subling<br>dm | ort C:<br>gual 5 µg<br>nLT<br>=X) | Sublin<br>µg d | ort D:<br>gual 25<br>mLT<br>=X) | Coh<br>Plac | olingual<br>orts:<br>cebo<br>=X) | Route | blingual<br>Subjects<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subjects <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| At least one severe (Grade 3) unsolicited adverse event | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | х |
| Related | х | X | x | х | X | х | х | X | х | х | X | х | x | x | х | х |
| Unrelated | Х | х | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| At least one serious adverse event <sup>b</sup> | X | X | X | X | X | X | x | X | X | X | X | X | X | X | x | х |
| At least one related, serious adverse event | х | х | х | х | х | х | х | х | х | х | х | х | Х | х | х | х |
| At least one adverse event leading to early termination <sup>c</sup> | х | х | Х | х | х | х | х | х | х | х | X | х | х | X | х | х |
| Study withdrawal for any reason | х | x | X | х | х | х | х | х | х | x | x | х | X | х | x | x |
| Discontinuation of study vaccination for any reason | х | Х | X | х | X | х | Х | X | х | х | X | х | X | X | х | х |

N = Number of subjects in the Safety Population

#### **Table 92:** Overall Summary of Adverse Events - Intradermal & Pooled Cohorts

[Implementation note: Treatment groups are Cohort E: Intradermal 0.3  $\mu$ g dmLT (N=X), Cohort E: Intradermal Placebo (N=X), and All Intradermal Route Subjects (N=X). All Subjects (N=X) will be added at the end.]

<sup>&</sup>lt;sup>a</sup> Subjects are counted once for each category regardless of the number of events.

<sup>&</sup>lt;sup>b</sup> A listing of Serious Adverse Events is included in Table 122.

<sup>&</sup>lt;sup>c</sup> As reported on the Adverse Event eCRF.

Table 93: Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Oral & Sublingual Cohorts

| MedDRA Preferred<br>Term | MedDRA System<br>Organ Class | | Cohort<br>I 5 µg<br>(N=X | dmLT | 0 | Cohortoral 25 dmL (N=X | 5μg<br>T | _ | Oral C<br>Placel<br>(N=X | | \$ | Oral l<br>Subjec<br>(N=X | | Sub | Cohort<br>lingua<br>dmL'<br>(N=X | ıl 5 μg<br>T | Subli | ohort<br>ingual<br>dmL'<br>(N=X | l 25 μg<br>Τ | ( | Subli<br>Cohor<br>Placel<br>(N=X | bo | Rou | Sublin<br>ite Sul<br>(N=X | bjects |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Event | S | | | | | | | | | | | | | | | | | | | | | | | | |
| All | All | X | X | X | X | x | X | X | x | X | X | x | X | x | X | X | X | X | X | X | X | X | X | X | X |
| PT1 | SOC1 | X | X | X | X | x | х | Х | x | X | X | x | X | х | X | X | х | X | X | X | X | х | X | X | X |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | | | | | | | |
| Other (Non-serious) Ad | dverse Events | | | | | | | | | | | | | | | | | | | | | | | | |
| All | All | X | X | X | X | х | Х | X | х | Х | X | х | X | х | X | X | х | x | X | X | X | х | X | x | X |
| PT1 | SOC1 | X | X | X | X | Х | X | X | X | Х | X | х | X | X | X | X | X | X | X | X | X | X | X | х | X |
| Etc. | Etc. | | | | | | | | | | | | | | | | | | | | | | | | |

N = number of subjects in the Safety Population (number of subjects at risk).

Events= total frequency of events reported.

Tables with similar format:

Table 94: Adverse Events Occurring in 5% of Subjects in Any Treatment Group by MedDRA System Organ Class and Preferred Term, and Treatment Group – Intradermal & Pooled Cohorts

[Implementation note: Treatment groups are Cohort E: Intradermal 0.3  $\mu$ g dmLT (N=X), Cohort E: Intradermal Placebo (N=X), and All Intradermal Route Subjects (N=X). All Subjects (N=X) will be added at the end.]

Table 95: Serious Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Oral & Sublingual Cohorts

Table 96: Serious Adverse Events by MedDRA System Organ Class and Preferred Term, and Treatment Group – Intradermal & Pooled Cohorts

[Implementation note: Treatment groups are Cohort E: Intradermal 0.3  $\mu$ g dmLT (N=X), Cohort E: Intradermal Placebo (N=X), and All Intradermal Route Subjects (N=X). All Subjects (N=X) will be added at the end.]

n= number of subjects reporting event.

#### 14.3.1.1 Solicited Adverse Events

Table 97: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort A: Oral 5 µg dmLT

| | | Post Dose 1<br>(N=X) | | | Post Dose 2<br>(N=X) | | | Post Dose 3<br>(N=X) | | | Post Any Dose (N=X) | e |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | х | xx | x.x, x.x | х | xx | x.x, x.x | х | XX | x.x, x.x | х | xx | x.x, x.x |
| Any Systemic Symptom | | | | | | | | | | | | |
| Fever | | | | | | | | | | | | |
| Feverishness | | | | | | | | | | | | |
| Fatigue | | | | | | | | | | | | |
| Malaise | | | | | | | | | | | | |
| Myalgia | | | | | | | | | | | | |
| Headache | | | | | | | | | | | | |
| Any Local Symptom | | | | | | | | | | | | |
| Irritation of the Oral<br>Cavity or Tongue | | | | | | | | | | | | |
| Diarrhea | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | |
| Abdominal Discomfort | | | | | | | | | | | | |

Note: N=Number of subjects in the Safety Population

Tables with similar format:

Table 98: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort B: Oral 25 μg dmLT

Table 99: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – All Oral Cohorts: Placebo

### Table 100: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort C: Sublingual 5 µg dmLT

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

### Table 101: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort D: Sublingual 25 µg dmLT

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

# Table 102: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – All Sublingual Cohorts: Placebo

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

## Table 103: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort Ε: Intradermal 0.3 μg dmLT

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

### Table 104: Number and Percentage of Subjects Experiencing Solicited Events with 95% Confidence Intervals by Symptom, Dose, and Treatment Group – Cohort E: Intradermal Placebo

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

Table 105: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort A: Oral 5 μg dmLT

| | | | Post Dose | 1 | | Post Dose 2 | , | | Post Dose 3 | | | Post Any Dos | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | (N=X) | L | | (N=X) | 4 | | (N=X) | | | (N=X) | е |
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Any Symptom | None | X | xx | x.x, x.x | X | XX | x.x, x.x | X | xx | X.X, X.X | X | XX | x.x, x.x |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Systemic Symp | toms | | | | | | | | | _ | | | |
| Any Systemic<br>Symptom | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Malaise | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |

| | | | Post Dose 1<br>(N=X) | | | Post Dose 2<br>(N=X) | | | Post Dose 3<br>(N=X) | | | Post Any Dos<br>(N=X) | e |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| <b>Local Symptom</b> | S | | | | | | | | | | | | |
| Any Local<br>Symptom | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Irritation of the<br>Oral Cavity or<br>Tongue | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Diarrhea | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |

| | | | Post Dose 1 (N=X) | I | | Post Dose 2<br>(N=X) | | | Post Dose 3<br>(N=X) | 3 | | Post Any Do<br>(N=X) | se |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI | n | % | 95% CI |
| Nausea | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Vomiting | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | |
| Abdominal<br>Discomfort | None | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | |
| N. M. M. | Severe | | | | | | | | | | . 1 | | |

Note: N = Number of subjects in the Safety Population who received the specified dose. Severity is the maximum severity reported over all solicited symptoms post dosing for each subject.

Tables with similar format:

- Table 106: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose Cohort B: Oral 25 μg dmLT
- Table 107: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose All Oral Cohorts: Placebo
- Table 108: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose Cohort C: Sublingual 5 µg dmLT

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

Table 109: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort D: Sublingual 25 µg dmLT

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

### Table 110: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – All Sublingual Cohorts: Placebo

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

### Table 111: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort E: Intradermal 0.3 µg dmLT

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

### Table 112: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Maximum Severity, Dose – Cohort E: Intradermal Placebo

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

Table 113: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort A: Oral 5 µg dmLT, Dose 1

| | | Pre- | Dose | Post- | -Dose | Da | y 1 | Da | ıy 2 | Da | ıy 3 | Da | ıy 4 | Da | ıy 5 | Da | ıy 6 | Da | ıy 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any<br>Symptom | None | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx | х | xx |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Systemic Sym | ptoms | | • | • | • | | • | • | • | | • | • | • | • | • | | • | • | |
| Any<br>Systemic<br>Symptom | None | х | xx | х | xx | x | xx | х | xx | х | xx | х | xx | x | xx | х | xx | X | xx |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Fever | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Feverishness | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Fatigue | None | | | | | | | | | | | | | | | | | | |

| | | Pre- | -Dose | Post- | -Dose | Da | ny 1 | Da | y 2 | Da | y 3 | Da | ıy 4 | Da | ıy 5 | Da | ny 6 | Da | ny 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Malaise | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Myalgia | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Headache | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Local Sympto | oms | | | | | | | | | | | | | | | | | | |
| Any Local<br>Symptom | None | x | xx | x | xx | x | xx | x | xx | х | xx | x | xx | x | xx | x | xx | x | xx |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |

| | | Pre- | Dose | Post- | -Dose | Da | ay 1 | Da | y 2 | Da | y 3 | Da | ıy 4 | Da | y 5 | Da | ıy 6 | Da | y 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Irritation of<br>the Oral<br>Cavity or<br>Tongue | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Diarrhea | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Nausea | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Vomiting | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |
| Abdominal<br>Discomfort | None | | | | | | | | | | | | | | | | | | |
| | Mild | | | | | | | | | | | | | | | | | | |
| | Moderate | | | | | | | | | | | | | | | | | | |

| | | Pre-Dose | | Post- | Dose | Da | y 1 | Da | y 2 | Da | y 3 | Da | y 4 | Da | y 5 | Da | y 6 | Da | y 7 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Severe | | | | | | | | | | | | | | | | | | |
| | Not Reported | | | | | | | | | | | | | | | | | | |

Note: N = Number of subjects in the Safety Population who received the specified dose. Severity is the maximum severity reported post dosing for each subject for each day.

#### Tables with similar format:

- Table 114: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group Cohort A: Oral 5 µg dmLT, Dose 2
- Table 115: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group Cohort A: Oral 5 µg dmLT, Dose 3
- Table 116: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group Cohort B: Oral 25 μg dmLT, Dose 1
- Table 117: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group Cohort B: Oral 25 µg dmLT, Dose 2
- Table 118: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group Cohort B: Oral 25 μg dmLT, Dose 3
- Table 119: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group All Oral Cohorts: Placebo, Dose 1
- Table 120: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group All Oral Cohorts: Placebo, Dose 2
- Table 121: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group All Oral Cohorts: Placebo, Dose 3
- Table 122: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group Cohort C: Sublingual 5 μg dmLT, Dose 1

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

### Table 123: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort C: Sublingual 5 μg dmLT, Dose 2

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

Table 124: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort C: Sublingual 5 μg dmLT, Dose 3

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

Table 125: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort D: Sublingual 25 μg dmLT, Dose 1

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

Table 126: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort D: Sublingual 25 μg dmLT, Dose 2

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

Table 127: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort D: Sublingual 25 μg dmLT, Dose 3

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

Table 128: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Sublingual Cohorts: Placebo Dose 1

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

Table 129: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Sublingual Cohorts: Placebo, Dose 2

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

### Table 130: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – All Sublingual Cohorts: Placebo, Dose 3

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, or headache. Local symptoms presented will be irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.]

## Table 131: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal 0.3 µg dmLT, Dose 1

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

## Table 132: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal 0.3 µg dmLT, Dose 2

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

### Table 133: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal Placebo, Dose 1

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

### Table 134: Number and Percentage of Subjects Experiencing Solicited Events by Symptom, Severity, Dose, Day Post Dosing, and Treatment Group – Cohort E: Intradermal Placebo, Dose 2

[Implementation note: Systemic symptoms presented will be fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort. Local symptoms presented will be injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles or hardened mass.]

Table 135: Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 2 by Treatment Group

| Treatment Group | | Dose 2 – Subjects with No<br>Symptoms | Dose 2 – Subjects with Mild<br>or Greater Symptoms | Dose 2 – Total Number of<br>Subjects |
|---|---|---|---|---|
| Systemic Symptoms | | · | | |
| Cohort A: Oral 5 µg dmLT | Dose 1 Subject with No Symptoms | x (%) | x (%) | x (%) |
| | Dose 1 Subjects with Mild or Greater Symptoms | x (%) | x (%) | x (%) |
| | Dose 1 Total Number of Subjects | x (%) | x (%) | x (100%) |
| Cohort B: Oral 25 µg dmLT | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| All Oral Cohorts: Placebo | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort C: Sublingual 5 μg dmLT | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort D: Sublingual 25 µg dmLT | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| All Sublingual Cohorts: Placebo | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort E: Intradermal 5 µg dmLT | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort E: Intradermal Placebo | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |

| Treatment Group | | Dose 2 – Subjects with No<br>Symptoms | Dose 2 – Subjects with Mild<br>or Greater Symptoms | Dose 2 – Total Number of<br>Subjects |
|---|---|---|---|---|
| Local Symptoms | | | | |
| Cohort A: Oral 5 µg dmLT | Dose 1 Subjects with No Symptoms | x (%) | x (%) | х (%) |
| | Dose 1 Subjects with Mild or Greater Symptoms | x (%) | x (%) | х (%) |
| | Dose 1 Total Number of Subjects | x (%) | x (%) | x (100%) |
| Cohort B: Oral 25 μg dmLT | Dose 1 Subjects with No Symptoms | | x (%) x (%) x (%) x (%) | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| All Oral Cohorts: Placebo | Dose 1 Subjects with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort C: Sublingual 5 µg dmLT | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort D: Sublingual 25 µg dmLT | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| All Sublingual Cohorts: Placebo | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort E: Intradermal 5 µg dmLT | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |
| Cohort E: Intradermal Placebo | Dose 1 Subject with No Symptoms | | | |
| | Dose 1 Subjects with Mild or Greater Symptoms | | | |
| | Dose 1 Total Number of Subjects | | | |

Note: Denominators for percentages are the number of subjects in the Safety Population who received the first and second dose. [x] subjects did not get the second dose and are not included in this table.

#### Table 136: Number and Percentage of Subjects Experiencing Solicited Events for Dose 1 Compared with Dose 3 by Treatment Group

[Implementation note: Footnote will be "Note: Denominators for percentages are the number of subjects in the Safety Population who received the first and third dose. [x] subjects did not get the third dose and are not included in this table."]

#### Table 137: Number and Percentage of Subjects Experiencing Solicited Events for Dose 2 Compared with Dose 3 by Treatment Group

[Implementation note: Footnote will be "Note: Denominators for percentages are the number of subjects in the Safety Population who received the second and third dose. [x] subjects did not get the third dose and are not included in this table."]

#### 14.3.1.2 Unsolicited Adverse Events

### 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

### **Table 138:** Listing of Serious Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | No. of Days<br>Post Dose<br>the Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Subject ID: , Treatment Group: , AE Number: | | | | | | | | | | | |
| | | T | | | | | | T | | | | |
| Comments: | Comments: | | | | | | | | | | | |
| Subject ID | Subject ID: , Treatment Group: , AE Number: | | | | | | | | | | | |
| Comments: | Comments: | | | | | | | | | | | |

#### Table 139: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days<br>Post<br>Associated<br>Dose<br>(Duration) | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID: , Tr | Subject ID: , Treatment Group: , AE Number: | | | | | | | | | |
| | T | | | | T | | T | | | |
| Comments: | Comments: | | | | | | | | | |
| Subject ID: , Tr | eatment Group:, | AE Number: | | | | | | | | |
| Comments: | , | | | | | | | | | |

### 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

(not included in SAP, but this is a placeholder for the CSR)

### 14.3.4 Abnormal Laboratory Value Listings (by Subject)

### Table 140: Listing of Abnormal Laboratory Results - Chemistry

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued Due<br>to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|
Table 141:
 Listing of Abnormal Laboratory Results - Hematology

| Subject<br>ID | Treatment<br>Group | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Action Taken<br>with Study<br>Treatment | Subject<br>Discontinued Due<br>to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

## 14.3.5 Displays of Laboratory Results

## 14.3.5.1 Chemistry Results

Table 142: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Chemistry Parameter

| | | | No | one | | ild /<br>ade 1 | l l | erate/<br>ide 2 | | ere/<br>ide 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 μg dmLT | х | х | XX | х | xx | x | xx | х | xx | х | xx |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 7 Days Post-<br>Dose 3 <sup>a</sup> | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual Placebo | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort. Albumin was not evaluated at this visit.

<sup>&</sup>lt;sup>b</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

Table 143: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Creatinine

| | | | No | one | | ild/<br>ade 1 | | lerate/<br>ade 2 | | rere/ | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 μg dmLT | х | х | xx | х | xx | х | xx | х | XX | х | xx |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 7 Days Post-<br>Dose 3 <sup>a</sup> | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual Placebo | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 36 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>b</sup> Day 57 for Oral & Sublingual Cohorts

Table 144: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Alanine Aminotransferase

| | | | No | one | | ild/<br>ide 1 | | erate/<br>ide 2 | | vere/<br>ade 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | Х | х | xx | X | xx | X | XX | X | xx | х | XX |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 7 Days Post-Dose 3 <sup>a</sup> | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual Placebo | | | | | | | | | | | |
| 28 Days Post-Dose 3 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity Post Baseline | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 36 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>b</sup> Day 57 for Oral & Sublingual Cohorts

Table 145: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Albumin

| | | | N | one | | ild/<br>ade 1 | | erate/<br>ide 2 | | vere/<br>ide 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 μg dmLT | Х | Х | xx | х | XX | х | XX | х | XX | х | xx |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Table 146: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Total Bilirubin

| | | No | one | | | | | | | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Cohort A: Oral 5 µg dmLT | X | x | XX | X | XX | X | xx | x | XX | X | XX |
| Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| All Oral Cohorts: Placebo | | | | | | | | | | | |
| Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| Cohort E: Intradermal Placebo | | | | | | | | | | | |
| Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| All Oral Cohorts: Placebo | | | | | | | | | | | |
| Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| All Oral Cohorts: Placebo | | | | | | | | | | | |
| Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| Cohort E: Intradermal Placebo | | | | | | | | | | | |
| | Cohort A: Oral 5 µg dmLT Cohort B: Oral 25 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT Cohort D: Sublingual 25 µg dmLT All Sublingual Cohorts: Placebo Cohort E: Intradermal 0.3 µg dmLT Cohort B: Oral 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort D: Sublingual 5 µg dmLT All Sublingual Cohorts: Placebo Cohort A: Oral 5 µg dmLT All Sublingual Cohorts: Placebo Cohort C: Sublingual 25 µg dmLT All Oral Cohorts: Placebo Cohort A: Oral 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort D: Sublingual 25 µg dmLT All Sublingual Cohorts: Placebo Cohort E: Intradermal 0.3 µg dmLT | Cohort A: Oral 5 µg dmLT Cohort B: Oral 25 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT Cohort D: Sublingual 25 µg dmLT All Sublingual Cohorts: Placebo Cohort E: Intradermal 0.3 µg dmLT Cohort B: Oral 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort D: Sublingual 5 µg dmLT All Sublingual Cohorts: Placebo Cohort A: Oral 5 µg dmLT All Sublingual Cohorts: Placebo Cohort C: Sublingual 25 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 µg dmLT All Sublingual Cohorts: Placebo Cohort D: Sublingual 25 µg dmLT All Sublingual Cohorts: Placebo Cohort E: Intradermal 0.3 µg dmLT | Treatment Group Cohort A: Oral 5 μg dmLT X X Cohort B: Oral 25 μg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 μg dmLT All Sublingual Cohorts: Placebo Cohort E: Intradermal 0.3 μg dmLT Cohort B: Oral 25 μg dmLT Cohort B: Oral 25 μg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 μg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 μg dmLT All Oral Cohorts: Placebo Cohort A: Oral 5 μg dmLT All Sublingual Cohorts: Placebo Cohort C: Sublingual 25 μg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 μg dmLT Cohort D: Sublingual 5 μg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 μg dmLT All Oral Cohorts: Placebo Cohort C: Sublingual 5 μg dmLT All Oral Cohorts: Placebo Cohort D: Sublingual 25 μg dmLT All Sublingual Cohorts: Placebo Cohort D: Sublingual 25 μg dmLT All Sublingual Cohorts: Placebo Cohort E: Intradermal 0.3 μg dmLT | Cohort A: Oral 5 µg dmLT | Treatment Group N N N N N N N N N N N N N | Treatment Group N N N N N N N N N N N N N | Treatment Group N N N N N N N N N N N N N | Treatment Group N N N N N N N N N N N N N | Treatment Group N N N N N N N N N N N N N | None Grade 1 Grade 2 Grade 3 | None Grade 1 Grade 2 Grade 3 Miss |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group -**Table 147:** Creatinine (µmol/L)

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 μg dmLT | X | xx.x | XX.X | XX.X | xx.x, xx.x |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 7 Days Post-Dose 3 <sup>a</sup> | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | Cohort D: Sublingual Placebo | | | | | |
| 7 Days Post-Dose 3 <sup>a</sup> ,<br>Change from Baseline | Cohort D: Sublingual 25 μg dmLT | | | | | |
| | Cohort D: Sublingual Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>b</sup> | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>b</sup> ,<br>Change from Baseline | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 36 for Oral & Sublingual Cohorts <sup>b</sup> Day 57 for Oral & Sublingual Cohorts

Table 148: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Alanine Aminotransferase (U/L)

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 µg dmLT | X | xx.x | XX.X | XX.X | xx.x, xx.x |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 7 Days Post-Dose 3 <sup>a</sup> | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | Cohort D: Sublingual Placebo | | | | | |
| 7 Days Post-Dose 3 <sup>a</sup> , Change from Baseline | Cohort D: Sublingual 25 μg dmLT | | | | | |
| | Cohort D: Sublingual Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>b</sup> ,<br>Change from Baseline | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 36 for Oral & Sublingual Cohorts; Day 50 for Intradermal Cohort

<sup>&</sup>lt;sup>b</sup> Day 57 for Oral & Sublingual Cohorts; Day 71 for Intradermal Cohort

Table 149: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Albumin (g/dL)

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 µg dmLT | X | xx.x | XX.X | XX.X | xx.x, xx.x |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> ,<br>Change from Baseline | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Table 150: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Total Bilirubin ( $\mu mol/L$ )

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 µg dmLT | X | xx.x | XX.X | XX.X | xx.x, xx.x |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 µg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> ,<br>Change from Baseline | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

## 14.3.5.2 Hematology Results

Table 151: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Any Hematology Parameter

| Any Hematology<br>Parameter | | | N | one | | ild /<br>ade 1 | | erate/<br>ide 2 | | ere/<br>ide 3 | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | X | х | XX | х | xx | х | xx | х | xx | х | XX |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity Post<br>Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Table 152: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – White Blood Cell Count

| | | | No | one | Gr | ild/<br>ade<br>1<br>ow) | Gr | ild/<br>ade<br>1<br>igh) | Gra | erate/<br>ide 2<br>ow) | Gra | erate/<br>ide 2<br>igh) | Gra | rere/<br>ide 3<br>ow) | Gra | ere/<br>de 3 | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | х | х | xx | Х | xx | X | XX | Х | XX | Х | xx | х | xx | х | xx | х | xx |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| 28 Days<br>Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| Max<br>Severity Post<br>Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Table 153: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Absolute Neutrophil Count

| | | | No | one | | ild/<br>ide 1 | | erate/<br>ide 2 | | rere/<br>ide 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | х | x | xx | х | xx | x | XX | х | XX | x | xx |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

**Table 154:** Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group - Hemoglobin

| | | | No | one | | ild/<br>ade 1 | | lerate/<br>ade 2 | | vere/<br>ade 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 μg dmLT | х | х | XX | х | XX | X | xx | Х | xx | х | XX |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>a</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments. N=Number of subjects in the Safety Population <sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Table 155: Laboratory Results by Parameter, Maximum Severity, Time Point, and Treatment Group – Platelets

| | | | No | one | | ild/<br>ide 1 | l l | erate/<br>ide 2 | | vere/<br>ide 3 | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | X | X | XX | X | XX | Х | XX | X | XX | X | xx |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group -**Table 156:** White Blood Cell Count (109/L)

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 μg dmLT | X | xx.x | XX.X | XX.X | xx.x, xx.x |
| | Cohort B: Oral 25 μg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | |
| 20 24,01 000 2000 | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> ,<br>Change from Baseline | Cohort A: Oral 5 µg dmLT | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

Note: N = Number of subjects in the Safety Population <sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Table 157: Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group – Absolute Neutrophil Count (109/L)

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 µg dmLT | X | xx.x | XX.X | xx.x | xx.x, xx.x |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 µg dmLT | | | | | |
| 20 24,01000 2000 0 | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> ,<br>Change from Baseline | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group -**Table 158:** Hemoglobin (mg/dL)

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 μg dmLT | X | xx.x | XX.X | XX.X | xx.x, xx.x |
| | Cohort B: Oral 25 μg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 µg dmLT | | | | | |
| 20 Buyo 1 oot Bose 5 | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> ,<br>Change from Baseline | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

Note: N = Number of subjects in the Safety Population <sup>a</sup> Day 57 for Oral & Sublingual Cohorts

Laboratory Summary Statistics by Parameter, Time Point, and Treatment Group -**Table 159:** Platelets (10<sup>9</sup>/L)

| Time Point | Treatment Group | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | Cohort A: Oral 5 μg dmLT | X | xx.x | XX.X | XX.X | xx.x, xx.x |
| | Cohort B: Oral 25 μg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | |
| | Cohort E: Intradermal Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> | Cohort A: Oral 5 µg dmLT | | | | | |
| 20 Days 1 03t D030 3 | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |
| 28 Days Post-Dose 3 <sup>a</sup> ,<br>Change from Baseline | Cohort A: Oral 5 μg dmLT | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | |
| | All Oral Cohorts: Placebo | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | |

Note: N = Number of subjects in the Safety Population <sup>a</sup> Day 57 for Oral & Sublingual Cohorts

## 14.3.6 Displays of Vital Signs

Table 160: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Any Assessment

| | | | No | one | M | ild | Mod | erate | Sev | ere | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 μg dmLT | х | Х | XX | х | XX | Х | XX | X | XX | Х | XX |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 7 Days Post-Dose 1 <sup>a</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| Dose 2 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 7 Days Post-Dose 2 <sup>c</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |

| | | | No | one | M | ild | Mod | erate | Sev | ere | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| Dose 3 <sup>d</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| 7 Days Post-Dose 3 <sup>e</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| 28 Days Post-Dose 3 <sup>f</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| 85 Days Post-Dose 3g | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | |
| 180 Days Post-Dose 3h | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | |
| Max Severity Post Baseline | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |

| | | | No | ne | M | ild | Mod | erate | Sev | ere | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 29 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>f</sup> Day 57 for Oral & Sublingual Cohorts

g Day 114 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>h</sup> Day 209 for Oral & Sublingual Cohorts

Table 161: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Temperature

| | | | No | one | M | ild | Mod | lerate | Sev | ere | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 μg dmLT | X | х | XX | х | XX | х | XX | х | XX | х | xx |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 7 Days Post-<br>Dose 1 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| Dose 2 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| 7 Days Post-<br>Dose 2 <sup>c</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |
| Dose 3 <sup>d</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |

| | | | N | one | М | ild | Mod | lerate | Sev | ere | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| 7 Days Post-<br>Dose 3 <sup>e</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>f</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |
| 85 Days Post-<br>Dose 3 <sup>g</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | |
| 180 Days<br>Post-Dose 3 <sup>h</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | |

| | | | No | ne | M | ild | Mod | erate | Sev | ere | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | |

<sup>&</sup>lt;sup>a</sup> Day 8

<sup>&</sup>lt;sup>b</sup> Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort

<sup>&</sup>lt;sup>c</sup> Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort

<sup>&</sup>lt;sup>d</sup> Day 29 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>e</sup> Day 36 for Oral & Sublingual Cohorts

f Day 57 for Oral & Sublingual Cohorts g Day 114 for Oral & Sublingual Cohorts

h Day 209 for Oral & Sublingual Cohorts

Table 162: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Pulse

| | | | No | one | | ild<br>ow) | | ild<br>igh) | | lerate<br>ow) | | erate<br>igh) | | vere<br>ow) | | vere<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | х | X | XX | Х | XX | Х | xx | Х | xx | Х | XX | X | XX | Х | XX | х | XX |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 1 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| Dose 2 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 μg dmLT | | | | | | | | | | | | | | | | | |

| | | | No | one | 1 | ild<br>ow) | I | ild<br>igh) | | lerate<br>ow) | | erate<br>gh) | | vere<br>ow) | | vere<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 2 <sup>c</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| Dose 3 <sup>d</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 3 <sup>e</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>f</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | _ | | | | | | | | | | | | | | | |

| | | | No | one | | ild<br>ow) | | ild<br>igh) | | lerate<br>ow) | | erate<br>gh) | Sev<br>(Lo | ere<br>ow) | | vere<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 85 Days Post-<br>Dose 3 <sup>g</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | | | | | | | |
| 180 Days Post-<br>Dose 3 <sup>h</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |

| | | | No | one | | ild<br>ow) | (Hi | ild<br>gh) | | erate<br>ow) | | erate<br>gh) | Sev<br>(Lo | | (Hi | ere<br>gh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

<sup>&</sup>lt;sup>a</sup> Day 8

b Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort
Capay 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort
Day 29 for Oral & Sublingual Cohorts
Day 36 for Oral & Sublingual Cohorts

f Day 57 for Oral & Sublingual Cohorts

g Day 114 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>h</sup> Day 209 for Oral & Sublingual Cohorts

Table 163: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Systolic Blood Pressure

| | | | No | one | | (ild<br>ow) | | ild<br>igh) | | lerate<br>ow) | | erate<br>igh) | | vere<br>ow) | | vere<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | х | х | XX | X | XX | х | XX | X | XX | X | XX | X | XX | X | XX | х | xx |
| | Cohort B: Oral 25 μg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 1 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| Dose 2 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |

| | | | No | one | | ild<br>ow) | | ild<br>igh) | | erate<br>ow) | | erate<br>gh) | | vere<br>ow) | | vere<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 2 <sup>c</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| Dose 3 <sup>d</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 3 <sup>e</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>f</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |

| | | | No | one | | ild<br>ow) | | ild<br>igh) | | erate<br>ow) | | erate<br>gh) | | vere<br>ow) | | vere<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 85 Days Post-<br>Dose 3 <sup>g</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | | | | | | | |
| 180 Days<br>Post-Dose 3 <sup>h</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |

| | | | No | one | Mi<br>(Lo | | | ild<br>gh) | Mod<br>(Lo | erate<br>ow) | Mod<br>(Hi | erate<br>gh) | Sev<br>(Lo | | (Hi | ere<br>(gh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

N = Number of subjects in the Safety Population.

<sup>a</sup> Day 8

b Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort
c Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort
d Day 29 for Oral & Sublingual Cohorts
c Day 36 for Oral & Sublingual Cohorts

f Day 57 for Oral & Sublingual Cohorts

g Day 114 for Oral & Sublingual Cohorts

<sup>h</sup> Day 209 for Oral & Sublingual Cohorts

Table 164: Vital Signs by Assessment, Maximum Severity, Time Point, and Treatment Group – Diastolic Blood Pressure

| | | | N | one | | ild<br>ow) | | lild<br>igh) | | lerate<br>ow) | | lerate<br>igh) | | vere<br>ow) | | vere<br>igh) | Mis | ssing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Baseline | Cohort A: Oral 5 µg dmLT | X | Х | XX | X | XX | х | xx | х | xx | X | XX | X | xx | X | xx | х | XX |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 1 <sup>a</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| Dose 2 <sup>b</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 μg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |

| | | | No | one | | ild<br>ow) | M<br>(Hi | | | erate<br>ow) | | erate<br>igh) | | vere<br>ow) | | vere<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 2 <sup>c</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| Dose 3 <sup>d</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 7 Days Post-<br>Dose 3 <sup>e</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 28 Days Post-<br>Dose 3 <sup>f</sup> | Cohort A: Oral 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | _ | | | | | | | | | | | | | | | |

| | | | No | one | | ild<br>ow) | M<br>(Hi | | | erate<br>ow) | Mod<br>(Hi | erate<br>gh) | | vere<br>ow) | | ere<br>igh) | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Treatment Group | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| 85 Days Post-<br>Dose 3 <sup>g</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | | | | | | | |
| 180 Days Post-<br>Dose 3 <sup>h</sup> | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual Placebo | | | | | | | | | | | | | | | | | |
| Max Severity<br>Post Baseline | Cohort A: Oral 5 μg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort B: Oral 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Oral Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort C: Sublingual 5 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort D: Sublingual 25 µg dmLT | | | | | | | | | | | | | | | | | |
| | All Sublingual Cohorts: Placebo | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal 0.3 µg dmLT | | | | | | | | | | | | | | | | | |
| | Cohort E: Intradermal Placebo | | | | | | | | | | | | | | | | | |
| | | | No | one | M<br>(Lo | ild<br>ow) | M<br>(Hi | ild<br>gh) | | erate<br>ow) | | erate<br>igh) | | vere<br>Ow) | Sev<br>(Hi | | Mis | sing |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | <b>Treatment Group</b> | N | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |

Note: The "Max Post Baseline" rows indicate the maximum severity experienced by each subject at any time point post baseline, including unscheduled assessments.

N = Number of subjects in the Safety Population.

<sup>&</sup>lt;sup>a</sup> Day 8

b Day 15 for Oral & Sublingual Cohorts; Day 22 for Intradermal Cohort
c Day 22 for Oral & Sublingual Cohorts; Day 29 for Intradermal Cohort
d Day 29 for Oral & Sublingual Cohorts
c Day 36 for Oral & Sublingual Cohorts

f Day 57 for Oral & Sublingual Cohorts

g Day 114 for Oral & Sublingual Cohorts

<sup>&</sup>lt;sup>h</sup> Day 209 for Oral & Sublingual Cohorts

#### **APPENDIX 2. FIGURE MOCK-UPS**

#### LIST OF FIGURES

| Figure 1: | CONSORT Flow Diagram – Oral Cohorts | 263 |
|---|---|---|
| Figure 2: | CONSORT Flow Diagram – Sublingual Cohorts | 264 |
| Figure 3: | CONSORT Flow Diagram – Intradermal Cohort | 265 |
| Figure 4: | Serum IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 266 |
| Figure 5: | Serum IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 267 |
| Figure 6: | Serum IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population. | 267 |
| Figure 7: | Serum IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 267 |
| Figure 8: | Serum IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population | 267 |
| Figure 9: | Serum IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 267 |
| Figure 10: | Serum IgG Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 267 |
| Figure 11: | Serum IgG Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 267 |
| Figure 12: | Serum IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population, mITT Population | 267 |
| Figure 13: | Serum IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 268 |
| Figure 14: | Serum IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population | 268 |
| Figure 15: | Serum IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 268 |
| Figure 16: | Serum LT Neutralization Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 268 |
| Figure 17: | Serum LT Neutralization Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 268 |

| Figure 18: | Serum LT Neutralization Log-Titer over Time by Treatment Group – Sublingual, mITT Population Cohorts | 268 |
|---|---|---|
| Figure 19: | Serum LT Neutralization Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 268 |
| Figure 20: | Serum LT Neutralization Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population | 268 |
| Figure 21: | Serum LT Neutralization Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 268 |
| Figure 22: | ALS IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 269 |
| Figure 23: | ALS IgA Log-Titer over Time by Treatment Group – Oral Cohort, Per Protocol Population | 269 |
| Figure 24: | ALS IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population | 269 |
| Figure 25: | ALS IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 269 |
| Figure 26: | ALS IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population | 269 |
| Figure 27: | ALS IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 269 |
| Figure 28: | ALS IgG Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 269 |
| Figure 29: | ALS IgG Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 269 |
| Figure 30: | ALS IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population. | 269 |
| Figure 31: | ALS IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 270 |
| Figure 32: | ALS IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population. | 270 |
| Figure 33: | ALS IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | |
| Figure 34: | Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 270 |
| Figure 35: | Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population | |
| Figure 36: | Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population | |

| Figure 37: | Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 270 |
|---|---|---|
| Figure 38: | Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population | 270 |
| Figure 39: | Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 270 |
| Figure 40: | Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 271 |
| Figure 41: | Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 271 |
| Figure 42: | Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population | 271 |
| Figure 43: | Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 271 |
| Figure 44: | Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population | 271 |
| Figure 45: | Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 271 |
| Figure 46: | Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 271 |
| Figure 47: | Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 271 |
| Figure 48: | Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population | 271 |
| Figure 49: | Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 272 |
| Figure 50: | Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population | 272 |
| Figure 51: | Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 272 |
| Figure 52: | Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population | 272 |
| Figure 53: | Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment<br>Group – Oral Cohorts, Per Protocol Population | 272 |
| Figure 54: | Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment<br>Group – Sublingual Cohorts, mITT Population | 272 |
| Figure 55: | Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment<br>Group – Sublingual Cohorts, Per Protocol Population | 272 |

| Figure 56: | Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment<br>Group – Intradermal Cohort, mITT Population | 272 |
|---|---|---|
| Figure 57: | Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment<br>Group – Intradermal Cohort, Per Protocol Population | 272 |
| Figure 58: | Serum IgA Fold-Rise over Time by Treatment Group- Oral Cohorts, mITT Population | 273 |
| Figure 59: | Serum IgA Fold-Rise over Time by Treatment Group- Oral Cohorts, Per<br>Protocol Population | 274 |
| Figure 60: | Serum IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 274 |
| Figure 61: | Serum IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 274 |
| Figure 62: | Serum IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 274 |
| Figure 63: | Serum IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 274 |
| Figure 64: | Serum IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population | 274 |
| Figure 65: | Serum IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 274 |
| Figure 66: | Serum IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 274 |
| Figure 67: | Serum IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 275 |
| Figure 68: | Serum IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population. | 275 |
| Figure 69: | Serum IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 275 |
| Figure 70: | Serum LT Neutralization Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population | 275 |
| Figure 71: | Serum LT Neutralization Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 275 |
| Figure 72: | Serum LT Neutralization Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 275 |
| Figure 73: | • | |
| Figure 74: | Serum LT Neutralization Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | |

| Figure 75: | Serum LT Neutralization Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 275 |
|---|---|---|
| Figure 76: | ALS IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population | 276 |
| Figure 77: | ALS IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 276 |
| Figure 78: | ALS IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 276 |
| Figure 79: | ALS IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 276 |
| Figure 80: | ALS IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 276 |
| Figure 81: | ALS IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 276 |
| Figure 82: | ALS IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population | 276 |
| Figure 83: | ALS IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 276 |
| Figure 84: | ALS IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 276 |
| Figure 85: | ALS IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 277 |
| Figure 86: | ALS IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 277 |
| Figure 87: | ALS IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 277 |
| Figure 88: | Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population | 277 |
| Figure 89: | Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 277 |
| Figure 90: | Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 277 |
| Figure 91: | Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | |
| Figure 92: | Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | |
| Figure 93: | Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | |

| Figure 94: | Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group — Oral Cohorts, mITT Population | 278 |
|---|---|---|
| Figure 95: | Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 278 |
| Figure 96: | Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 278 |
| Figure 97: | Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group — Sublingual Cohorts, Per Protocol Population | 278 |
| Figure 98: | Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group — Intradermal Cohort, mITT Population | 278 |
| Figure 99: | Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group — Intradermal Cohort, Per Protocol Population | 278 |
| Figure 100: | Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population | 278 |
| Figure 101: | Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population | 278 |
| Figure 102: | Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 278 |
| Figure 103: | Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 279 |
| Figure 104: | Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 279 |
| Figure 105: | Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population | 279 |
| Figure 106: | Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group Oral Cohorts, mITT Population | 279 |
| Figure 107: | Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group Oral Cohorts, Per Protocol Population | 279 |
| Figure 108: | Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population | 279 |
| Figure 109: | Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population | 279 |
| Figure 110: | Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group — Intradermal Cohort, mITT Population | 279 |
| Figure 111: | Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group — Intradermal Cohort, Per Protocol Population | 279 |
| Figure 112: | T-cell Effector function - CD4/IFNg (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | |

| Figure 113: T-cell Effector function - CD4/IFNg (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | 280 |
|---|---|
| Figure 114: T-cell Effector function - CD4/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 280 |
| Figure 115: T-cell Effector function - CD4/TNFa (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 280 |
| Figure 116: T-cell Effector function - CD4/TNFa (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | 280 |
| Figure 117: T-cell Effector function - CD4/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 280 |
| Figure 118: T-cell Effector function - CD4/MIP1b (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 280 |
| Figure 119: T-cell Effector function - CD4/MIP1b (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | 280 |
| Figure 120: T-cell Effector function - CD4/MIP1b (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 281 |
| Figure 121: T-cell Effector function - CD4/CD107a (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 281 |
| Figure 122: T-cell Effector function - CD4/CD107a (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 281 |
| Figure 123: T-cell Effector function - CD4/CD107a (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 281 |
| Figure 124: T-cell Effector function - CD4/IL-2 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | |
| Figure 125: T-cell Effector function - CD4/IL-2 (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | |
| Figure 126: T-cell Effector function - CD4/IL-2 (%) Rise over Time by Treatment Group - Intradermal Cohort, mITT Population | |
| Figure 127: T-cell Effector function - CD4/IL-17A (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 281 |
| Figure 128: T-cell Effector function - CD4/IL-17A (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | |
| Figure 129: T-cell Effector function - CD4/IL-17A (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 282 |
| Figure 130: T-cell Effector function - CD4 Tem/IFNg (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | |
| Figure 131: T-cell Effector function - CD4 Tem/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | |

| | Γ-cell Effector function - CD4 Tem/IFNg (%) Rise over Time by Treatment<br>Group — Intradermal Cohort, mITT Population | 282 |
|---|---|---|
| _ | Γ-cell Effector function - CD4 Tem/TNFa (%) Rise over Time by Treatment<br>Group – Oral Cohort, mITT Population | 282 |
| _ | Γ-cell Effector function - CD4 Tem/TNFa (%) Rise over Time by Treatment<br>Group – Sublingual Cohort, mITT Population | 282 |
| • | Γ-cell Effector function - CD4 Tem/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 282 |
| _ | Γ-cell Effector function - CD4 Tem/MIP1b (%) Rise over Time by<br>Γreatment Group – Oral Cohort, mITT Population | 282 |
| | Γ-cell Effector function - CD4 Tem/MIP1b (%) Rise over Time by<br>Γreatment Group — Sublingual Cohort, mITT Population | 282 |
| _ | Γ-cell Effector function - CD4 Tem/MIP1b (%) Rise over Time by<br>Γreatment Group — Intradermal Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/CD107a (%) Rise over Time by<br>Γreatment Group – Oral Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/CD107a (%) Rise over Time by<br>Γreatment Group – Sublingual Cohort, mITT Population | 283 |
| • | Γ-cell Effector function - CD4 Tem/CD107a (%) Rise over Time by<br>Γreatment Group — Intradermal Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/IL-2 (%) Rise over Time by Treatment<br>Group – Oral Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/IL-2 (%) Rise over Time by Treatment Group — Sublingual Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/IL-17A (%) Rise over Time by<br>Freatment Group — Oral Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/IL-17A (%) Rise over Time by<br>Freatment Group – Sublingual Cohort, mITT Population | 283 |
| _ | Γ-cell Effector function - CD4 Tem/IL-17A (%) Rise over Time by<br>Freatment Group — Intradermal Cohort, mITT Population | 284 |
| _ | Γ-cell Effector function - CD8/IFNg (%) Rise over Time by Treatment<br>Group – Oral Cohort, mITT Population | 284 |
| | Γ-cell Effector function - CD8/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 284 |
| Figure 150: 7 | Γ-cell Effector function - CD8/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 284 |

| Figure 151: | T-cell Effector function - CD8/TNFa (%) Rise over Time by Treatment<br>Group - Oral Cohort, mITT Population | .284 |
|---|---|---|
| Figure 152: | T-cell Effector function - CD8/TNFa (%) Rise over Time by Treatment<br>Group - Sublingual Cohort, mITT Population | .284 |
| Figure 153: | T-cell Effector function - CD8/TNFa (%) Rise over Time by Treatment<br>Group – Intradermal Cohort, mITT Population. | .284 |
| Figure 154: | T-cell Effector function - CD8/MIP1b (%) Rise over Time by Treatment<br>Group - Oral Cohort, mITT Population | .284 |
| Figure 155: | T-cell Effector function - CD8/MIP1b (%) Rise over Time by Treatment<br>Group - Sublingual Cohort, mITT Population | .284 |
| Figure 156: | T-cell Effector function - CD8/MIP1b (%) Rise over Time by Treatment<br>Group – Intradermal Cohort, mITT Population | .285 |
| Figure 157: | T-cell Effector function - CD8/CD107a (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | .285 |
| Figure 158: | T-cell Effector function - CD8/CD107a (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | .285 |
| Figure 159: | T-cell Effector function - CD8/CD107a (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | .285 |
| Figure 160: | T-cell Effector function - CD8/IL-2 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | .285 |
| Figure 161: | T-cell Effector function - CD8/IL-2 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | .285 |
| Figure 162: | T-cell Effector function - CD8/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | .285 |
| Figure 163: | T-cell Effector function - CD8/IL-17A (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | .285 |
| Figure 164: | T-cell Effector function - CD8/IL-17A (%) Rise over Time by Treatment Group — Sublingual Cohort, mITT Population | .285 |
| Figure 165: | T-cell Effector function - CD8/IL-17A (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | .286 |
| Figure 166: | T-cell Effector function - CD8 Tem/IFNg (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | .286 |
| Figure 167: | T-cell Effector function - CD8 Tem/IFNg (%) Rise over Time by Treatment Group — Sublingual Cohort, mITT Population | .286 |
| Figure 168: | T-cell Effector function - CD8 Tem/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | .286 |
| Figure 169: | T-cell Effector function - CD8 Tem/TNFa (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | .286 |

| Figure 170: T-cell Effector function - CD8 Tem/TNFa (%) Rise over Time by Treatmen Group - Sublingual Cohort, mITT Population | t<br>286 |
|---|---|
| Figure 171: T-cell Effector function - CD8 Tem/TNFa (%) Rise over Time by Treatmen Group – Intradermal Cohort, mITT Population | |
| Figure 172: T-cell Effector function - CD8 Tem/MIP1b (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 286 |
| Figure 173: T-cell Effector function - CD8 Tem/MIP1b (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | 286 |
| Figure 174: T-cell Effector function - CD8 Tem/MIP1b (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 287 |
| Figure 175: T-cell Effector function - CD8 Tem/CD107a (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 287 |
| Figure 176: T-cell Effector function - CD8 Tem/CD107a (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 287 |
| Figure 177: T-cell Effector function - CD8 Tem/CD107a (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 287 |
| Figure 178: T-cell Effector function - CD8 Tem/IL-2 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 287 |
| Figure 179: T-cell Effector function - CD8 Tem/IL-2 (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | 287 |
| Figure 180: T-cell Effector function - CD8 Tem/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 287 |
| Figure 181: T-cell Effector function - CD8 Tem/IL-17A (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 287 |
| Figure 182: T-cell Effector function - CD8 Tem/IL-17A (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 287 |
| Figure 183: T-cell Effector function - CD8 Tem/IL-17A (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 288 |
| Figure 184: T-cell Homing - CD4/integrin a4b7 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | |
| Figure 185: T-cell Homing - CD4/integrin a4b7 (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population | |
| Figure 186: T-cell Homing - CD4/integrin a4b7 (%) Rise over Time by Treatment Group — Intradermal Cohort, mITT Population | |
| Figure 187: T-cell Homing - CD4/CCR6 (%) Rise over Time by Treatment Group – Ora Cohort, mITT Population | 1 |
| Figure 188: T-cell Homing - CD4/CCR6 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | |

| Figure 189: | T-cell Homing - CD4/CCR6 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 288 |
|---|---|---|
| Figure 190: | T-cell Homing - CD4/CCR4 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 288 |
| Figure 191: | T-cell Homing - CD4/CCR4 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 288 |
| Figure 192: | T-cell Homing - CD4/CCR4 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 289 |
| Figure 193: | T-cell Homing - CD4/CXCR3 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 289 |
| Figure 194: | T-cell Homing - CD4/CXCR3 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 289 |
| Figure 195: | T-cell Homing - CD4/CXCR3 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 289 |
| Figure 196: | T-cell Homing - CD4 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 289 |
| Figure 197: | T-cell Homing - CD4 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 289 |
| Figure 198: | T-cell Homing - CD4 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 289 |
| Figure 199: | T-cell Homing - CD8/integrin a4b7 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 289 |
| Figure 200: | T-cell Homing - CD8/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 289 |
| Figure 201: | T-cell Homing - CD8/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 290 |
| Figure 202: | T-cell Homing - CD8 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 290 |
| Figure 203: | T-cell Homing - CD8 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 290 |
| Figure 204: | T-cell Homing - CD8 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 290 |
| Figure 205: | T-cell pTfh - CD4/CXCR5 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 290 |
| Figure 206: | T-cell pTfh - CD4/CXCR5 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 290 |
| Figure 207: | T-cell pTfh - CD4/CXCR5 (%) Rise over Time by Treatment Group — Intradermal Cohort, mITT Population | 290 |

| Figure 208: | T-cell pTfh-homing - CXCR5/integrin a4b7 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 290 |
|---|---|---|
| Figure 209: | T-cell pTfh-homing - CXCR5/integrin a4b7 (%) Rise over Time by Treatment Group — Sublingual Cohort, mITT Population | 290 |
| Figure 210: | T-cell pTfh-homing - CXCR5/integrin a4b7 (%) Rise over Time by Treatment Group — Intradermal Cohort, mITT Population | 291 |
| Figure 211: | T-cell pTfh-homing - CXCR5/CCR6 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 291 |
| Figure 212: | T-cell pTfh-homing - CXCR5/CCR6 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 291 |
| Figure 213: | T-cell pTfh-homing - CXCR5/CCR6 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 291 |
| Figure 214: | T-cell pTfh-homing - CXCR5/CCR4 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 291 |
| | T-cell pTfh-homing - CXCR5/CCR4 (%) Rise over Time by Treatment Group — Sublingual Cohort, mITT Population | 291 |
| Figure 216: | T-cell pTfh-homing - CXCR5/CCR4 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 291 |
| Figure 217: | T-cell pTfh-homing - CXCR5/CXCR3 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 291 |
| Figure 218: | T-cell pTfh-homing - CXCR5/CXCR3 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 291 |
| Figure 219: | T-cell pTfh-homing - CXCR5/CXCR3 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 292 |
| Figure 220: | T-cell pTfh-effector function - CXCR5/IFNg (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population | 292 |
| Figure 221: | T-cell pTfh-effector function - CXCR5/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 292 |
| Figure 222: | T-cell pTfh-effector function - CXCR5/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 292 |
| Figure 223: | T-cell pTfh-effector function - CXCR5/TNFa (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | |
| Figure 224: | T-cell pTfh-effector function - CXCR5/TNFa (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 292 |
| Figure 225: | T-cell pTfh-effector function - CXCR5/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | |
| Figure 226: | T-cell pTfh-effector function - CXCR5/IL-2 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | |

| _ | T-cell pTfh-effector function - CXCR5/IL-2 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 292 |
|---|---|---|
| _ | T-cell pTfh-effector function - CXCR5/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 293 |
| | T-cell pTfh-effector function - CXCR5/IL-21 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 293 |
| _ | T-cell pTfh-effector function - CXCR5/IL-21 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 293 |
| _ | T-cell pTfh-effector function - CXCR5/IL-21 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 293 |
| _ | T-cell pTfh-effector function - CXCR5/CD154 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 293 |
| _ | T-cell pTfh-effector function - CXCR5/CD154 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 293 |
| _ | T-cell pTfh-effector function - CXCR5/CD154 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 293 |
| | T-cell pTfh-effector function - CXCR5/ICOS (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population | 293 |
| _ | T-cell pTfh-effector function - CXCR5/ICOS (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population | 293 |
| _ | T-cell pTfh-effector function - CXCR5/ICOS (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population | 294 |
| _ | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment - Cohort A: Oral 5 µg dmLT | 295 |
| _ | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment - Cohort B: Oral 25 μg dmLT | 296 |
| _ | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment – All Oral Cohorts: Placebo | 296 |
| _ | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment - Cohort C: Sublingual 5 μg dmLT | 296 |
| _ | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment - Cohort D: Sublingual 25 μg dmLT | 296 |
| _ | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment – All Sublingual Cohorts: Placebo | 296 |
| _ | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment –Cohort E: Intradermal 0.3 μg dmLT | 296 |
| Figure 245: | Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment – Cohort E: Intradermal Placebo | |

| Figure 246: Maximum Severity of Solicited Local Symptoms per Subject by Day Post<br>Treatment –Cohort A: Oral 5 µg dmLT | 297 |
|---|---|
| Figure 247: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment –Cohort B: Oral 25 µg dmLT | 298 |
| Figure 248: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment – All Oral Cohorts: Placebo | 298 |
| Figure 249: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment –Cohort C: Sublingual 5 µg dmLT | 298 |
| Figure 250: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment –Cohort D: Sublingual 25 µg dmLT | 298 |
| Figure 251: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment – All Sublingual Cohorts: Placebo | 298 |
| Figure 252: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment –Cohort E: Intradermal 0.3 µg dmLT | 298 |
| Figure 253: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment – Cohort E: Intradermal Placebo | 298 |
| Figure 254: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine, Oral Cohorts | 299 |
| Figure 255: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine, Sublingual Cohorts | 299 |
| Figure 256: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine, Intradermal Cohort | 299 |
| Figure 257: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Alanine Aminotransferase, Oral Cohorts | 300 |
| Figure 258: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Alanine Aminotransferase, Sublingual Cohorts | 300 |
| Figure 259: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Alanine Aminotransferase, Intradermal Cohort | 300 |
| Figure 260: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Total Bilirubin, Sublingual Cohorts | 300 |
| Figure 261: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Total Bilirubin, Intradermal Cohort | 300 |

| Figure 262: | | | Changes from Baseline by Albumin, Oral Cohorts | 300 |
|---|---|---|---|---|
| Figure 263: | | | Changes from Baseline by Albumin, Sublingual Cohorts | 300 |
| Figure 264: | | | Changes from Baseline by Albumin, Intradermal Cohort | 300 |
| Figure 265: | Laboratory Parameter | , and Treatment Group – | Changes from Baseline by<br>White Blood Cell, Oral | 300 |
| Figure 266: | Laboratory Parameter | , and Treatment Group – | Changes from Baseline by<br>White Blood Cell, Sublingual | 301 |
| Figure 267: | Laboratory Parameter | , and Treatment Group – | Changes from Baseline by<br>White Blood Cell, | 301 |
| Figure 268: | Laboratory Parameter | , and Treatment Group – | Changes from Baseline by<br>Absolute Neutrophil Count, | 301 |
| Figure 269: | Laboratory Parameter | , and Treatment Group – | Changes from Baseline by<br>Absolute Neutrophil Count, | 301 |
| Figure 270: | Laboratory Parameter | , and Treatment Group – | Changes from Baseline by<br>Absolute Neutrophil Count, | 301 |
| Figure 271: | Laboratory Parameter | , Sex, and Treatment Gro | Changes from Baseline by oup – Hemoglobin, Oral | 301 |
| Figure 272: | Laboratory Parameter | , Sex, and Treatment Gro | Changes from Baseline by pup – Hemoglobin, Sublingual | 301 |
| Figure 273: | Laboratory Parameter | , Sex, and Treatment Gro | Changes from Baseline by pup – Hemoglobin, | 301 |
| Figure 274: | | | Changes from Baseline by Platelets, Oral Cohorts | 302 |
| Figure 275: | • | | Changes from Baseline by Platelets, Sublingual Cohorts | 302 |
| Figure 276: | | | Changes from Baseline by Platelets, Intradermal Cohort | 302 |

#### 10.1 Disposition of Subjects

Figure 1: CONSORT Flow Diagram – Oral Cohorts



Figure 2: CONSORT Flow Diagram – Sublingual Cohorts



Figure 3: CONSORT Flow Diagram – Intradermal Cohort



# 14.2.2 Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point Figure 4: Serum IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: The figure below is an example only. Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]



Figures with similar format:

#### Figure 5: Serum IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 6: Serum IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 7: Serum IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 8: Serum IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 9: Serum IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

#### Figure 10: Serum IgG Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 11: Serum IgG Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 12: Serum IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 13: Serum IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 14: Serum IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 15: Serum IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 16: Serum LT Neutralization Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 17: Serum LT Neutralization Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 18: Serum LT Neutralization Log-Titer over Time by Treatment Group – Sublingual, mITT Population Cohorts

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 19: Serum LT Neutralization Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 20: Serum LT Neutralization Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 21: Serum LT Neutralization Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

#### Figure 22: ALS IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 23: ALS IgA Log-Titer over Time by Treatment Group – Oral Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 24: ALS IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 25: ALS IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 26: ALS IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 27: ALS IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

#### Figure 28: ALS IgG Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 29: ALS IgG Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 30: ALS IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 31: ALS IgG Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 32: ALS IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 33: ALS IgG Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 34: Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 35: Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 36: Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 37: Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

### Figure 38: Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 39: Fecal dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 40: Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 41: Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 42: Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 43: Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 44: Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 45: Fecal dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 46: Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 47: Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 48: Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 49: Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 50: Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT, and Cohort E: Intradermal Placebo.]

# Figure 51: Salivary dmLT-specific IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT, and Cohort E: Intradermal Placebo.]

## Figure 52: Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 53: Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 54: Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 55: Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 56: Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 57: Salivary dmLT-specific /Total IgA Log-Titer over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 1, 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

Figure 58: Serum IgA Fold-Rise over Time by Treatment Group- Oral Cohorts, mITT Population

[Implementation note: The figure below is an example only. Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]



#### Figures with similar format:

# Figure 59: Serum IgA Fold-Rise over Time by Treatment Group- Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 60: Serum IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 61: Serum IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 62: Serum IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 63: Serum IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

#### Figure 64: Serum IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 65: Serum IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 66: Serum IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 67: Serum IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 68: Serum IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 69: Serum IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 70: Serum LT Neutralization Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 71: Serum LT Neutralization Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 72: Serum LT Neutralization Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 73: Serum LT Neutralization Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, 57, and 114. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 74: Serum LT Neutralization Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 75: Serum LT Neutralization Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, 71, and 128. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

#### Figure 76: ALS IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 77: ALS IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 78: ALS IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 79: ALS IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 80: ALS IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

### Figure 81: ALS IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

#### Figure 82: ALS IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 83: ALS IgG Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 84: ALS IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 85: ALS IgG Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, and 36. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 86: ALS IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 87: ALS IgG Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, and 50. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 88: Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 89: Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 90: Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 91: Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 92: Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 93: Fecal dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 94: Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 95: Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 96: Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 97: Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 98: Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 99: Fecal dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 100: Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 101: Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 102: Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 103: Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 104: Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 105: Salivary dmLT-specific IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 106: Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 107: Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Oral Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 108: Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 109: Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Sublingual Cohorts, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 15, 22, 29, 36, and 57. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 110: Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 111: Salivary dmLT-specific/Total IgA Fold-Rise over Time by Treatment Group – Intradermal Cohort, Per Protocol Population

[Implementation note: Timepoints presented will be Study Day 8, 22, 29, 43, 50, and 71. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 112: T-cell Effector function - CD4/IFNg (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 113: T-cell Effector function - CD4/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

### Figure 114: T-cell Effector function - CD4/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 115: T-cell Effector function - CD4/TNFa (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 116: T-cell Effector function - CD4/TNFa (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

#### Figure 117: T-cell Effector function - CD4/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 118: T-cell Effector function - CD4/MIP1b (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 119: T-cell Effector function - CD4/MIP1b (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 120: T-cell Effector function - CD4/MIP1b (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 121: T-cell Effector function - CD4/CD107a (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 122: T-cell Effector function - CD4/CD107a (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

#### Figure 123: T-cell Effector function - CD4/CD107a (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 124: T-cell Effector function - CD4/IL-2 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209 Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 125: T-cell Effector function - CD4/IL-2 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 126: T-cell Effector function - CD4/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 127: T-cell Effector function - CD4/IL-17A (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 128: T-cell Effector function - CD4/IL-17A (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]
## Figure 129: T-cell Effector function - CD4/IL-17A (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 130: T-cell Effector function - CD4 Tem/IFNg (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 131: T-cell Effector function - CD4 Tem/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 132: T-cell Effector function - CD4 Tem/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 133: T-cell Effector function - CD4 Tem/TNFa (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 134: T-cell Effector function - CD4 Tem/TNFa (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 135: T-cell Effector function - CD4 Tem/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 136: T-cell Effector function - CD4 Tem/MIP1b (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 137: T-cell Effector function - CD4 Tem/MIP1b (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 138: T-cell Effector function - CD4 Tem/MIP1b (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 139: T-cell Effector function - CD4 Tem/CD107a (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 140: T-cell Effector function - CD4 Tem/CD107a (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

### Figure 141: T-cell Effector function - CD4 Tem/CD107a (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 142: T-cell Effector function - CD4 Tem/IL-2 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

### Figure 143: T-cell Effector function - CD4 Tem/IL-2 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 144: T-cell Effector function - CD4 Tem/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 145: T-cell Effector function - CD4 Tem/IL-17A (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 146: T-cell Effector function - CD4 Tem/IL-17A (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 147: T-cell Effector function - CD4 Tem/IL-17A (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 148: T-cell Effector function - CD8/IFNg (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 149: T-cell Effector function - CD8/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 150: T-cell Effector function - CD8/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 151: T-cell Effector function - CD8/TNFa (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 152: T-cell Effector function - CD8/TNFa (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 153: T-cell Effector function - CD8/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 154: T-cell Effector function - CD8/MIP1b (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209 Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 155: T-cell Effector function - CD8/MIP1b (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 156: T-cell Effector function - CD8/MIP1b (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 157: T-cell Effector function - CD8/CD107a (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 158: T-cell Effector function - CD8/CD107a (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 159: T-cell Effector function - CD8/CD107a (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 160: T-cell Effector function - CD8/IL-2 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 161: T-cell Effector function - CD8/IL-2 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 162: T-cell Effector function - CD8/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 163: T-cell Effector function - CD8/IL-17A (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 164: T-cell Effector function - CD8/IL-17A (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 165: T-cell Effector function - CD8/IL-17A (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 166: T-cell Effector function - CD8 Tem/IFNg (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 167: T-cell Effector function - CD8 Tem/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

#### Figure 168: T-cell Effector function - CD8 Tem/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 169: T-cell Effector function - CD8 Tem/TNFa (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 170: T-cell Effector function - CD8 Tem/TNFa (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 171: T-cell Effector function - CD8 Tem/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 172: T-cell Effector function - CD8 Tem/MIP1b (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 173: T-cell Effector function - CD8 Tem/MIP1b (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 174: T-cell Effector function - CD8 Tem/MIP1b (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 175: T-cell Effector function - CD8 Tem/CD107a (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 176: T-cell Effector function - CD8 Tem/CD107a (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 177: T-cell Effector function - CD8 Tem/CD107a (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 178: T-cell Effector function - CD8 Tem/IL-2 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 179: T-cell Effector function - CD8 Tem/IL-2 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 180: T-cell Effector function - CD8 Tem/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 181: T-cell Effector function - CD8 Tem/IL-17A (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 182: T-cell Effector function - CD8 Tem/IL-17A (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 183: T-cell Effector function - CD8 Tem/IL-17A (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 184: T-cell Homing - CD4/integrin a4b7 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 185: T-cell Homing - CD4/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

### Figure 186: T-cell Homing - CD4/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 187: T-cell Homing - CD4/CCR6 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 188: T-cell Homing - CD4/CCR6 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209 Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 189: T-cell Homing - CD4/CCR6 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 190: T-cell Homing - CD4/CCR4 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 191: T-cell Homing - CD4/CCR4 (%) Rise over Time by Treatment Group - Sublingual Cohort, mITT Population

## Figure 192: T-cell Homing - CD4/CCR4 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 193: T-cell Homing - CD4/CXCR3 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 194: T-cell Homing - CD4/CXCR3 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

### Figure 195: T-cell Homing - CD4/CXCR3 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 196: T-cell Homing - CD4 Tem/integrin a4b7 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

### Figure 197: T-cell Homing - CD4 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 198: T-cell Homing - CD4 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 199: T-cell Homing - CD8/integrin a4b7 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 200: T-cell Homing - CD8/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 201: T-cell Homing - CD8/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 202: T-cell Homing - CD8 Tem/integrin a4b7 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209 Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 203: T-cell Homing - CD8 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 204: T-cell Homing - CD8 Tem/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 205: T-cell pTfh - CD4/CXCR5 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 206: T-cell pTfh - CD4/CXCR5 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 207: T-cell pTfh - CD4/CXCR5 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 208: T-cell pTfh-homing - CXCR5/integrin a4b7 (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 209: T-cell pTfh-homing - CXCR5/integrin a4b7 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 210: T-cell pTfh-homing - CXCR5/integrin a4b7 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 211: T-cell pTfh-homing - CXCR5/CCR6 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209 Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 212: T-cell pTfh-homing - CXCR5/CCR6 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209 Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 213: T-cell pTfh-homing - CXCR5/CCR6 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 214: T-cell pTfh-homing - CXCR5/CCR4 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 215: T-cell pTfh-homing - CXCR5/CCR4 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

# Figure 216: T-cell pTfh-homing - CXCR5/CCR4 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 217: T-cell pTfh-homing - CXCR5/CXCR3 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 218: T-cell pTfh-homing - CXCR5/CXCR3 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 219: T-cell pTfh-homing - CXCR5/CXCR3 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 220: T-cell pTfh-effector function - CXCR5/IFNg (%) Rise over Time by Treatment Group – Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 221: T-cell pTfh-effector function - CXCR5/IFNg (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

### Figure 222: T-cell pTfh-effector function - CXCR5/IFNg (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 223: T-cell pTfh-effector function - CXCR5/TNFa (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 224: T-cell pTfh-effector function - CXCR5/TNFa (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209 Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 225: T-cell pTfh-effector function - CXCR5/TNFa (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 226: T-cell pTfh-effector function - CXCR5/IL-2 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

# Figure 227: T-cell pTfh-effector function - CXCR5/IL-2 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

## Figure 228: T-cell pTfh-effector function - CXCR5/IL-2 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

## Figure 229: T-cell pTfh-effector function - CXCR5/IL-21 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 230: T-cell pTfh-effector function - CXCR5/IL-21 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

#### Figure 231: T-cell pTfh-effector function - CXCR5/IL-21 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 232: T-cell pTfh-effector function - CXCR5/CD154 (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 233: T-cell pTfh-effector function - CXCR5/CD154 (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo.]

## Figure 234: T-cell pTfh-effector function - CXCR5/CD154 (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

# Figure 235: T-cell pTfh-effector function - CXCR5/ICOS (%) Rise over Time by Treatment Group - Oral Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 22, 36, 57, 114, and 209. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo.]

## Figure 236: T-cell pTfh-effector function - CXCR5/ICOS (%) Rise over Time by Treatment Group – Sublingual Cohort, mITT Population

# Figure 237: T-cell pTfh-effector function - CXCR5/ICOS (%) Rise over Time by Treatment Group – Intradermal Cohort, mITT Population

[Implementation note: Timepoints presented will be Study Day 29, 50, 71, 128, and 223. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo.]

#### 14.3.1.1 Solicited Adverse Events

Figure 238: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment - Cohort A: Oral 5 µg dmLT

[Implementation Note: The figure below is an example only. 3 panels will be presented for doses 1, 2, and 3 at Post Dose Days 1 through 7.]



Figures with similar format:

- Figure 239: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment Cohort B: Oral 25 µg dmLT
- Figure 240: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment All Oral Cohorts: Placebo
- Figure 241: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment Cohort C: Sublingual 5 µg dmLT
- Figure 242: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment Cohort D: Sublingual 25 µg dmLT
- Figure 243: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment All Sublingual Cohorts: Placebo
- Figure 244: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment Cohort E: Intradermal 0.3 µg dmLT

[Implementation Note: 2 panels will be presented for doses 1 and 2 at Post Dose Days 1 through 7.]

Figure 245: Maximum Severity of Solicited Systemic Symptoms per Subject by Day Post Treatment – Cohort E: Intradermal Placebo

[Implementation Note: 2 panels will be presented for doses 1 and 2 at Post Dose Days 1 through 7.]

Figure 246: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment – Cohort A: Oral 5 µg dmLT

[Implementation Note: The figure below is an example only. 3 panels will be presented for doses 1, 2, and 3 at Post Dose Days 1 through 7.]



#### Figures with similar format:

- Figure 247: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment Cohort B: Oral 25 µg dmLT
- Figure 248: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment All Oral Cohorts: Placebo
- Figure 249: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment Cohort C: Sublingual 5 µg dmLT
- Figure 250: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment Cohort D: Sublingual 25 µg dmLT
- Figure 251: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment All Sublingual Cohorts: Placebo
- Figure 252: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment Cohort E: Intradermal 0.3 µg dmLT

Implementation Note: 2 panels will be presented for doses 1 and 2 at Post Dose Days 1 through 7.]

Figure 253: Maximum Severity of Solicited Local Symptoms per Subject by Day Post Treatment – Cohort E: Intradermal Placebo

Implementation Note: 2 panels will be presented for doses 1 and 2 at Post Dose Days 1 through 7.]

#### 14.3.5 Displays of Laboratory Results

Figure 254: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine, Oral Cohorts

[Implementation note: The figure below is an example only. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo at Baseline and Study Days 36 and 57.]



Figures with similar format:

Figure 255: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine, Sublingual Cohorts

[Implementation note: Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo at Baseline and Study Days 36 and 57.]

Figure 256: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Creatinine, Intradermal Cohort

[Implementation note: Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Days 50 and 71.]

## Figure 257: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Alanine Aminotransferase, Oral Cohorts

[Implementation note: Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo at Baseline and Study Days 36 and 57.]

Figure 258: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Alanine Aminotransferase, Sublingual Cohorts

[Implementation note: Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo at Baseline and Study Days 36 and 57.]

Figure 259: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Alanine Aminotransferase, Intradermal Cohort

[Implementation note: Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Days 50 and 71.]

Figure 260: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Total Bilirubin, Sublingual Cohorts

[Implementation note: Groups presented will be Cohort D: Sublingual 25 µg dmLT and Cohort D: Placebo at Baseline and Study Days 36 and 57.]

Figure 261: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Total Bilirubin, Intradermal Cohort

[Implementation note: Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Days 50 and 71.]

Figure 262: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Albumin, Oral Cohorts

[Implementation note: Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo at Baseline and Study Day 57.]

Figure 263: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Albumin, Sublingual Cohorts

[Implementation note: Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo at Baseline and Study Day 57.]

Figure 264: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Albumin, Intradermal Cohort

[Implementation note: Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Day 71.]

Figure 265: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – White Blood Cell, Oral Cohorts

[Implementation note: Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo at Baseline and Study Day 57.]

## Figure 266: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – White Blood Cell, Sublingual Cohorts

[Implementation note: Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, Jand All Sublingual Cohorts: Placebo at Baseline and Study Day 57.]

Figure 267: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – White Blood Cell, Intradermal Cohort

[Implementation note: Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Day 71.]

Figure 268: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Absolute Neutrophil Count, Oral Cohorts

[Implementation note: Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo at Baseline and Study Day 57.]

Figure 269: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Absolute Neutrophil Count, Sublingual Cohorts

[Implementation note: Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo at Baseline and Study Day 57.]

Figure 270: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Absolute Neutrophil Count, Intradermal Cohort

[Implementation note: Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Day 71.]

Figure 271: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, Sex, and Treatment Group – Hemoglobin, Oral Cohorts

[Implementation note: As Figure 143 with two panels for male and female participants. Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo at Baseline and Study Day 57.]

Figure 272: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, Sex, and Treatment Group – Hemoglobin, Sublingual Cohorts

[Implementation note: As Figure 143 with two panels for male and female participants. Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo at Baseline and Study Day 57.]

Figure 273: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, Sex, and Treatment Group – Hemoglobin, Intradermal Cohort

[Implementation note: As Figure 143 with two panels for male and female participants. Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Day 71.]

## Figure 274: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Platelets, Oral Cohorts

[Implementation note: Groups presented will be Cohort A: Oral 5 µg dmLT, Cohort B: Oral 25 µg dmLT, and All Oral Cohorts: Placebo at Baseline and Study Day 57.]

## Figure 275: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Platelets, Sublingual Cohorts

[Implementation note: Groups presented will be Cohort C: Sublingual 5 µg dmLT, Cohort D: Sublingual 25 µg dmLT, and All Sublingual Cohorts: Placebo at Baseline and Study Day 57.]

## Figure 276: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Treatment Group – Platelets, Intradermal Cohort

[Implementation note: Groups presented will be Cohort E: Intradermal 0.3 µg dmLT and Cohort E: Intradermal Placebo at Baseline and Study Day 71.]

#### APPENDIX 3. LISTINGS MOCK-UPS

#### **LISTINGS**

| Listing 1: | 16.2.1: Early Terminations or Discontinued Subjects | 306 |
|---|---|---|
| Listing 2: | 16.2.2.1: Subject-Specific Protocol Deviations | 307 |
| Listing 3: | 16.2.2.2: Non-Subject-Specific Protocol Deviations | 308 |
| Listing 4: | 16.2.3: Subjects Excluded from Analysis Populations | 309 |
| Listing 5: | 16.2.4.1: Demographic Data | 310 |
| Listing 6: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 311 |
| Listing 7: | 16.2.6.1: Individual Immunogenicity Response Data – Serum IgA & IgG | 313 |
| Listing 8: | 16.2.6.2: Individual Immunogenicity Response Data – Serum LT Neutralization | 313 |
| Listing 9: | 16.2.6.3: Individual Immunogenicity Response Data – ASC IgA & IgG | 313 |
| Listing 10: | 16.2.6.4: Individual Immunogenicity Response Data – ALS IgA & IgG | 314 |
| Listing 11: | 16.2.6.5: Individual Immunogenicity Response Data – ASC Homing Markers | 314 |
| Listing 12: | 16.2.6.6: Individual Immunogenicity Response Data – Fecal IgA | 315 |
| Listing 13: | 16.2.6.7: Individual Immunogenicity Response Data – Salivary IgA | 315 |
| Listing 14: | 16.2.6.8: Individual Immunogenicity Response Data – B-Memory Cell | 316 |
| Listing 15: | 16.2.6.9: Individual Immunogenicity Response Data – T Cell Memory Responses by CyTOF | 316 |
| Listing 16: | 16.2.7.1: Solicited Events – Systemic Symptoms Oral Cohorts | 318 |
| Listing 17: | 16.2.7.1: Solicited Events – Systemic Symptoms Sublingual Cohorts | 318 |
| Listing 18: | 16.2.7.1: Solicited Events – Systemic Symptoms Intradermal Cohorts | 318 |
| Listing 19: | 16.2.7.2: Solicited Events – Local Symptoms Oral Cohorts | 319 |
| Listing 20: | 16.2.7.2: Solicited Events – Local Symptoms Sublingual Cohorts | 319 |
| Listing 21: | 16.2.7.2: Solicited Events – Local Symptoms Intradermal Cohorts | 319 |
| Listing 22: | 16.2.7.3: Unsolicited Adverse Events | 320 |
| Listing 23: | 16.2.8.1: Clinical Laboratory Results – Chemistry | 321 |
| Listing 24: | 16.2.8.2: Clinical Laboratory Results – Hematology | 322 |
| Listing 25: | 16.2.9.1: Vital Signs | 323 |
| Listing 26: | 16.2.9.2: Physical Exam Findings | 324 |
| Listing 27: | 16.2.10: Concomitant Medications | 325 |

| Version | 1.0 |
|---------|-----|
| 6AUG20 | )21 |

| 200 |
|-----|
| 326 |
| 326 |
| 327 |
| 327 |
| 327 |

#### 16.1.6: Listing of Subjects Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

#### 16.2 Database Listings by Subject

#### **16.2.1 Discontinued Subjects**

#### **Listing 1:** 16.2.1: Early Terminations or Discontinued Subjects

| Treatment Group | Subject ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

#### 16.2.2 Protocol Deviations

#### **Listing 2:** 16.2.2.1: Subject-Specific Protocol Deviations

| Treatment<br>Group | Subject ID | DV Number | Deviation | Deviation<br>Category | Study Day | Reason for<br>Deviation | Deviation<br>Resulted<br>in AE? | Deviation Resulted<br>in Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### **Listing 3:** 16.2.2.2: Non-Subject-Specific Protocol Deviations

| Site | Start Date | Deviation | End Date | Reason for<br>Deviation | Deviation<br>Resulted in<br>Subject<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.3 Subjects Excluded from the Immunogenicity Analysis

#### Listing 4: 16.2.3: Subjects Excluded from Analysis Populations

| Treatment Group | Subject ID | Analyses in which<br>Subject is Included | Analyses from which<br>Subject is Excluded | Results Available? | Reason Subject Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, ITT, PP] | [e.g., Safety, ITT, PP, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

#### 16.2.4 Demographic Data

#### Listing 5: 16.2.4.1: Demographic Data

| Treatment Group | Subject ID | Sex | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|

#### Listing 6: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

| Treatment<br>Group | Subject ID | MH Number | Medical History Term | Condition Start Day | Condition End Day | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|---|

#### 16.2.5 Compliance and/or Drug Concentration Data

Not applicable.

#### 16.2.6 Individual Immunogenicity Response Data

Listing 7: 16.2.6.1: Individual Immunogenicity Response Data – Serum IgA & IgG

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | IgA Titer | IgA Fold Rise | IgG Titer | IgG Fold Rise |
|---|---|---|---|---|---|---|---|

#### Listing 8: 16.2.6.2: Individual Immunogenicity Response Data – Serum LT Neutralization

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | Titer | Fold Rise |
|---|---|---|---|---|---|

#### Listing 9: 16.2.6.3: Individual Immunogenicity Response Data – ASC IgA & IgG

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | IgA<br>ASC / 10 <sup>6</sup> PBMC | IgG<br>ASC / 10 <sup>6</sup> PBMC |
|---|---|---|---|---|---|

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | IgA<br>ASC / 10 <sup>6</sup> PBMC | IgG<br>ASC / 10 <sup>6</sup> PBMC |
|---|---|---|---|---|---|

#### Listing 10: 16.2.6.4: Individual Immunogenicity Response Data – ALS IgA & IgG

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | IgA Titer | IgA Fold Rise | IgG Titer | IgG Fold Rise |
|---|---|---|---|---|---|---|---|

#### **Listing 11:** 16.2.6.5: Individual Immunogenicity Response Data – ASC Homing Markers

| | | | | IgA | | Ig | gG |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject ID | Planned<br>Time Point | Actual Study<br>Day | dmLT-specific IgA Gut<br>Homing ASC (α4/β7+) | Total IgA Gut Homing ASC (α4/β7+) | dmLT-specific IgA Gut<br>Homing ASC (α4/β7+) | Total IgG Gut Homing ASC (α4/β7+) |

| | | | | IgA | | IgG | |
|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Subject ID | Planned<br>Time Point | Actual Study<br>Day | dmLT-specific IgA Gut<br>Homing ASC (α4/β7+) | Total IgA Gut Homing ASC (α4/β7+) | dmLT-specific IgA Gut<br>Homing ASC (α4/β7+) | Total IgG Gut Homing ASC (α4/β7+) |

#### Listing 12: 16.2.6.6: Individual Immunogenicity Response Data – Fecal IgA

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | dmLT specific<br>IgA Titer | dmLT specific IgA<br>Fold-Rise | dmLT specific/ Total<br>IgA Titer | dmLT specific/ Total<br>IgA Fold-Rise |
|---|---|---|---|---|---|---|---|

#### Listing 13: 16.2.6.7: Individual Immunogenicity Response Data – Salivary IgA

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | dmLT specific<br>IgA Titer | dmLT specific IgA<br>Fold-Rise | dmLT specific/ Total<br>IgA Titer | dmLT specific/ Total<br>IgA Fold-Rise |
|---|---|---|---|---|---|---|---|

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | dmLT specific<br>IgA Titer | dmLT specific IgA<br>Fold-Rise | dmLT specific/ Total<br>IgA Titer | dmLT specific/ Total<br>IgA Fold-Rise |
|---|---|---|---|---|---|---|---|

#### Listing 14: 16.2.6.8: Individual Immunogenicity Response Data – B-Memory Cell

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | IgA dmLT-specific | IgA dmLT-specific<br>/IgA total | IgG dmLT-specific | IgG dmLT-specific<br>/IgG total |
|---|---|---|---|---|---|---|---|

#### Listing 15: 16.2.6.9: Individual Immunogenicity Response Data – T Cell Memory Responses by CyTOF

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | Assay | Cell<br>Expression | Result |
|---|---|---|---|---|---|---|

| Treatment Group | Subject ID | Planned Time Point | Actual Study Day | Assay | Cell<br>Expression | Result |
|---|---|---|---|---|---|---|

#### 16.2.7 Adverse Events

**Listing 16:** 16.2.7.1: Solicited Events – Systemic Symptoms Oral Cohorts

| Treatment<br>Group | Subject ID | Dose Number | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity | Attributed to<br>Alternate<br>Etiology? <sup>b</sup> | Alternate Etiology |
|---|---|---|---|---|---|---|---|---|
| | | | | MA | | | | |
| | | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

Listings with similar format:

**Listing 17:** 16.2.7.1: Solicited Events – Systemic Symptoms Sublingual Cohorts

**Listing 18:** 16.2.7.1: Solicited Events – Systemic Symptoms Intradermal Cohorts

<sup>&</sup>lt;sup>b</sup> Grade 3 events only.

**Listing 19:** 16.2.7.2: Solicited Events – Local Symptoms Oral Cohorts

| Treatment Group | Subject ID | Dose Number | Post Dose Day | Assessmenta | Symptom | Severity |
|---|---|---|---|---|---|---|
| | | | | MA | | |
| | | | | Clinic | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by subject on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.)

Listings with similar format:

**Listing 20:** 16.2.7.2: Solicited Events – Local Symptoms Sublingual Cohorts

**Listing 21:** 16.2.7.2: Solicited Events – Local Symptoms Intradermal Cohorts

#### Listing 22: 16.2.7.3: Unsolicited Adverse Events

| Adverse<br>Event | Associated with Dose No. | No. of Days Post Associated Dose (Duration) | Severity | SAE? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken with<br>Study<br>Treatment | Subject<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System<br>Organ Class | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | | | | | | | | | | | |
| Treatment ( | Group: , Subject | ID: , AE Numbe | er: | | | | | | | | |
| Comments: | | | | | | | | | | ' | |
| Note: For a | dditional details | s about SAEs, se | ee Table 122. | | | | | | | | |

#### 16.2.8 Individual Laboratory Measurements

#### **Listing 23:** 16.2.8.1: Clinical Laboratory Results – Chemistry

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study Day | Sex | Age (years) | Laboratory Parameter (Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

#### **Listing 24:** 16.2.8.2: Clinical Laboratory Results – Hematology

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual<br>Study<br>Day | Sex | Age<br>(years) | Laboratory Parameter<br>(Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.9 Vital Signs and Physical Exam Findings

Listing 25: 16.2.9.1: Vital Signs

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Temperature<br>(°C) | Systolic Blood<br>Pressure<br>(mmHg) | Diastolic Blood<br>Pressure<br>(mmHg) | Heart Rate<br>(beats/min) | Weight<br>(kg) | Height (cm) |
|---|---|---|---|---|---|---|---|---|---|

#### Listing 26: 16.2.9.2: Physical Exam Findings

| Treatment<br>Group | Subject ID | Planned Time<br>Point | Actual Study<br>Day | Body System | Abnormal Finding | Reported as an AE?<br>(AE Description; Number) |
|---|---|---|---|---|---|---|

#### **16.2.10** Concomitant Medications

#### **Listing 27:** 16.2.10: Concomitant Medications

| Treatment<br>Group | Subject ID | CM<br>Number | Medication | Medication Start<br>Day | Medication End<br>Day | Indication | Taken for an AE?<br>(AE Description;<br>Number) | Taken for a condition<br>on Medical History?<br>(MH Description;<br>Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.11 Pregnancy Reports

**Listing 28:** 16.2.11.1: Pregnancy Reports – Maternal Information

| Treatment<br>Group | Subject<br>ID | Pregnancy<br>Number | Study Day<br>Corresponding<br>to Estimated<br>Date of<br>Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or<br>Post-Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 29: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | | | | Live Births | 6 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>b</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

<sup>&</sup>lt;sup>a</sup> Preterm Birth

<sup>&</sup>lt;sup>b</sup> Term Birth

#### **Listing 30:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Subject<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

#### **Listing 31:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Subject<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome<br>(for this<br>Fetus) | Fetal Distress During Labor and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital<br>Anomalies? | Autopsy<br>Performed? | If Autopsy, Etiology<br>for Still Birth<br>Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

#### **Listing 32:** 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Subject<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|